# Supplementary Appendix: Study Protocol and Statistical Analysis Plan

**Trial:** Pragmatic Investigation of optimal Oxygen Targets (PILOT) trial

**Manuscript:** Lower, intermediate, and higher oxygen saturation targets for

mechanically ventilated critically ill adults

ClinicalTrials.gov: NCT03026322

Authors: Matthew W. Semler; Jonathan D. Casey; Bradley D. Lloyd; Pamela

G. Hastings; Margaret A. Hays; Joanna L. Stollings; Kevin G. Buell;

John H. Brems; Edward T. Qian; Kevin P. Seitz; Li Wang; Christopher J. Lindsell; Robert E. Freundlich; Jonathan P.

Wanderer; Jin H. Han; Gordon R. Bernard; Wesley H. Self; Todd W. Rice; for the PILOT Investigators and the Pragmatic Critical

Care Research Group.

# This Supplementary Appendix contains the following items:

1) Original Trial Protocol [dated 5/1/2018]

- 2) Final Trial Protocol [dated 4/7/2021]
- 3) Summary of changes to Trial Protocol
- 4) Original Statistical Analysis Plan [dated 4/2/2021]
- 5) Final Statistical Analysis Plan [dated 10/28/2021]
- 6) Summary of changes to Statistical Analysis Plan

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

# <u>Preliminary Investigation of optimal Oxygen Targets</u> (PILOT) trial

### Version 1.0

# **Principal Investigator**

Matthew W. Semler, MD, MSc
Department of Medicine
Division of Allergy, Pulmonary, and Critical Care Medicine
Vanderbilt University School of Medicine

#### Mentors

Gordon R. Bernard, MD, Wesley H. Self, MD, MPH, &
Todd W. Rice, MD, MSc
Department of Medicine
Division of Allergy, Pulmonary, and Critical Care Medicine
Vanderbilt University School of Medicine

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

# **Table of Contents:**

# Study Schema

- 1.0 Study Summary
- 2.0 Background
- 3.0 Rationale, Aims, and Hypotheses
- 4.0 Study Description
- 5.0 <u>Inclusion/Exclusion Criteria</u>
- 6.0 <u>Enrollment/Randomization</u>
- 7.0 Study Procedures
- 8.0 Risks and Benefits
- 9.0 Adverse Events
- 10.0 <u>Study Withdrawal/Discontinuation</u>
- 11.0 <u>Statistical Considerations</u>
- 12.0 Privacy/Confidentiality Issues
- 13.0 Follow-up and Record Retention
- 14.0 <u>References</u>

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

# 1.0 Study Summary

Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

**Background:** Mechanical ventilation of ICU patients universally involves titration of the fraction of inspired oxygen ( $FiO_2$ ) to maintain arterial oxygen saturation ( $SpO_2$ ). Despite decades of ICU practice, however, the optimal  $SpO_2$  target remains unknown. Higher  $SpO_2$  targets (96-100%) provide a margin of safety against hypoxia but increase exposure to hyperoxia. Lower  $SpO_2$  targets (88-92%) minimize hyperoxia, but may increase the risk of hypoxia. An intermediate  $SpO_2$  target (92-96%) may avoid the risks of both hyperoxia and hypoxia, or may expose patients intermittently to both sets of risks. Current guidelines offer divergent recommendations as to the optimal  $SpO_2$  target and clinical safety and efficacy data are lacking. Therefore, we propose a 2,250-patient cluster-randomized cluster-crossover trial comparing a lower  $SpO_2$  target (90%), an intermediate  $SpO_2$  target (94%), and a higher  $SpO_2$  target (98%) with regard to the outcome of days alive and free of invasive mechanical ventilation.

#### **Primary Aim:**

 To compare the effect of higher, intermediate, and lower SpO<sub>2</sub> targets on days alive and free of invasive mechanical ventilation among mechanically ventilated critically ill adults.

### **Primary Hypotheses:**

Use of a lower SpO<sub>2</sub> target (90%) for mechanically ventilated ICU patients will
result in more days alive and free of invasive mechanical ventilation than use of
an intermediate SpO<sub>2</sub> target (94%) or a higher SpO<sub>2</sub> target (98%).

#### **Inclusion Criteria:**

 We will include adults (≥ 18 years old) receiving mechanical ventilation through an endotracheal tube or tracheostomy who are admitted to the study ICU or for whom admission to the study ICU from the emergency department is planned.

# **Exclusion Criteria:**

We will exclude patients who are pregnant or who are prisoners.

**Consent:** Because [1] the study enrolls only patients who would have been exposed to oxygen therapy as a part of clinical care outside of the study, [2] all  $SpO_2$  targets examined are currently used in routine care in the study ICU, [3] no high-quality data suggest that the choice of  $SpO_2$  target affects clinical outcomes, and [4] during the trial treating clinicians retain discretion to control the  $SpO_2$  target when felt to be required for the safe treatment a specific patient, we feel the study qualifies as minimal risk.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

Given the minimal risk, the implementation of  $SpO_2$  targets at an ICU level, and the impracticability of consenting each patient during initiation of mechanical ventilation in the ICU or emergency department, we will request a waiver of informed consent.

**Randomization:** In the PILOT trial, the entire study ICU will be assigned to a single  $SpO_2$  target (cluster-randomized) and the ICU will switch between lower, intermediate, and higher  $SpO_2$  targets every two months in a randomly generated sequence (cluster-crossover).

#### **Study Interventions:**

- **Lower SpO<sub>2</sub> Target** FiO<sub>2</sub> will be titrated according to an oxygen therapy protocol to a target SpO<sub>2</sub> of 90% with a range considered compliant of 88-92%.
- Intermediate SpO<sub>2</sub> Target FiO<sub>2</sub> will be titrated according to an oxygen therapy protocol to a target SpO<sub>2</sub> of 94% with a range considered compliant of 92-96%.
- **Higher SpO<sub>2</sub> Target** FiO<sub>2</sub> will be titrated according to an oxygen therapy protocol to a target SpO<sub>2</sub> of 98% with a range considered compliant of 96-100%.

#### **Primary Outcome:**

• Ventilator-free days (VFDs) to study day 28, defined as the number of days from liberation from invasive mechanical ventilation to day 28 after enrollment.

### **Secondary Outcomes:**

- Secondary Clinical Outcomes: ICU mortality, in-hospital mortality, vasopressorfree days, duration of vasopressor receipt, renal replacement therapy-free days, duration of renal replacement therapy receipt, ICU-free days, ICU-length of stay, hospital length of stay.
- Secondary Organ Function Outcomes: daily SOFA score, creatinine, lactate, presence of acute respiratory distress syndrome, Stage II or greater AKI by KDIGO criteria.
- Secondary Safety Outcomes: Atrial arrhythmia, ventricular arrhythmia, cardiac arrest, pneumothorax.
- Secondary Feasibility Outcomes: SpO<sub>2</sub>, SaO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, percentage of SpO<sub>2</sub> values outside target range, <88% with FiO<sub>2</sub> <1.0, PaO<sub>2</sub> < 55 with FiO<sub>2</sub> <1.0, SpO<sub>2</sub> >98% with FiO<sub>2</sub> > 0.21, PaO<sub>2</sub> >120 with FiO<sub>2</sub> >0.21, episodes of SpO<sub>2</sub> ≤ 85% lasting > 5 minutes, PaO<sub>2</sub>/FiO<sub>2</sub> ratio.
- Secondary Process of Care Outcomes: Tidal volume, positive end expiratory
  pressure, peak airway pressure, net fluid balance, receipt of mandatory
  ventilator mode, number of arterial blood gasses, hemoglobin, red cell
  transfusion.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

# 2.0 Background

Each year 2-3 million intensive care unit (ICU) patients receive invasive mechanical ventilation,<sup>1–3</sup> at a cost of more than \$20 billion dollars.<sup>4,5</sup> Despite recent advances,<sup>6</sup> inhospital mortality among mechanically ventilated ICU patients remains 25-35%,<sup>7</sup> and survivors often face cognitive, psychiatric, and physical dysfunction.<sup>8–11</sup>

Mechanical ventilation of ICU patients universally involves titration of the fraction of inspired oxygen (FiO<sub>2</sub>) to maintain arterial oxygen saturation (SpO<sub>2</sub>). Despite decades of ICU practice, however, the optimal SpO<sub>2</sub> target remains unknown. Higher SpO<sub>2</sub> targets (96-100%) provide a margin of safety against hypoxemia, but may increase exposure to excess FiO<sub>2</sub>, hyperoxemia, and tissue hyperoxia, causing oxidative damage, <sup>12-14</sup> inflammation, <sup>15,16</sup> and increased alveolar-capillary permeability. Lower SpO<sub>2</sub> targets (88-92%) minimize hyperoxia, <sup>6,18,19</sup> but may increase the risk of hypoxemia, tissue hypoxia, and organ dysfunction. An intermediate SpO<sub>2</sub> target (92-96%) may avoid the risks of both hyperoxia and hypoxia, or, conversely, may expose patients intermittently to both sets of risks.

Current guidelines offer divergent recommendations – ranging from tolerating SpO $_2$  values as low as 88% (ARDS Network) $^{22,23}$  to pursuing SpO $_2$  values as high as 98% (British Thoracic Society) $^{24}$ . The relative risks and benefits of different SpO $_2$  targets have been extensively examined in the setting of the neonatal ICU, $^{25-28}$  but have only been investigated in adult ICU patients in three small trials. $^{29-31}$  Targeting lower SpO $_2$  resulted in improved survival in one trial and trends toward improved survival in the other two.

In clinical practice, however, hyperoxemia remains common.<sup>32,33</sup> In our recent observational study of 2,200 mechanically ventilated ICU patients at 50 centers across

the United States (see Figure), the majority of patients had a lowest PaO<sub>2</sub> value on the first study day > 100 mm Hg (~SpO<sub>2</sub> > 97%). The wide variation in current practice (frequently favoring higher SpO<sub>2</sub> targets), conflicting guidelines, and pilot trial data favoring lower SpO<sub>2</sub> targets have led to calls for a large, randomized trial to determine the effect of SpO<sub>2</sub> target on patient outcomes.<sup>18</sup>



Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

#### 3.0 Rationale, Aims, and Hypotheses

In order to determine the effect of SpO<sub>2</sub> targets during mechanical ventilation of critically ill adults on clinical outcomes, a randomized trial is needed.

### **Study Aims:**

• **Primary:** To compare the effect of higher, intermediate, and lower SpO<sub>2</sub> targets on days alive and free of invasive mechanical ventilation among mechanically ventilated critically ill adults.

### Secondary:

- To evaluate the effect of the same intervention in the same population on pre-specified Secondary Clinical Outcomes, Secondary Organ Function Outcomes, Secondary Safety Outcomes, Secondary Feasibility Outcomes, and Secondary Process of Care Outcomes.
- To evaluate the effect of the same intervention on days alive and free of invasive mechanical ventilation in clinically relevant pre-specified patient subgroups.

# **Study Hypotheses:**

• **Primary:** Use of a lower SpO<sub>2</sub> target (90%) for mechanically ventilated ICU patients will result in more days alive and free of invasive mechanical ventilation than use of an intermediate SpO<sub>2</sub> target (94%) or a higher SpO<sub>2</sub> target (98%).

#### Secondary:

- Compared with use of an intermediate SpO<sub>2</sub> target (94%) or higher SpO<sub>2</sub> target (98%), use of a lower SpO<sub>2</sub> target (90%) for mechanically ventilated ICU patients will result in:
  - Lower ICU and in-hospital mortality
  - No difference between in other Secondary Clinical Outcomes
  - Lower daily SOFA score
  - Lower incidence of acute respiratory distress syndrome
  - No difference in other Secondary Organ Function Outcomes
  - No difference in Secondary Safety Outcomes
  - Lower SpO<sub>2</sub>, SaO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, and incidence of SpO<sub>2</sub> >98% with FiO<sub>2</sub> > 0.21 or PaO<sub>2</sub> >120 with FiO<sub>2</sub> >0.21
  - Higher  $PaO_2/FiO_2$  ratio and incidence of  $SpO_2 < 88\%$  with  $FiO_2 < 1.0$  or  $PaO_2 < 55$  with  $FiO_2 < 1.0$
  - No difference in episodes of SpO<sub>2</sub> ≤ 85% lasting > 5 minutes
  - No difference in Secondary Process of Care Outcomes

#### 4.0 Study Description

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

In order to address the aims outlined above, we propose the Preliminary Investigation of optimal Oxygen Targets (PILOT) trial. The PILOT trial will be a prospective, unblinded, cluster-randomized, cluster-crossover trial conducted between July 1, 2018 and June 30, 2021 in the medical ICU at Vanderbilt University Medical Center examining the effect of SpO<sub>2</sub> targets on days alive and free of mechanical ventilation among mechanically ventilated ICU patients. For the 36 months of the PILOT trial, the entire medical ICU will be assigned to a single SpO<sub>2</sub> target and the ICU will switch between lower, intermediate, and higher SpO<sub>2</sub> targets every two months in a randomly generated sequence (Figure below). Patients who fulfill inclusion criteria without meeting exclusion criteria will be enrolled at the initiation of mechanical ventilation in the study ICU or in the emergency department when admission to the study ICU is planned. The PILOT trial will control only the SpO<sub>2</sub> target and all other aspects of patients clinical care will remain at the discretion of the treating clinicians.

| | Study Year 1 | | | | | | Study Year 2 | | | | | | | Study Year 3 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug | Sept-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun |
| | 2018 | | | | 20 | 19 | | | 2020 | | | | | | 2021 | | |
| High | Mid. | Low | Mid. | Low | High | Low | Mid. | High | High | Mid. | Low | Mid. | High | Low | Mid. | High | Low |

The study ICU was randomly assigned to an SpO<sub>2</sub> target for each two-month block.

 $High = SpO_2 \text{ target } 98\% \text{ (range } 96-100\%); Mid. = SpO_2 \text{ target } 94\% \text{ (range } 92-96\%); Low = SpO_2 \text{ target } 90\% \text{ (range } 88-92\%); Mid. = SpO_2 \text{ target } 90\% \text{ (range } 98-92\%); Mid. = SpO_2 \text{ (range } 98-92\%); Mid. = SpO_2 \text{ (range } 98-92\%); Mid. = SpO_2 \text{ (range } 9$ 

#### 5.0 Inclusion and Exclusion Criteria

#### 5.1 Inclusion Criteria:

- 1. Age  $\geq$  18 years
- 2. Receiving mechanical ventilation through an endotracheal tube or tracheostomy
- 3. Admitted to the study ICU or admission to the study ICU from the emergency department is planned

#### 5.2 Exclusion Criteria:

- 1. Known pregnancy or beta hCG level greater than the laboratory upper limit of normal in a patient capable of becoming pregnant
- 2. Known to be a prisoner

# 6.0 Enrollment/Randomization

#### 6.1 Study Sites:

- Medical Intensive Care Unit at Vanderbilt University Medical Center
- Emergency Department at Vanderbilt University Medical Center

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

**6.2 Study Population:** All adults located in the study ICU (or for whom admission to the study ICU from the emergency department is planned) for whom the treating clinicians have decided invasive mechanical ventilation is required will be enrolled unless meeting exclusion criteria. Patients will be included regardless of age, gender, race, weight or body mass index, initial oxygen saturation, or other clinical factors.

**6.3 Enrollment:** All adult patients who do not meet exclusion criteria will be enrolled immediately upon receipt of invasive mechanical ventilation in the study ICU or in the emergency department when admission to the study ICU is planned.

#### 6.4 Consent:

All patients receiving invasive mechanical ventilation in an intensive care unit receive oxygen therapy titrated to maintain  $SpO_2$  as a part of routine care. In clinical practice, 98% of  $SpO_2$  values experienced by mechanically ventilated adults fall between 88-100%. Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: [1] tolerating  $SpO_2$  values as low as 88% (NIH/NHLBI ARDS Network),  $^{22}$  [2] titrating within the range 92-96% (Thoracic Society of Australia and New Zealand),  $^{34}$  or [3] pursuing  $SpO_2$  values as high as 98% (British Thoracic Society). We have  $SpO_2$  target (90%), intermediate  $SpO_2$  target (94%), and higher  $SpO_2$  target (98%) examined in this study are all intermittently used in routine care in the study ICU and recommended by at least one international guideline. There are currently no high-quality data to suggest that one  $SpO_2$  target is better than the others with regard to clinical outcomes. Although there are no clear data to support the choice of  $SpO_2$  target, during the PILOT trial, treating clinicians in the study ICU will be allowed to change the  $SpO_2$  target at any point if it is felt to be required for the safe treatment a specific patient.

Because the interventions studied [1] are used as part of routine care in the study ICU, [2] are interventions o which the patient would be expected even if not participating in the study, [3] have no prior data to suggest the superiority of one approach over the other, and [4] are equivalent options from the perspective of the treating clinicians (otherwise the treating clinician retains control of  $SpO_2$  target), we feel the study presents minimal risk.

Additionally, obtaining informed consent prior to participation in the study would be impractical. Endotracheal intubation and initiation of mechanical ventilation for critically ill patients is frequently a time-sensitive procedure. Despite the availability of a formal informed consent document for the endotracheal intubation and initiation of mechanical ventilation, time allows discussion of risks and benefits in less than 10% of airway management events in the study ICU. The oxygen titration protocol used to target SpO2 in this trial begins immediately at the initiation of mechanical ventilation to capture the period of mechanical ventilation with the highest risk for hyperoxia and hypoxia. Moreover, in this cluster-randomized trial, the entire ICU is assigned to a single SpO<sub>2</sub> target delivered by the unit's respiratory therapist through a unit-wide oxygen

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

titration protocol. Obtaining informed consent from every eligible patient in the ICU each day would be logistically infeasible and patients who declined to participate would need to be transferred between ICUs which might adversely impact their care.

Because the study presents minimal risk, would not adversely affect the welfare or privacy rights of the participant, and consent would be impracticable, we will request a waiver of informed consent.

#### 6.5 Randomization:

During each two-month block of the study, the ICU will be assigned to either a higher  $SpO_2$  target (98%), an intermediate  $SpO_2$  target (94%), or a lower  $SpO_2$  target (90%). The order of study group assignments will be generated by computerized randomization using permuted blocks of 3 to minimize the impact of seasonal variation. The last 7 days of each two-month block will be a washout period during which the ICU will continue to target the assigned  $SpO_2$  but new patients will not be enrolled. Assuming a duration of mechanical ventilation similar to that observed for mechanically ventilated patients admitted to the study ICU in a prior year (median 3 [IQR 3-5] days), a 7-day washout period will ensure that 98% patients do not experience a "crossover" from one assigned  $SpO_2$  target to another.

#### 7.0 Study Procedures

# 7.1 Study Interventions

**Choice of SpO<sub>2</sub> targets:** In clinical practice, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adults fall between 88-100%.<sup>32,33</sup> Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: [1] tolerating SpO<sub>2</sub> values as low as 88% (NIH/NHLBI ARDS Network),<sup>22</sup> [2] titrating within the range 92-96% (Thoracic Society of Australia and New Zealand),<sup>34</sup> or [3] pursuing SpO<sub>2</sub> values as high as 98% (British Thoracic Society).<sup>24</sup> The PILOT trial will

have three study groups, each emulating an approach to SpO<sub>2</sub> targets represented in guidelines and clinical practice (Table).

| Study Group | SpO <sub>2</sub> target | SpO <sub>2</sub> range | PaO <sub>2</sub> target | PaO₂ range |
|---|---|---|---|---|
| Lower SpO <sub>2</sub> target | 90% | 88-92% | 60 mm Hg | 55-65 mm Hg |
| Intermediate SpO <sub>2</sub> target | 94% | 92-96% | 70 mm Hg | 65-80 mm Hg |
| Higher SpO <sub>2</sub> target | 98% | 96-100% | 110 mm Hg | > 80 mm Hg |

The  $SpO_2$  target and range of  $SpO_2$  values considered to be compliant are displayed for each study group.  $PaO_2$  will be used to guide oxygen titration for participants without functioning pulse oximetry monitoring.

**SpO<sub>2</sub> versus PaO<sub>2</sub>:** SpO<sub>2</sub> is measured continuously via non-invasive pulse oximetry for nearly all mechanically ventilated ICU patients. In contrast, PaO<sub>2</sub> is assessed via arterial puncture intermittently and selectively, particularly among more severely ill patients

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

earlier in their clinical course. Similar to prior studies of oxygen therapy during mechanical ventilation<sup>29</sup>, the PILOT trial will target ranges of  $SpO_2$  for all patients with functioning non-invasive pulse oximetry monitoring. For patients in the PILOT trial for whom non-invasive pulse oximetry monitoring is unavailable (e.g., inadequate plethysmography signal due to hypoperfusion),  $PaO_2$  values corresponding to the assigned  $SpO_2$  target will be used to guide oxygen therapy (see above Table).<sup>35</sup>

Oxygen Titration Protocol: In current usual care in the study ICU, titration of  $FiO_2$  to maintain  $SpO_2$  for mechanically ventilated adults is performed by respiratory therapists, with input from nurses and physicians. Other aspects of mechanical ventilation (selection of tidal volume, titration of positive end-expiratory pressure, screening for spontaneous breathing trials) are governed by respiratory therapy protocols jointly developed by respiratory therapy and physician leaders. In preparation for the PILOT trial, we have collaborated with respiratory therapy leaders in the study ICU to develop an oxygen titration protocol for each  $SpO_2$  target group (see Figure below). Each block of the study, the mechanical ventilators in the study ICU will be outfitted by study personnel with paper copies of the oxygen titration protocol targeting the assigned  $SpO_2$ . The oxygen titration protocol will also be available to respiratory therapists, nurses, and physicians through the electronic order entry system.





Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center



<u>Initiation of Mechanical Ventilation:</u> The oxygen titration protocol guides respiratory therapists and treating clinicians to begin titrating FiO2 to the target SpO2 value within 15 minutes of the initiation of mechanical ventilation in the participating ED or ICU. This initial 15-minute window is intended to give the treating clinicians adequate time after emergent tracheal intubation to stabilize the patient's hemodynamics and initiate basic ventilator settings, but also to intervene early enough to control the FiO2 and SpO2 during the critical early period of mechanical ventilation when exposure to excess FiO2 and hyperoxemia is most common.

<u>Oxygen Titration during Mechanical Ventilation:</u> SpO<sub>2</sub> will be assessed by continuous pulse oximetry. The respiratory therapist managing the patient's ventilator will target an SpO<sub>2</sub> value of 98% in the higher SpO<sub>2</sub> group, 94% in the intermediate SpO<sub>2</sub> group, and 90% in the lower SpO<sub>2</sub> group. The respiratory therapist will titrate FiO<sub>2</sub> as directed by the oxygen titration protocol when SpO<sub>2</sub> values are outside of the range 96-98% in the higher SpO<sub>2</sub> group, 92-96% in the intermediate SpO<sub>2</sub> group, and 88-92% in the lower SpO<sub>2</sub> group. SpO<sub>2</sub> will be reassessed 5 minutes after each change in FiO<sub>2</sub>.

<u>Liberation from Mechanical Ventilation:</u> Each day of mechanical ventilation, all patients in the study ICU are assessed for safety of a spontaneous awakening trial (SAT) and spontaneous breathing trial (SBT)<sup>36</sup> using the SAT and SBT safety criteria from the

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

Awakening and Breathing Controlled trial.<sup>37</sup> To prevent patients in the higher SpO<sub>2</sub> target group from experiencing delays in qualifying for an SBT based on receipt of higher FiO<sub>2</sub> to achieve the higher SpO<sub>2</sub> target, during the PILOT trial we will allow patients in all groups to qualify for an SBT with an FiO<sub>2</sub>  $\leq$  0.6. Definitions of SAT and SBT failure and the ventilator settings and duration of the SBT will not be changed from those used in the ABC trial and during usual care in the study ICU. For patients who have passed an SBT and SAT, the decision to discontinue invasive mechanical ventilation will be made by the treating clinicians.

**Modification of SpO<sub>2</sub> Targets:** At any time during the course of the study, if a treating clinician feels an SpO<sub>2</sub> target other than that assigned by the study is required for the safe treatment of a specific patient, the SpO<sub>2</sub> target for that patient may be modified. To modify the target, the supervising physician will complete a one-page SpO<sub>2</sub> target modification sheet documenting the rationale for modifying the target and prompting reassessment of the need for modification every twelve hours. Details of each SpO<sub>2</sub> target modification will be collected and monitored. In our prior cluster-crossover trial using the same approach to modification of therapy assignment, treating clinicians exercised the ability to modify the assigned therapy for < 5% of patients.<sup>38</sup>

Anticipated examples of conditions for which treating clinicians may elect to override the assigned SpO2 target include:

- pneumothorax,
- pneumomediastinum,
- carbon monoxide poisoning,
- decompression sickness,
- bleomycin toxicity,
- paraguat toxicity

SpO<sub>2</sub> Monitoring: For all mechanically ventilated patients in the study ICU, SpO<sub>2</sub> is continuously monitored using Nellcor™ SpO<sub>2</sub> Adhesive Sensors (Medtronic, Minneapolis, MN), which measure changes in red and infrared light absorption in an arteriolar bed throughout the pulse cycle to report a non-normalized real-time plethysmographic waveform and arterial hemoglobin saturation values averaged over the prior 6 seconds with a mean difference between SpO<sub>2</sub> and SaO<sub>2</sub> < 2% for SpO<sub>2</sub> values 80-100%.<sup>39</sup> Plethysmography and SpO<sub>2</sub> values are displayed [1] on IntelliVue MP90 bedside patient monitors (PHILIPS, Amsterdam, Netherlands) in each ICU room, [2] on telemetry monitors located at ICU nursing stations and adjacent to the respiratory therapy office, and [3] in real-time in the institutional EHR, available from any physical location. SpO<sub>2</sub> values are archived every 60 seconds into an intuitional data warehouse.<sup>40,41</sup> Collecting SpO<sub>2</sub> values every 60 seconds will allow the PILOT trial report with far greater accuracy the incidence, severity, and duration of desaturation than prior trials in which SpO<sub>2</sub> values were collected every 4-24 hours.<sup>29,30</sup>

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

**Feedback on SpO<sub>2</sub> Target Adherence:** [1] During the study, the IntelliVue MP90 bedside patient monitors in each room will be set to generate a low priority alarm for SpO<sub>2</sub> values 1-3% outside the assigned target range and a high priority alarm for SpO<sub>2</sub> values ≥ 4% outside the assigned target range (see Figure below). For example, for patients in the lower SpO<sub>2</sub> target group, SpO<sub>2</sub> values 88-92% will generate no alarm, SpO<sub>2</sub> values 85-87% or 93-95% will generate a low priority alarm, and SpO<sub>2</sub> values ≤ 84% or ≥ 96% will generate a high-priority alarm. [2] For the first 6 months of the PILOT trial, study personnel will remotely monitor SpO<sub>2</sub> values in real-time 8am-5pm Monday through

Friday and during a 10% sample of night and weekend hours to identify instances of lag between out of range SpO<sub>2</sub> values and FiO<sub>2</sub> titration, provide feedback and reinforcement to bedside nurses and respiratory therapists, and identify any barriers to SpO<sub>2</sub> target compliance. [3] For the entire period of the PILOT trial, study personnel will attend quarterly respiratory therapy group meetings, monthly nursing unit board meetings, and



monthly ICU physician leadership meetings to educate staff about the study, solicit safety concerns and adverse events, and identify and address barriers to  $SpO_2$  target compliance. This approach to daily monitoring and intermittent feedback to clinical personnel successfully achieved 95% compliance with the assigned intervention in a prior cluster-crossover trial in the same ICU.<sup>38</sup>

**Co-interventions:** Institutional protocols in the study setting will ensure that mechanically ventilated patients in PILOT receive: [1] ventilation targeting 6 mL/kg of predicted body weight and plateau pressure  $\leq$  30 cm H<sub>2</sub>O,<sup>6</sup> [2] PEEP titration according to the ARDSNet Lower PEEP/higher FiO<sub>2</sub> table (except for patients with severe ARDS, for

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

whom the Higher PEEP/lower  $FiO_2$  table is applied),  $^{42,43}$  [3] management of pain, agitation, and delirium  $^{44}$  targeting Critical Care Pain Observation Tool (CPOT),  $^{45}$  Richmond Agitation-Sedation Scale (RASS),  $^{46,47}$  and Confusion Assessment Method for the ICU (CAM-ICU) scores,  $^{48,49}$  and [4] daily spontaneous awakening trials (SAT) and spontaneous breathing trials (SBT).  $^{36,37}$ 

- **7.2 Blinding:** Similar to prior  $SpO_2$  target studies among critically ill adults<sup>29,30</sup>, patients and clinicians will not be blinded to study group assignment. Observer bias will be minimized by use of objective endpoints collected *in duplicate* by [1] study personnel blinded to group assignment and [2] automated data extraction from the EHR (see *Data Collection* below).
- **7.3 Data Collection:** The PILOT trial will primarily use structured data collected in routine clinical care, exported daily from the institution's EHR into an Enterprise Data Warehouse, along with data from the patient registration, billing, and laboratory clinical information systems. We have previously validated the quality of this method of data collection against the reference standard of two-physician manual chart review, <sup>50</sup> and the planned approach to electronic dataset generation for the PILOT trial has already been successfully employed for the conduct of three prior pragmatic trials. <sup>38,38,51</sup>

#### **Electronically extracted data elements will include:**

Enrollment (Day 0): age; sex; race; ethnicity; height, weight; APACHE II score; SOFA score; Glasgow Coma Scale score; Elixhauser Comorbidity Index; vital signs (temperature, heart rate, systolic blood pressure, diastolic blood pressure, SpO<sub>2</sub>); mechanical ventilator settings (mode, set and exhaled tidal volume, set and actual respiratory rate, positive end-expiratory pressure, peak pressure, FiO<sub>2</sub>); serum laboratory values (white blood cell count, hemoglobin, platelet count, sodium, potassium, bicarbonate, creatinine, bilirubin, alanine aminotransferase, aspartate aminotransferase, lactate, arterial pH, PaO<sub>2</sub>, SaO<sub>2</sub>).

<u>Daily On-Study (Days 0-28):</u> Vital signs, ventilator settings, and serum laboratory values (as above); net fluid balance; receipt of red cell transfusion; number of arterial blood gases; SOFA score; ARDS by Berlin criteria;<sup>56</sup> Stage II or greater AKI by KDIGO criteria;<sup>57</sup> atrial arrhythmia, ventricular arrhythmia, cardiac arrest, or pneumothorax.

<u>Termination (Days 0-28)</u>: Vital status at 28 days; time of liberation from invasive mechanical ventilation; receipt and duration of vasopressors; receipt and duration of renal replacement therapy; duration of ICU and hospital admission.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

Data elements collected manually by study personnel will include: [1] all data elements for a randomly selected 10% of participants to ensure the quality of electronically extracted data, [2] all primary and secondary outcomes collected at study termination for 100% of participants to ensure duplicate data collection of key study outcomes, and [3] any data elements for which electronic data extraction has not been developed and validated, including etiology of respiratory failure, indication for mechanical ventilation, protocol violations, and adverse events. Data will be stored, curated, and secured in the online database, REDCap.<sup>58</sup>

#### 7.4 Outcome Measures

**Primary Outcome:** Ventilator-free days (VFDs) to study day 28, defined as the number of days from liberation from invasive mechanical ventilation to day 28 after enrollment. Patients who continue to receive invasive mechanical ventilation at day 28 or have died prior to day 28 will receive zero VFDs. For patients who return to invasive mechanical ventilation and are subsequently liberated from invasive mechanical ventilation prior to day 28, VFDs will be counted from final liberation from mechanical ventilation. We chose VFDs as the primary outcome for the PILOT trial as choice of SpO<sub>2</sub> target may simultaneously affect both mortality and duration of invasive mechanical ventilation.

# **Secondary Clinical Outcomes:**

- 1. ICU mortality
- 2. In-hospital mortality
- 3. Vasopressor-free days
- 4. Duration of vasopressor receipt
- 5. Renal replacement therapy-free days
- 6. Duration of renal replacement therapy receipt
- 7. ICU-free days
- 8. ICU-length of stay
- 9. Hospital length of stay.

**Secondary Organ Function Outcomes:** (All secondary organ function outcomes will employ only laboratory values and imaging obtained as a part of routine clinical care)

- 1. Daily SOFA score
- 2. Daily creatinine
- 3. Daily lactate
- 4. Presence of acute respiratory distress syndrome
- 5. Stage II or greater AKI by KDIGO criteria

### **Secondary Safety Outcomes:**

- 1. Atrial arrhythmia
- 2. Ventricular arrhythmia

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

- 3. Cardiac arrest
- 4. Pneumothorax.

### **Secondary Feasibility Outcomes:**

- 1. SpO<sub>2</sub>
- 2. SaO<sub>2</sub>
- 3. FiO<sub>2</sub>
- 4. PaO<sub>2</sub>
- 5. Percentage of SpO<sub>2</sub> values outside target range
- 6. <88% with FiO<sub>2</sub> <1.0
- 7.  $PaO_2 < 55$  with  $FiO_2 < 1.0$
- 8.  $SpO_2 > 98\%$  with  $FiO_2 > 0.21$
- 9.  $PaO_2 > 120$  with  $FiO_2 > 0.21$
- 10. Episodes of SpO<sub>2</sub>  $\leq$  85% lasting > 5 minutes
- 11. PaO<sub>2</sub>/FiO<sub>2</sub> ratio

#### **Secondary Process of Care Outcomes:**

- 1. Tidal volume
- 2. Positive end expiratory pressure
- 3. Peak airway pressure
- 4. Net fluid balance
- 5. Receipt of mandatory ventilator mode
- 6. Number of arterial blood gasses
- 7. Hemoglobin
- 8. Red cell transfusion

#### 8.0 Risks and Benefits:

Among adult patients for whom the treating clinicians have decided invasive mechanical ventilation is required, there are currently no established risks or benefits to targeting a higher, intermediate, or lower SpO<sub>2</sub>. At this time, there is no reason to believe that participation in this study would expose patients to greater medical risks or benefits than those experienced by critically ill patients receiving invasive mechanical ventilation as a part of routine care. The greater benefit of the study would be to society in the form of improved understanding of safe and effective provision of oxygen therapy during mechanical ventilation for critically ill patients.

A potential risk to patients participating in this study involves the collection of protected health information (PHI). In order to limit the associated risks, the minimum amount of PHI necessary for study conduct will be collected. After collection, the data will be stored in a secure online database (REDCap) only accessible by the investigators. After publication, a de-identified database will be generated to protect participant privacy.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

# 9.0 Safety Monitoring and Adverse Events:

### 9.1 Safety Monitoring

The PILOT trial will take place in a high-acuity clinical care environment during delivery of a high-acuity procedure required for routine clinical care. During the time of the study intervention, the patient will have a critical care or emergency medicine nurse with a low patient-to-nurse staffing ratio, immediate access to a respiratory therapist, and a team of critical care physicians physically located on the study unit twenty-four hours a day. As a part of routine care all patients will be receiving continuous invasive or non-invasive monitoring of heart rate, blood pressure, respiratory rate, and oxygen saturation.

Study personnel will monitor compliance with the study inclusion and exclusion criteria, study protocol, and study safety measures daily. Study personnel will be readily available to answer questions at any time from patients, legally authorized representatives, or treating clinicians. If, at any point in a patient's clinical course, the treating clinicians believe an SpO2 target different from the assigned target is required for the safe treatment of the patient, the SpO2 target will be modified to the target the treating clinicians judge to be safest.

A structured plan for prospective collection of study outcomes has been specified, in addition to a process by which Adverse Events and Serious Adverse Events will be managed and reported as required to regulatory bodies.

A Data and Safety Monitoring Board (DSMB) will be appointed to oversee the study. The DSMB will be available throughout the trial to monitor enrollment, protocol compliance, safety, and adverse events. Additionally the DSMB will perform an interim analysis for safety and efficacy.

#### 9.2 Adverse Event Reporting

A system has been established to report and track clinical outcomes and adverse events (AEs). Study personnel will monitor the safety of subjects and follow AEs until the event resolves or is explained.

<u>Clinical Outcomes (not considered Adverse Events).</u> In this study of critically ill patients who are at high risk for death or other adverse outcomes due to their underlying critical illness, clinical outcomes, including death and organ dysfunction, will be systematically tracked (collected in the case report form) and will be included as part of the analyses for this study. For the purposes of reporting, death and organ dysfunction will not be recorded as AEs unless the investigator believes the event may have been caused by the study or is more severe or prolonged than expected given the underlying critical illness. This approach—considering death and organ dysfunction as outcomes rather than AEs

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

and systemically tracking expected outcomes for analysis rather than solely recording individual AEs—is common in ICU trials because these outcomes/events occur commonly in the ICU and this system mandates that data regarding death, organ dysfunction, and expected outcomes be tracked systematically for all patients and analyzed appropriately. Clinical outcomes will be systemically tracked throughout the study period. Listed below are events that will be tracked as primary or secondary clinical outcomes and will not therefore be reported as AEs during this study (unless believed to be study related and more severe or prolonged than expected given the underlying critical illness):

- 1. Death (all deaths occurring prior to hospital discharge will be reported on the CRF in the vital status at hospital discharge section);
- 2. Recurrence of respiratory failure, including need for re-intubation or non-invasive mechanical ventilation, presence of acute respiratory distress syndrome, or presence of pneumothorax;
- Circulatory failure, including cardiac arrest or shock with or without receipt of vasopressors;
- 4. Incidence of sustained atrial and ventricular arrhythmias;
- 5. Acute kidney injury, including leading to increased creatinine or receipt of renal replacement therapy;
- 6. Hepatic injury or failure leading to increased bilirubin, AST, or ALT;
- 7. Coagulation derangements leading to elevated PT/INR or PTT, DIC, thrombocytopenia, or thrombocytosis;
- 8. Lactic acidosis;
- 9. Delirium, disability, and physical or cognitive impairment believed to be newly acquired;
- 10. All values for SpO<sub>2</sub>, SaO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, or PaO<sub>2</sub>/FiO<sub>2</sub> ratio;
- 11. All values for vital signs (e.g., temperature, respiratory rate, SpO2);
- 12. Receipt of co-interventions (e.g., net fluid balance, number of arterial blood gasses, red cell transfusion)
- 13. Duration of ICU admission, ICU readmission;
- 14. Duration of hospitalization, hospital readmission;
- 15. Alterations in routine labs, including chemistries, complete blood counts, liver function tests, and hemostasis profiles.

Adverse Event Classifications. An Adverse Event (AE) will be any untoward medical occurrence for a patient enrolled in the trial that is not tracked as a clinical outcome, regardless of whether the event is considered study related or not. All AEs occurring during the observational study period will be recorded on the CRF. All AEs will then be assessed as to whether they are (1) related to study procedures, (2) serious, and/or (3) unexpected according to the following definitions:

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

I. <u>Related to study procedures.</u> AEs that the investigator suspects are related to the study will be classified as study related. Certainty of relatedness is not required as long as a reasonable possibility exists that the AE is related to a study procedure.

- II. <u>Serious.</u> AEs that meet any of the criteria below will be considered Serious Adverse Events (SAEs):
  - a. Results in death
  - Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event and NOT an event that hypothetically might have caused death if it would have been more severe)
  - c. Prolongs an existing hospitalization
  - d. Results in persistent or significant disability or incapacity
  - e. Results in a congenital anomaly or birth defect
  - f. Important medical event that requires an intervention to prevent any of a-e above.
- III. <u>Unexpected.</u> AEs that are more severe or prolonged than expected based on the investigator's discretion will be considered Unexpected.

The PILOT trial will monitor, track, and report all Clinical Outcomes and AEs as required by regulatory bodies.

<u>Communication and Reporting of Adverse Events</u>. In order to ensure proper and timely reporting of all adverse events, there will be a clear communication plan for all study personnel to follow. AEs will be recorded in the AE CRF in the electronic database and reported to the PI within 5 days of occurrence. The PI will provide a report of all AEs annually to the IRB and DSMB as part of the annual review process as required. All SAEs will be reported to the PI within 72 hours of occurrence. The PI will, in turn, report all SAEs to the IRB, DSMB, and funding body within 7 calendar days of occurrence.

#### 9.3 Frequency of Monitoring and Interim Analysis.

Study personnel will continuously monitor enrollment, protocol compliance, and AEs and SAEs throughout the course of the trial. Annually, the DSMB will formally review enrollment, protocol compliance, and AEs and SAEs as part of a formal DSMB meeting. Additionally, the DSMB will be available to convene a meeting at any point in the course of the trial to review urgent issues related to AEs, protocol compliance, or unexpected adverse events. Study personnel and DSMB members will adhere to the expectations for reporting and managing AEs and unexpected adverse events outlined in the DSMB charter.

<u>Interim Analysis.</u> In addition to ongoing monitoring of safety throughout the trial, the DSMB will conduct a single interim analysis for efficacy and safety at the

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

anticipated halfway point of the PILOT trial. The interim analysis will include patients enrolled during the first 18 months of the trial. The stopping boundary for efficacy will be met if the P value for the difference between groups is <0.001. Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05). Given the minimal risk nature of the study and current use of all SpO<sub>2</sub> target as a part of usual care, there will be no stopping boundary for futility. The DSMB will reserve the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety.

- **9.4 Data and Safety Monitoring Board (DSMB).** A formal independent DSMB will oversee the conduct of the trial and the planned interim analysis. The DSMB will be composed of at least one physician outside the study institution experienced in the conduct of critical care clinical trials and one biostatistical expert who will assist with study monitoring and performance of the interim analysis.
- **9.5 Data Monitoring Plan**. To ensure data are accurately and completely collected during the PILOT trial, the study team will follow a specific Data Monitoring Plan. All clinical outcomes will be collected in duplicate by both electronic data collection and by the study nurse. All study data from random sample of 10% of study records will be collected in duplicate by electronic data collection and by the study nurse. Each of these records will also be reviewed annually by the primary investigator to ensure data collection is accurate, complete, and current. The study biostatistician will run periodic data cleans throughout the study looking for outliers or overtly erroneous data. This Monitoring Plan will serve as a method for identifying and resolving systematic problems and therefore increase data quality. We will submit progress reports to the local IRB annually, or more frequently if requested.

# 10.0 Study Withdrawal/Discontinuation

Patients can be withdrawn from study participation in the following circumstances:

- The investigator decides that the patient should be withdrawn for safety considerations.
- There is a significant protocol violation in the judgment of the PI.

The reason and date of every withdrawal will be recorded in the patient study records. Follow-up will be performed for all patients who discontinue due to an adverse event or any other safety parameter. Follow-up will also be performed for all patients who end participation in the protocol for another reason, but who also have an adverse event or other safety parameter that could have led to discontinuation. Follow-up will be conducted until the condition has resolved, until diagnosis of the adverse event or

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

safety parameter is deemed chronic and stable, or as long as clinically appropriate. This follow-up will be documented in the patient study record as well.

#### 11.0 Statistical Considerations

<u>Power calculation</u>. In a prior cluster-randomized cluster-crossover trial in the same ICU,<sup>51</sup> 880 mechanically ventilated adults were enrolled per year (73.3 per month), with a median of 22 VFDs [IQR 0-25 VFDs] and an intra-cluster intra-period correlation of 0.01. During the planned 36 month PILOT trial, we estimate 2,640 mechanically ventilated adults will be admitted to the study ICU, of whom 390 will be excluded during washout periods and 2,250 will be enrolled. With a total enrollment of 2,250 patients, a standard deviation in the primary outcome of VFDs of 11.4 days, and a two-sided alpha of 0.05, *the PILOT trial will have 92 percent statistical power to detect an absolute reduction in VFDs of 2.0 days* (similar to the numerical difference in VFDs between SpO<sub>2</sub> target groups reported in prior studies<sup>29,30</sup>).

| Proposed effect modifiers to be included in model | | |
|---|---|---|
| | Lower SpO <sub>2</sub> target<br>better | Higher SpO <sub>2</sub> target<br>better |
| Demographic | | ↑Age |
| Comorbidities | Supplemental $O_2$ , COPD | ↑NYHA stage of CHF,<br>Coronary disease |
| Acute illnesses | Cardiac arrest,<br>Myocardial<br>infarction,<br>ARDS, Pneumonia,<br>Sepsis | Ischemic stroke,<br>Status epilepticus,<br>Acute kidney injury |
| Severity of illness | ↑SOFA score | |
| Vent Settings | $\uparrow$ static compliance,<br>$\downarrow$ PaO <sub>2</sub> /FiO <sub>2</sub> | |
| Lab values | ↑WBC, ↓Platelets,<br>↓Albumin | ↓Hemoglobin,<br>↓Bicarbonate |
| representation in st | modifiers not included in i<br>tudy ICU: Traumatic brain<br>r organ transplant or surgi | injury, Post-operative |
| | tes included in the model:<br>enrollment duration of me | |

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

<u>Primary analysis</u>. The primary analysis will be an intention-to-treat comparison of the number of VFDs experienced by patients in each study group using the Kruskal–Wallis test. Secondary analyses will include [1] intention-to-treat comparisons of the prespecified secondary outcomes between study groups; [2] intention-to-treat comparison of the SpO<sub>2</sub> target groups with regard to ventilator free days using a generalized linear mixed-effects model adjusting for fixed effects (age, sex, race, source of admission, vasopressor receipt, acute diagnosis) and random effects (study period) to account for intra-period correlation, and [3] examination of the differential effects of the intervention for patients with different baseline characteristics (heterogeneity of treatment effect) (see Figure below).

All of secondary analyses will be considered hypothesis-generating, and no corrections for multiple comparisons will be performed. No imputations will be made for missing baseline or on-study laboratory or physiologic data. Continuous variables will be described as mean and standard deviation or median and 25th percentile – 75th percentile or bootstrapped 95% confidence intervals as appropriate. Categorical variables will be given as number and percentage. All between-group comparisons with continuous variables will be performed using Kruskal–Wallis tests; categorical variables will be compared with chi-square testing or Fisher's exact test as appropriate. A complete pre-specified statistical analysis plan will be published prior to the completion of enrollment.

#### **Interim Analysis**

We will plan for the DSMB to conduct a single interim analysis for efficacy and safety at the anticipated halfway point of the trial. The interim analysis will include patients enrolled during the first 18 months of the trial. The stopping boundary for efficacy will be met if the P value for the difference between groups is <0.001. Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05). Given the minimal risk nature of the study and current use of all SpO<sub>2</sub> target as a part of usual care, there will be no stopping boundary for futility. The DSMB will reserve the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety.

## 12.0 Privacy/Confidentiality Issues

At no time during the course of this study, its analysis, or its publication will patient identities be revealed in any manner. The minimum necessary data containing patient or provider identities will be collected. All patients will be assigned a unique study ID number for tracking. Data collected from the medical record will be entered into the secure online database REDCap. Hard copies of the treating clinician

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

modification of SpO<sub>2</sub> target sheet will be stored in a locked room until after the completion of enrollment and data cleaning. Once data are verified and the database is locked, all hard copies of data collection forms will be destroyed. All data will be maintained in the secure online database REDCap until the time of study publication. At the time of publication, a de-identified version of the database will be generated.

# 13.0 Follow-up and Record Retention

Patients will be followed after enrollment for 28 days or until hospital discharge, whichever occurs first. Data collected from the medical record will be entered into the secure online database REDCap. Once data are verified and the database is locked, all hard copies of data collection forms will be destroyed. All data will be maintained in the secure online database REDCap until the time of study publication. At the time of publication, a de-identified version of the database will be generated.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

#### 14.0 References

1. Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med 2010;38(10):1947–53.

- 2. Wunsch H, Angus DC, Harrison DA, Linde-Zwirble WT, Rowan KM. Comparison of medical admissions to intensive care units in the United States and United Kingdom. Am J Respir Crit Care Med 2011;183(12):1666–73.
- 3. Adhikari NKJ, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet Lond Engl 2010;376(9749):1339–46.
- 4. Dasta JF, McLaughlin TP, Mody SH, Piech CT. Daily cost of an intensive care unit day: the contribution of mechanical ventilation. Crit Care Med 2005;33(6):1266–71.
- 5. Halpern NA, Pastores SM. Critical care medicine in the United States 2000-2005: an analysis of bed numbers, occupancy rates, payer mix, and costs. Crit Care Med 2010;38(1):65–71.
- 6. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. The Acute Respiratory Distress Syndrome Network. N Engl J Med 2000;342(18):1301–8.
- 7. Esteban A, Frutos-Vivar F, Muriel A, et al. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med 2013;188(2):220–30.
- 8. Herridge MS, Cheung AM, Tansey CM, et al. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med 2003;348(8):683–93.
- 9. Herridge MS, Tansey CM, Matté A, et al. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med 2011;364(14):1293–304.
- 10. Kahn JM, Benson NM, Appleby D, Carson SS, Iwashyna TJ. Long-term acute care hospital utilization after critical illness. JAMA 2010;303(22):2253–9.
- 11. Pandharipande PP, Girard TD, Jackson JC, et al. Long-term cognitive impairment after critical illness. N Engl J Med 2013;369(14):1306–16.
- 12. Fridovich I. Oxygen toxicity: a radical explanation. J Exp Biol 1998;201(Pt 8):1203–9.
- 13. Heffner JE, Repine JE. Pulmonary strategies of antioxidant defense. Am Rev Respir Dis 1989;140(2):531–54.
- 14. Freeman BA, Crapo JD. Hyperoxia increases oxygen radical production in rat lungs and lung mitochondria. J Biol Chem 1981;256(21):10986–92.
- 15. Waxman AB, Einarsson O, Seres T, et al. Targeted lung expression of interleukin-11 enhances murine tolerance of 100% oxygen and diminishes hyperoxia-induced DNA fragmentation. J Clin Invest 1998;101(9):1970–82.
- 16. Griffith DE, Garcia JG, James HL, Callahan KS, Iriana S, Holiday D. Hyperoxic exposure in humans. Effects of 50 percent oxygen on alveolar macrophage leukotriene B4 synthesis. Chest 1992;101(2):392–7.
- 17. Davis WB, Rennard SI, Bitterman PB, Crystal RG. Pulmonary oxygen toxicity. Early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med 1983;309(15):878–83.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

18. Aggarwal NR, Brower RG. Targeting normoxemia in acute respiratory distress syndrome may cause worse short-term outcomes because of oxygen toxicity. Ann Am Thorac Soc 2014;11(9):1449–53.

- 19. Meade MO, Cook DJ, Guyatt GH, et al. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA J Am Med Assoc 2008;299(6):637–45.
- 20. Eastwood G, Bellomo R, Bailey M, et al. Arterial oxygen tension and mortality in mechanically ventilated patients. Intensive Care Med 2012;38(1):91–8.
- 21. de Jonge E, Peelen L, Keijzers PJ, et al. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care Lond Engl 2008;12(6):R156.
- 22. National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network, Rice TW, Wheeler AP, et al. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA J Am Med Assoc 2012;307(8):795–803.
- 23. Rice TW, Wheeler AP, Thompson BT, et al. Enteral omega-3 fatty acid, gammalinolenic acid, and antioxidant supplementation in acute lung injury. JAMA J Am Med Assoc 2011;306(14):1574–81.
- O'Driscoll BR, Howard LS, Earis J, Mak V, British Thoracic Society Emergency Oxygen Guideline Group, BTS Emergency Oxygen Guideline Development Group. BTS guideline for oxygen use in adults in healthcare and emergency settings. Thorax 2017;72(Suppl 1):ii1-ii90.
- 25. Supplemental Therapeutic Oxygen for Prethreshold Retinopathy Of Prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. Pediatrics 2000;105(2):295–310.
- 26. SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network, Carlo WA, Finer NN, et al. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med 2010;362(21):1959–69.
- 27. Schmidt B, Whyte RK, Asztalos EV, et al. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. JAMA 2013;309(20):2111–20.
- 28. BOOST II United Kingdom Collaborative Group, BOOST II Australia Collaborative Group, BOOST II New Zealand Collaborative Group, et al. Oxygen saturation and outcomes in preterm infants. N Engl J Med 2013;368(22):2094–104.
- 29. Panwar R, Hardie M, Bellomo R, et al. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med 2016;193(1):43–51.
- 30. Girardis M, Busani S, Damiani E, et al. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA 2016;316(15):1583–9.
- 31. Asfar P, Schortgen F, Boisramé-Helms J, et al. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med [Internet] 2017 [cited 2017 Feb 20]; Available from: http://linkinghub.elsevier.com/retrieve/pii/S2213260017300462

Principal Investigators: Matt Semler Version Date: 5/1/2018
Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial Institution/Hospital: Vanderbilt University Medical Center

- 32. Panwar R, Capellier G, Schmutz N, et al. Current oxygenation practice in ventilated patients-an observational cohort study. Anaesth Intensive Care 2013;41(4):505–14.
- 33. Suzuki S, Eastwood GM, Peck L, Glassford NJ, Bellomo R. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care 2013;28(5):647–54.
- 34. Beasley R, Chien J, Douglas J, et al. Thoracic Society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: "Swimming between the flags." Respirol Carlton Vic 2015;20(8):1182–91.
- 35. Severinghaus JW. Simple, accurate equations for human blood O2 dissociation computations. J Appl Physiol 1979;46(3):599–602.
- 36. Stollings JL, Foss JJ, Ely EW, et al. Pharmacist leadership in ICU quality improvement: coordinating spontaneous awakening and breathing trials. Ann Pharmacother 2015;49(8):883–91.
- 37. Girard TD, Kress JP, Fuchs BD, et al. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet Lond Engl 2008;371(9607):126–34.
- 38. Semler MW, Noto MJ, Stollings J, et al. Effect Of Saline Versus Balanced Crystalloids On Major Adverse Kidney Events In The Medical Intensive Care Unit: The Salt Randomized Trial. Am J Respir Crit Care Med 2016;193:A4290.
- 39. Harris BU, Char DS, Feinstein JA, Verma A, Shiboski SC, Ramamoorthy C. Accuracy of Pulse Oximeters Intended for Hypoxemic Pediatric Patients. Pediatr Crit Care Med J Soc Crit Care Med World Fed Pediatr Intensive Crit Care Soc 2016;17(4):315–20.
- 40. Ehrenfeld JM, Funk LM, Van Schalkwyk J, Merry AF, Sandberg WS, Gawande A. The incidence of hypoxemia during surgery: evidence from two institutions. Can J Anaesth J Can Anesth 2010;57(10):888–97.
- 41. Lopez MG, Pretorius M, Shotwell MS, et al. The Risk of Oxygen during Cardiac Surgery (ROCS) trial: study protocol for a randomized clinical trial. Trials 2017;18(1):295.
- 42. Brower RG, Lanken PN, MacIntyre N, et al. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med 2004;351(4):327–36.
- 43. Briel M, Meade M, Mercat A, et al. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA J Am Med Assoc 2010;303(9):865–73.
- 44. Barr J, Fraser GL, Puntillo K, et al. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med 2013;41(1):263–306.
- 45. Gélinas C, Fortier M, Viens C, Fillion L, Puntillo K. Pain assessment and management in critically ill intubated patients: a retrospective study. Am J Crit Care Off Publ Am Assoc Crit-Care Nurses 2004;13(2):126–35.
- 46. Sessler CN, Grap MJ, Brophy GM. Multidisciplinary management of sedation and analgesia in critical care. Semin Respir Crit Care Med 2001;22(2):211–26.

Study Title: Preliminary Investigation of optimal Oxygen Targets (PILOT) trial

Institution/Hospital: Vanderbilt University Medical Center

- 47. Ely EW, Truman B, Shintani A, et al. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA 2003;289(22):2983–91.
- 48. Ely EW, Margolin R, Francis J, et al. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med 2001;29(7):1370–9.
- 49. Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med 1990;113(12):941–8.
- 50. Semler MW, Rice TW, Shaw AD, et al. Identification of Major Adverse Kidney Events Within the Electronic Health Record. J Med Syst 2016;40(7):167.
- 51. for the Isotonic Solutions and Major Adverse Renal Events Trial (SMART) Investigators, the Pragmatic Critical Care Research Group, Semler MW, et al. Balanced crystalloids versus saline in the intensive care unit: study protocol for a cluster-randomized, multiple-crossover trial. Trials [Internet] 2017 [cited 2017 Mar 17];18(1). Available from: http://trialsjournal.biomedcentral.com/articles/10.1186/s13063-017-1871-1
- 52. Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med 1985;13(10):818–29.
- 53. Vincent JL, Moreno R, Takala J, et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med 1996;22(7):707–10.
- 54. Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet Lond Engl 1974;2(7872):81–4.
- 55. Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care 1998;36(1):8–27.
- 56. ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, et al. Acute respiratory distress syndrome: the Berlin Definition. JAMA J Am Med Assoc 2012;307(23):2526–33.
- 57. Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney inter 2012;2(Suppl):1–138.
- 58. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42(2):377–81.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# <u>Pragmatic Investigation of optimal Oxygen Targets</u> (PILOT) trial

### Version 1.5

# **Principal Investigator**

Matthew W. Semler, MD, MSc
Department of Medicine
Division of Allergy, Pulmonary, and Critical Care Medicine
Vanderbilt University School of Medicine

#### **Mentors**

Gordon R. Bernard, MD, Wesley H. Self, MD, MPH, &
Todd W. Rice, MD, MSc
Department of Medicine
Division of Allergy, Pulmonary, and Critical Care Medicine
Vanderbilt University School of Medicine

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# **Table of Contents:**

# Study Schema

- 1.0 Study Summary
- 2.0 Background
- 3.0 Rationale, Aims, and Hypotheses
- 4.0 Study Description
- 5.0 <u>Inclusion/Exclusion Criteria</u>
- 6.0 <u>Enrollment/Randomization</u>
- 7.0 Study Procedures
- 8.0 Risks and Benefits
- 9.0 Adverse Events
- 10.0 <u>Study Withdrawal/Discontinuation</u>
- 11.0 <u>Statistical Considerations</u>
- 12.0 Privacy/Confidentiality Issues
- 13.0 Follow-up and Record Retention
- 14.0 <u>References</u>

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# 1.0 Study Summary

Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) trial

**Background:** Mechanical ventilation of ICU patients universally involves titration of the fraction of inspired oxygen (FiO<sub>2</sub>) to maintain arterial oxygen saturation (SpO<sub>2</sub>). Despite decades of ICU practice, however, the optimal SpO<sub>2</sub> target remains unknown. Higher SpO<sub>2</sub> targets (96-100%) provide a margin of safety against hypoxia but increase exposure to hyperoxia. Lower SpO<sub>2</sub> targets (88-92%) minimize hyperoxia, but may increase the risk of hypoxia. An intermediate SpO<sub>2</sub> target (92-96%) may avoid the risks of both hyperoxia and hypoxia, or may expose patients intermittently to both sets of risks. Current guidelines offer divergent recommendations as to the optimal SpO<sub>2</sub> target and clinical safety and efficacy data are lacking. Therefore, we propose a 2,250-patient cluster-randomized cluster-crossover trial comparing a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%), an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%), and a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%) with regard to the outcome of days alive and free of invasive mechanical ventilation.

#### **Primary Aim:**

 To compare the effect of higher, intermediate, and lower SpO₂ targets on days alive and free of invasive mechanical ventilation among mechanically ventilated critically ill adults.

#### **Primary Hypothesis:**

• Use of a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%) for mechanically ventilated ICU patients will result in more days alive and free of invasive mechanical ventilation than use of an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%) or a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%).

#### **Inclusion Criteria:**

 We will include adults (≥ 18 years old) receiving mechanical ventilation through an endotracheal tube or tracheostomy who are admitted to the study ICU or for whom admission to the study ICU from the emergency department is planned.

#### **Exclusion Criteria:**

• We will exclude patients who are pregnant or who are prisoners.

**Consent:** Because [1] the study enrolls only patients who would have been exposed to oxygen therapy as a part of clinical care outside of the study, [2] all  $SpO_2$  targets examined are currently used in routine care in the study ICU, [3] no high-quality data suggest that the choice of  $SpO_2$  target affects clinical outcomes, and [4] during the trial

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

treating clinicians retain discretion to control the  $SpO_2$  target when felt to be required for the safe treatment a specific patient, we feel the study qualifies as minimal risk. Given the minimal risk, the implementation of  $SpO_2$  targets at an ICU level, and the impracticability of consenting each patient during initiation of mechanical ventilation in the ICU or emergency department, we will request a waiver of informed consent.

**Randomization:** In the PILOT trial, the entire study ICU will be assigned to a single  $SpO_2$  target (cluster-randomized) and the ICU will switch between lower, intermediate, and higher  $SpO_2$  targets every two months in a randomly generated sequence (cluster-crossover).

### **Study Interventions:**

- Lower SpO<sub>2</sub> Target FiO<sub>2</sub> will be titrated to a target SpO<sub>2</sub> of 90% with a goal range of 88-92%.
- Intermediate SpO<sub>2</sub> Target FiO<sub>2</sub> will be titrated to a target SpO<sub>2</sub> of 94% with a goal range of 92-96%.
- **Higher SpO<sub>2</sub> Target** FiO<sub>2</sub> will be titrated accord to a target SpO<sub>2</sub> of 98% with a goal range of 96-100%.

#### **Primary Outcome:**

 Ventilator-free days (VFDs) to study day 28, defined as the number of calendar days alive and free of invasive mechanical ventilation from the final receipt of invasive mechanical ventilation through 28 days after enrollment.

# **Secondary Outcome:**

 28-day in-hospital mortality, defined as death from any cause between enrollment and the first of hospital discharge or 28 days after enrollment.

### **Exploratory Outcomes:**

- Exploratory Clinical Outcomes: ICU mortality, vasopressor-free days, renal replacement therapy-free days, ICU-free days, hospital-free days.
- Exploratory Organ Function Outcomes: daily non-respiratory SOFA score, creatinine, lactate, presence of acute respiratory distress syndrome, Stage II or greater AKI by KDIGO criteria.
- Exploratory Safety Outcomes: Atrial arrhythmia, ventricular arrhythmia, cardiac arrest with return of spontaneous circulation, pneumothorax or pneumomediastinum, ischemic stroke, myocardial infarction

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# 2.0 Background

Each year 2-3 million intensive care unit (ICU) patients receive invasive mechanical ventilation,<sup>1–3</sup> at a cost of more than \$20 billion dollars.<sup>4,5</sup> Despite recent advances,<sup>6</sup> inhospital mortality among mechanically ventilated ICU patients remains 25-35%,<sup>7</sup> and survivors often face cognitive, psychiatric, and physical dysfunction.<sup>8–11</sup>

Mechanical ventilation of ICU patients universally involves titration of the fraction of inspired oxygen (FiO<sub>2</sub>) to maintain arterial oxygen saturation (SpO<sub>2</sub>). Despite decades of ICU practice, however, the optimal SpO<sub>2</sub> target remains unknown. Higher SpO<sub>2</sub> targets (96-100%) provide a margin of safety against hypoxemia, but may increase exposure to excess FiO<sub>2</sub>, hyperoxemia, and tissue hyperoxia, causing oxidative damage, <sup>12-14</sup> inflammation, <sup>15,16</sup> and increased alveolar-capillary permeability. Lower SpO<sub>2</sub> targets (88-92%) minimize hyperoxia, <sup>6,18,19</sup> but may increase the risk of hypoxemia, tissue hypoxia, and organ dysfunction. An intermediate SpO<sub>2</sub> target (92-96%) may avoid the risks of both hyperoxia and hypoxia, or, conversely, may expose patients intermittently to both sets of risks.

Current guidelines offer divergent recommendations – ranging from tolerating  $SpO_2$  values as low as 88% (ARDS Network)<sup>22,23</sup> to pursuing  $SpO_2$  values as high as 98% (British Thoracic Society)<sup>24</sup>. The relative risks and benefits of different  $SpO_2$  targets have been extensively examined in the setting of the neonatal ICU,<sup>25–28</sup> but have only been investigated in adult ICU patients in three small trials.<sup>29–31</sup> Targeting lower  $SpO_2$  resulted in improved survival in one trial and trends toward improved survival in the other two.

In clinical practice, however, hyperoxemia remains common.<sup>32,33</sup> In our recent observational study of 2,200 mechanically ventilated ICU patients at 50 centers across

the United States (see Figure), the majority of patients had a lowest PaO<sub>2</sub> value on the first study day > 100 mm Hg (~SpO<sub>2</sub> > 97%). The wide variation in current practice (frequently favoring higher SpO<sub>2</sub> targets), conflicting guidelines, and pilot trial data favoring lower SpO<sub>2</sub> targets have led to calls for a large, randomized trial to determine the effect of SpO<sub>2</sub> target on patient outcomes.<sup>18</sup>



Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

#### 3.0 Rationale, Aims, and Hypotheses

In order to determine the effect of SpO<sub>2</sub> targets during mechanical ventilation of critically ill adults on clinical outcomes, a randomized trial is needed.

### **Study Aims:**

• **Primary:** To compare the effect of higher, intermediate, and lower SpO<sub>2</sub> targets on days alive and free of invasive mechanical ventilation among mechanically ventilated critically ill adults.

#### • Secondary:

- To evaluate the effect of the same intervention in the same population on the pre-specified Secondary Outcome and on pre-specified Exploratory Clinical Outcomes, Exploratory Organ Function Outcomes, and Exploratory Safety Outcomes.
- To evaluate the effect of the same intervention on days alive and free of invasive mechanical ventilation in clinically relevant pre-specified patient subgroups.

#### **Study Hypotheses:**

- **Primary:** Use of a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%) for mechanically ventilated ICU patients will result in more days alive and free of invasive mechanical ventilation (*Primary Outcome*) than use of an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%) or a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%).
- Secondary: Use of a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%) for mechanically ventilated ICU patients will result in lower 28-day in-hospital mortality (*Secondary Outcome*) than use of an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%) or a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%).

#### 4.0 Study Description

In order to address the aims outlined above, we propose the Pragmatic Investigation of optimal Oxygen Targets (PILOT) trial. The PILOT trial will be a prospective, un-blinded, cluster-randomized, cluster-crossover trial conducted between July 1, 2018 and August 31, 2021 in the medical ICU at Vanderbilt University Medical Center examining the effect of  $SpO_2$  targets on days alive and free of mechanical ventilation among mechanically ventilated ICU patients. For the 36 months of enrollment in the PILOT trial, the entire medical ICU will be assigned to a single  $SpO_2$  target and the ICU will switch between lower, intermediate, and higher  $SpO_2$  targets every two months in a

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

randomly generated sequence (Figure below). Patients who fulfill inclusion criteria without meeting exclusion criteria will be enrolled at the initiation of mechanical ventilation in the study ICU or in the emergency department when admission to the study ICU is planned. The PILOT trial will control only the SpO<sub>2</sub> target and all other aspects of patients' clinical care will remain at the discretion of the treating clinicians.

| Study Year 1 | | | | | | Study Year 2 | | | | | | Study Year 3 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar<br>& Jun | Jul-<br>Aug | Sept-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug |
| | 2018 | | | | 2019 | | | | | 2020 | | | | 2021 | | | |
| High | Mid. | Low | Mid | Low | High | Low | Mid. | High | High | Mid. | Low | Mid. | High | Low | Mid. | High | Low |

The study ICU was randomly assigned to an SpO2 target for each two-month block. The study did not enroll in April and May of 2020 secondary to the COVID-19 pandemic. High = SpO2 target 98% (range 96-100%), Mid. = SpO2 target 94% (range 92-96%), Low = SpO2 target 90% (range 88-92%)

#### 5.0 Inclusion and Exclusion Criteria

#### 5.1 Inclusion Criteria:

- 1. Age ≥ 18 years
- 2. Receiving mechanical ventilation through an endotracheal tube or tracheostomy
- 3. Admitted to the study ICU or admission to the study ICU from the emergency department is planned

#### **5.2** Exclusion Criteria:

- 1. Known pregnancy or beta hCG level greater than the laboratory upper limit of normal in a patient capable of becoming pregnant
- 2. Known to be a prisoner

### 6.0 Enrollment/Randomization

### 6.1 Study Sites:

- Medical Intensive Care Unit at Vanderbilt University Medical Center
- Emergency Department at Vanderbilt University Medical Center
- **6.2 Study Population:** All adults located in the study ICU (or for whom admission to the study ICU from the emergency department is planned) for whom the treating clinicians have decided invasive mechanical ventilation is required will be enrolled unless meeting exclusion criteria. Patients will be included regardless of age, gender, race, weight or body mass index, initial oxygen saturation, or other clinical factors.
- **6.3 Enrollment:** All adult patients who do not meet exclusion criteria will be enrolled immediately upon receipt of invasive mechanical ventilation in the study ICU or in the emergency department when admission to the study ICU is planned.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

#### 6.4 Consent:

All patients receiving invasive mechanical ventilation in an intensive care unit receive oxygen therapy titrated to maintain SpO<sub>2</sub> as a part of routine care. In clinical practice, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adults fall between 88-100%. 32,33 Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: [1] tolerating SpO<sub>2</sub> values as low as 88% (NIH/NHLBI ARDS Network), 22 [2] titrating within the range 92-96% (Thoracic Society of Australia and New Zealand), 34 or [3] pursuing SpO<sub>2</sub> values as high as 98% (British Thoracic Society).<sup>24</sup> The lower SpO<sub>2</sub> target (target 90% and goal range 88-92%), intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%), and higher SpO<sub>2</sub> target (target 98% and goal range 96-100%) examined in this study are all intermittently used in routine care in the study ICU and within the range recommended by at least one international guideline. There are currently no high-quality data to suggest that one SpO<sub>2</sub> target is better than the others with regard to clinical outcomes. Although there are no clear data to support the choice of SpO<sub>2</sub> target, during the PILOT trial, treating clinicians in the study ICU will be allowed to change the SpO<sub>2</sub> target at any point if it is felt to be required for the safe treatment a specific patient.

Because the interventions studied [1] are used as part of routine care in the study ICU, [2] are interventions to which the patient would be exposed even if not participating in the study, [3] have no prior data to suggest the superiority of one approach over the other, and [4] are equivalent options from the perspective of the treating clinicians (otherwise the treating clinician retains control of  $SpO_2$  target), we feel the study presents minimal risk.

Additionally, obtaining informed consent prior to participation in the study would be impractical. Endotracheal intubation and initiation of mechanical ventilation for critically ill patients is frequently a time-sensitive procedure. Despite the availability of a formal informed consent document for the endotracheal intubation and initiation of mechanical ventilation, time allows discussion of risks and benefits in less than 10% of airway management events in the study ICU. The oxygen titration protocol used to target SpO<sub>2</sub> in this trial begins immediately at the initiation of mechanical ventilation to capture the period of mechanical ventilation with the highest risk for hyperoxia and hypoxia. Moreover, in this cluster-randomized trial, the entire ICU is assigned to a single SpO<sub>2</sub> target delivered by the unit's respiratory therapists through a unit-wide oxygen titration protocol. Obtaining informed consent from every eligible patient in the ICU each day would be logistically infeasible and patients who declined to participate would need to be transferred between ICUs which might adversely impact their care.

Because the study presents minimal risk, would not adversely affect the welfare or privacy rights of the participant, and consent would be impracticable, we will request a waiver of informed consent.

### 6.5 Information for Patients, Families, or Surrogates about the Study:
Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

Although the study will be conducted with waiver of informed consent, we will implement a process by which patients, families, or surrogates may be made aware of the study and receive investigators' contact information in order to solicit additional information about the study, ask questions, or express concerns. An information sheet providing an IRB-approved lay language summary of the study activities and containing the contact information for investigators (who will remain available throughout the study period to provide additional information to patients and families upon request) will be made available in the following manner:

- 1. Throughout the study period, the information sheet will be posted in at least two glass display cases, one near the public entrance to the medical ICU and one near the mid-point of the medical ICU.
- 2. Throughout the study period, the information sheet will be included in the welcome packet of information about the medical ICU, which is distributed at the time of ICU admission to available families or surrogates by the medical receptionist or charge nurse as a part of routine clinical care.
- 3. Throughout the study period, copies of the information sheet will be available in a brochure holder on the display table in the medical ICU family waiting room.
- 4. Throughout the study period, additional copies of the information sheet will be available in the physician and respiratory therapy offices to be provided to patients, families, or surrogates with questions or concerns about the study.

Unlike an informed consent document, the information sheet will not be distributed by research personnel directly to participants but will be made generally available in the study setting to patients, families, and surrogates. There may be patients in the study who do not receive information about the study (e.g., a patient without family or surrogate who is admitted to the ICU with coma). There may be patients who are not in the study who do receive information about the study (e.g., a patient admitted to the medical ICU on high-flow nasal cannula who does not require invasive mechanical ventilation).

In order to ensure and record the execution of the above approach to providing information about the study, the primary investigator will:

1. Throughout the study period, audit in-person at least every fourteen (14) days to confirm that the most recent IRB-approved information sheet is posted in at least two glass display cases in the medical ICU. At least twice a year take a photograph of the most recent IRB-approved information sheet in one of the glass display cases in the medical ICU. Store the photographs with the date and time that they were taken electronically in the study files and in hard copy in the study binder.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

2. Throughout the study period, audit in-person at least every fourteen (14) days to confirm that copies of the most recent IRB-approved information sheet are available in a brochure holder on the display table in the medical ICU family waiting room. At least twice a year, take a photograph of the most recent IRB-approved information sheets in a brochure holder on the display table in the medical ICU family waiting room. Store the photographs with the date and time that they were taken electronically in the study files and in hard copy in the study binder.

- 3. Throughout the study period, audit in-person at least every fourteen (14) days to confirm that additional copies of the information sheet are available in the physician and respiratory therapy offices to be provided to patients, families, or surrogates with questions or concerns about the study.
- 4. Record and complete a case report form in the study database detailing contact about the study between patients, families, and surrogates and study personnel.

#### 6.6 Randomization:

During each two-month block of the study, the ICU will be assigned to either a higher  $SpO_2$  target (target 98% and goal range 96-100%), an intermediate  $SpO_2$  target (target 94% and goal range 92-96%), or a lower  $SpO_2$  target (target 90% and goal range 88-92%). The order of study group assignments will be generated by computerized randomization using permuted blocks of 3 to minimize the impact of seasonal variation. The last 7 days of each two-month block will be a washout period during which the ICU will continue to target the assigned  $SpO_2$  but new patients will not be included in the primary analysis. Assuming a duration of mechanical ventilation similar to that observed for mechanically ventilated patients admitted to the study ICU in a prior year (median 3 [IQR 3-5] days), a 7-day washout period will ensure that 98% patients do not experience a "crossover" from one assigned  $SpO_2$  target to another.

#### 7.0 Study Procedures

#### 7.1 Study Interventions

**Choice of SpO<sub>2</sub> targets:** In clinical practice, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adults fall between 88-100%.<sup>32,33</sup> Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: [1] tolerating SpO<sub>2</sub> values as low as 88% (NIH/NHLBI ARDS Network),<sup>22</sup> [2] titrating within the range 92-96% (Thoracic Society of Australia and New Zealand),<sup>34</sup> or

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

[3] pursuing SpO<sub>2</sub> values as high as 98% (British Thoracic Society).<sup>24</sup> The PILOT trial will have three study groups, each emulating an approach to SpO<sub>2</sub> targets represented in guidelines and clinical practice (Table).

| Study Group | SpO <sub>2</sub> target | SpO <sub>2</sub> range | PaO <sub>2</sub> target | PaO <sub>2</sub> range |
|---|---|---|---|---|
| Lower SpO <sub>2</sub> target | 90% | 88-92% | 60 mm Hg | 55-65 mm Hg |
| Intermediate SpO <sub>2</sub> target | 94% | 92-96% | 70 mm Hg | 65-80 mm Hg |
| Higher SpO <sub>2</sub> target | 98% | 96-100% | 110 mm Hg | > 80 mm Hg |

The  $SpO_2$  target and range of  $SpO_2$  values considered to be compliant are displayed for each study group.  $PaO_2$  will be used to guide oxygen titration for participants without functioning pulse oximetry monitoring.

**SpO<sub>2</sub> versus PaO<sub>2</sub>:** SpO<sub>2</sub> is measured continuously via non-invasive pulse oximetry for nearly all mechanically ventilated ICU patients. In contrast, PaO<sub>2</sub> is assessed via arterial puncture intermittently and selectively, particularly among more severely ill patients earlier in their clinical course. Similar to prior studies of oxygen therapy during mechanical ventilation<sup>29</sup>, the PILOT trial will target ranges of SpO<sub>2</sub> for all patients with functioning non-invasive pulse oximetry monitoring. For patients in the PILOT trial for whom non-invasive pulse oximetry monitoring is unavailable (e.g., inadequate plethysmography signal due to hypoperfusion), PaO<sub>2</sub> values corresponding to the assigned SpO<sub>2</sub> target will be used to guide oxygen therapy (see above Table).<sup>35</sup>

**Oxygen Titration:** In the study ED and ICU, and in the United States generally, titration of FiO<sub>2</sub> to maintain SpO<sub>2</sub> for mechanically ventilated adults is most commonly performed by respiratory therapists, with input from nurses and physicians. Other aspects of mechanical ventilation (selection of tidal volume, titration of positive end-expiratory pressure, screening for spontaneous breathing trials) are governed by respiratory therapy protocols jointly developed by respiratory therapy and physician leaders. In preparation for the PILOT trial, we collaborated with respiratory therapy leaders in the study ED and ICU to adapt existing ventilator management protocols to provide guidance for respiratory therapists in titrating FiO<sub>2</sub> to achieve each of the three study SpO<sub>2</sub> targets.

<u>Initiation of Mechanical Ventilation:</u> The study protocol guides respiratory therapists and treating clinicians to begin titrating  $FiO_2$  to the target  $SpO_2$  value within 15 minutes of the initiation of mechanical ventilation in the participating ED or ICU. This initial 15-minute window is intended to give the treating clinicians adequate time after emergent tracheal intubation to stabilize the patient's hemodynamics and initiate basic ventilator settings, but also to intervene early enough to control the  $FiO_2$  and  $SpO_2$  during the

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

critical early period of mechanical ventilation when exposure to excess FiO<sub>2</sub> and hyperoxemia is most common.

Oxygen Titration during Mechanical Ventilation: SpO<sub>2</sub> will be assessed by continuous pulse oximetry. The respiratory therapist managing the patient's ventilator will target an SpO<sub>2</sub> value of 98% in the higher SpO<sub>2</sub> group, 94% in the intermediate SpO<sub>2</sub> group, and 90% in the lower SpO<sub>2</sub> group. The respiratory therapist will titrate FiO<sub>2</sub> as directed by the oxygen titration protocol when SpO<sub>2</sub> values are outside of the range 96-100% in the higher SpO<sub>2</sub> group, 92-96% in the intermediate SpO<sub>2</sub> group, and 88-92% in the lower SpO<sub>2</sub> group. Respiratory therapists and other treating clinicians may also titrate FiO<sub>2</sub> when SpO<sub>2</sub> values are not outside the range considered to be at goal in order to achieve SpO<sub>2</sub> values closer to the assigned SpO<sub>2</sub> target, to facilitate weaning from mechanical ventilation, or for other clinical reasons. SpO<sub>2</sub> will be reassessed 5 minutes after each change in FiO<sub>2</sub> or sooner if clinically indicated. Study protocol determines the SpO<sub>2</sub> target from enrollment until the first of: (1) extubation from invasive mechanical ventilation, (2) transfer out of a participating study location, (3) completion of an SpO<sub>2</sub> target modification sheet by treating clinicians, or (4) end of the two-month study period. Study protocol does not determine the SpO<sub>2</sub> target during time-periods in which the patient is not physically located in a study location (e.g., during transport) or when  $FiO_2$  is not being titrated to achieve an  $SpO_2$  target (e.g., when an  $FiO_2$  of 1.0 is being administered for a procedure).

Liberation from Mechanical Ventilation: Each day of mechanical ventilation, all patients in the study ICU are assessed for safety of a spontaneous awakening trial (SAT) and spontaneous breathing trial (SBT)<sup>36</sup> using the SAT and SBT safety criteria from the Awakening and Breathing Controlled trial.<sup>37</sup> To prevent patients in the higher SpO<sub>2</sub> target group from experiencing delays in qualifying for an SBT based on receipt of higher FiO<sub>2</sub> to achieve the higher SpO<sub>2</sub> target, during the PILOT trial we will allow patients in all groups to qualify for an SAT and SBT regardless of their current FiO<sub>2</sub> or PEEP settings, as long as the other SAT and SBT Safety Screen criteria are met and treating clinicians feel performance of an SAT and SBT is safe. Definitions of SAT and SBT failure and the ventilator settings and duration of the SBT will not be changed from those used in the ABC trial and during usual care in the study ICU. For patients who have passed an SAT and SBT, the decision to discontinue invasive mechanical ventilation will be made by the treating clinicians.

**Modification of SpO<sub>2</sub> Targets:** At any time during the course of the study, if a treating clinician or a patient, family member, or surrogate feels an  $SpO_2$  target other than that assigned by the study is required for the safe treatment of a specific patient, the  $SpO_2$  target for that patient may be modified. To modify the target, the supervising physician will complete a one-page  $SpO_2$  target modification sheet documenting the rationale for modifying the target. Details of each  $SpO_2$  target modification will be collected and

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

monitored. In our prior cluster-crossover trial using the same approach to modification of therapy assignment, treating clinicians exercised the ability to modify the assigned therapy for < 5% of patients.<sup>38</sup>

Anticipated examples of conditions for which treating clinicians may elect to override the assigned SpO<sub>2</sub> target include:

- pneumothorax
- pneumomediastinum
- carbon monoxide poisoning
- decompression sickness
- bleomycin toxicity
- paraquat toxicity

SpO<sub>2</sub> Monitoring: For all mechanically ventilated patients in the study ICU, SpO<sub>2</sub> is continuously monitored using Nellcor™ SpO<sub>2</sub> Adhesive Sensors (Medtronic, Minneapolis, MN), which measure changes in red and infrared light absorption in an arteriolar bed throughout the pulse cycle to report a non-normalized real-time plethysmographic waveform and arterial hemoglobin saturation values averaged over the prior 6 seconds with a mean difference between SpO<sub>2</sub> and SaO<sub>2</sub> < 2% for SpO<sub>2</sub> values 80-100%.<sup>39</sup> Plethysmography and SpO<sub>2</sub> values are displayed [1] on IntelliVue MP90 bedside patient monitors (PHILIPS, Amsterdam, Netherlands) in each ICU room, [2] on telemetry monitors located at ICU nursing stations and adjacent to the respiratory therapy office, and [3] in real-time in the institutional EHR, available from any physical location. SpO<sub>2</sub> values are archived every 60 seconds into an intuitional data warehouse.<sup>40,41</sup> Collecting SpO<sub>2</sub> values every 60 seconds will allow the PILOT trial report with far greater accuracy the incidence, severity, and duration of desaturation than prior trials in which SpO<sub>2</sub> values were collected every 4-24 hours.<sup>29,30</sup>

**Feedback on SpO<sub>2</sub> Target Adherence:** [1] During the study, the IntelliVue MP90 bedside patient monitors in each room will be set to generate an alarm for SpO<sub>2</sub> values outside the range considered to be at goal for the assigned SpO<sub>2</sub> target group. For example, for patients in the intermediate SpO<sub>2</sub> target group, SpO<sub>2</sub> values 92-96% generate no alarm, whereas SpO<sub>2</sub> values ≤ 91% or ≥ 97% generate an alarm alerting nursing staff and respiratory therapy to the out-of-range value. [2] Study personnel will remotely monitor SpO<sub>2</sub> values every four hours from 4 AM through 10 PM Monday through Friday and during a 10% sample of night and weekend hours to identify instances of lag between out of range SpO<sub>2</sub> values and FiO<sub>2</sub> titration, provide feedback and reinforcement to bedside nurses and respiratory therapists, and identify any barriers to SpO<sub>2</sub> target compliance. [3] Study personnel will attend respiratory therapy group meetings, nursing unit board meetings, and ICU physician leadership meetings to educate staff about the study, solicit safety concerns and adverse events, and identify and address barriers to SpO<sub>2</sub> target compliance. This approach to daily monitoring and

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

intermittent feedback to clinical personnel successfully achieved 95% compliance with the assigned intervention in a prior cluster-crossover trial in the same ICU.<sup>38</sup>

**Co-interventions:** Institutional protocols in the study setting will ensure that mechanically ventilated patients in PILOT receive: [1] ventilation targeting 6 mL/kg of predicted body weight and plateau pressure  $\leq$  30 cm H<sub>2</sub>O,<sup>6</sup> [2] PEEP titration according to the ARDSNet Lower PEEP/higher FiO<sub>2</sub> table (except for patients with severe ARDS, for whom the Higher PEEP/lower FiO<sub>2</sub> table is applied),<sup>42,43</sup> [3] management of pain, agitation, and delirium<sup>44</sup> targeting Critical Care Pain Observation Tool (CPOT),<sup>45</sup> Richmond Agitation-Sedation Scale (RASS),<sup>46,47</sup> and Confusion Assessment Method for the ICU (CAM-ICU) scores,<sup>48,49</sup> and [4] daily spontaneous awakening trials (SAT) and spontaneous breathing trials (SBT).<sup>36,37</sup>

- **7.2 Blinding:** Similar to prior  $SpO_2$  target studies among critically ill adults<sup>29,30</sup>, patients and clinicians will not be blinded to study group assignment. Observer bias will be minimized by use of objective endpoints collected *in duplicate* by [1] study personnel blinded to group assignment and [2] automated data extraction from the EHR (see *Data Collection* below).
- **7.3 Data Collection:** The PILOT trial will primarily use structured data collected in routine clinical care, exported daily from the institution's EHR into an Enterprise Data Warehouse, along with data from the patient registration, billing, and laboratory clinical information systems. We have previously validated the quality of this method of data collection against the reference standard of two-physician manual chart review, <sup>50</sup> and the planned approach to electronic dataset generation for the PILOT trial has already been successfully employed for the conduct of three prior pragmatic trials. <sup>38,38,51</sup>

#### **Electronically extracted data elements will include:**

<u>Enrollment (Day 0)</u>: age; sex; race; ethnicity; height, weight; APACHE II score;<sup>52</sup> non-respiratory SOFA score;<sup>53</sup> Glasgow Coma Scale score;<sup>54</sup> Elixhauser Comorbidity Index;<sup>55</sup> history of present illness; vital signs (temperature, heart rate, systolic blood pressure, diastolic blood pressure, SpO<sub>2</sub>); mechanical ventilator settings (mode, set and exhaled tidal volume, set and actual respiratory rate, positive end-expiratory pressure, peak pressure, FiO<sub>2</sub>); serum laboratory values (white blood cell count, hemoglobin, platelet count, sodium, potassium, bicarbonate, creatinine, bilirubin, alanine aminotransferase, aspartate aminotransferase, lactate, arterial pH, PaO<sub>2</sub>, SaO<sub>2</sub>).

<u>Daily On-Study (Days 0-28):</u> Vital signs, ventilator settings, screening for and performance of spontaneous awakening trials and spontaneous breathing trials, and serum laboratory values (as above); receipt of red cell transfusion; number of arterial blood gases; non-respiratory SOFA score; ARDS by Berlin criteria; 56 Stage II or greater

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

AKI by KDIGO criteria;<sup>57</sup> atrial arrhythmia, ventricular arrhythmia, cardiac arrest, pneumothorax or pneumomediastinum, ischemic stroke, myocardial infarction.

<u>Termination (Days 0-28):</u> Vital status at 28 days; time of liberation from invasive mechanical ventilation; receipt and duration of vasopressors; receipt and duration of renal replacement therapy; duration of ICU and hospital admission.



Data elements collected manually by study personnel will include: [1] all data elements for a randomly selected 10% of participants to ensure the quality of electronically extracted data, [2] all primary and secondary outcomes collected at study termination for 100% of participants to ensure duplicate data collection of key study outcomes, and [3] any data elements for which electronic data extraction has not been developed and validated, including etiology of respiratory failure, indication for mechanical ventilation, protocol violations, and adverse events. Data will be stored, curated, and secured in the online database, REDCap.<sup>58</sup>

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

#### 7.4 Outcome Measures

# **Primary Outcome:**

The primary outcome is ventilator-free days (VFDs) to study day 28. VFDs will be defined as the number of calendar days alive and free of invasive mechanical ventilation from the final receipt of invasive mechanical ventilation through 28 days after enrollment. For the assessment of VFDs, the day of enrollment (defined as the day on which the patient first receives invasive mechanical ventilation in a participating study location), will be considered to be day 0. Outcome ascertainment will cease at the time of hospital discharge or 28 days after enrollment, whichever occurs first. Receipt of invasive mechanical ventilation will be considered to end when patients undergo the final tracheal extubation or disconnection of the ventilator from the endotracheal tube or tracheostomy tube between enrollment and 28 days after enrollment. Patients who continue to receive invasive mechanical ventilation at day 28 will receive zero VFDs. Patient who die prior to day 28 will receive zero VFDs. Patients who are discharged from the hospital prior to day 28 and are receiving invasive mechanical ventilation at the time of discharge will receive zero VFDs. Patients who are removed from invasive mechanical ventilation and are discharged from the hospital without invasive mechanical ventilation prior to 28 days will be assumed to remain free of invasive mechanical ventilation between hospital discharge and day 28. For patients who are removed from invasive mechanical ventilation, return to invasive mechanical ventilation, and are subsequently removed again from invasive mechanical ventilation prior to day 28, VFDs will be counted from the final receipt of invasive mechanical ventilation prior to day 28. We chose VFDs as the primary outcome for the PILOT trial as choice of SpO<sub>2</sub> target may simultaneously affect both mortality and duration of invasive mechanical ventilation.

#### **Secondary Outcome:**

The sole pre-specified secondary outcome is 28-day in-hospital mortality, defined as death from any cause between enrollment and the first of hospital discharge or 28 days after enrollment.

# **Exploratory Clinical Outcomes:**

- 1. ICU mortality
- 2. Vasopressor-free days
- 3. Renal replacement therapy-free days
- 4. ICU-free days
- 5. Hospital-free days

**Exploratory Organ Function Outcomes:** (All exploratory organ function outcomes will employ only laboratory values and imaging obtained as a part of routine clinical care)

1. Daily non-respiratory SOFA score

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

- 2. Daily creatinine
- 3. Daily lactate
- 4. Presence of acute respiratory distress syndrome
- 5. Stage II or greater AKI by KDIGO criteria

# **Exploratory Safety Outcomes:**

- 1. Atrial arrhythmia
- 2. Ventricular arrhythmia
- 3. Cardiac arrest
- 4. Pneumothorax or pneumomediastinum
- 5. Ischemic stroke
- 6. Myocardial infarction

# Measures of Separation between Groups:

- 1. SpO<sub>2</sub>
- 2. SaO<sub>2</sub>
- 3. FiO<sub>2</sub>
- 4. PaO<sub>2</sub>
- 5. Episodes of hypoxemia, including:
  - a.  $SpO_2 < 85\%$  for  $\geq 5$  minutes
  - b.  $SpO_2 < 80\%$  for  $\geq 5$  minutes
  - c.  $SpO_2 < 70\%$  for  $\ge 2$  minutes
- 6. Episodes of hyperoxemia, including:
  - a.  $SpO_2 > 98\%$  for  $\geq 5$  minutes
  - b.  $SpO_2 > 98\%$  for  $\ge 30$  minutes
- 7. Proportion of patients with a value for PaO2 < 55 mm Hg
- 8. Proportion of patients with a value for PaO2 > 120 mm Hg

# **Exploratory Processes of Care Outcomes:**

- 1. Tidal volume
- 2. Positive end expiratory pressure
- 3. Peak airway pressure
- 4. Receipt of mandatory ventilator mode
- 5. Number of arterial blood gasses
- 6. Hemoglobin
- 7. Red cell transfusion

#### 8.0 Risks and Benefits:

Among adult patients for whom the treating clinicians have decided invasive mechanical ventilation is required, there are currently no established risks or benefits to targeting a higher, intermediate, or lower SpO<sub>2</sub>. At this time, there is no reason to

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

believe that participation in this study would expose patients to greater medical risks or benefits than those experienced by critically ill patients receiving invasive mechanical ventilation as a part of routine care. The greater benefit of the study would be to society in the form of improved understanding of safe and effective provision of oxygen therapy during mechanical ventilation for critically ill patients.

A potential risk to patients participating in this study involves the collection of protected health information (PHI). In order to limit the associated risks, the minimum amount of PHI necessary for study conduct will be collected. After collection, the data will be stored in a secure online database (REDCap) only accessible by the investigators. After publication, a de-identified database will be generated to protect participant privacy.

# 9.0 Safety Monitoring and Adverse Events:

# 9.1 Safety Monitoring

The PILOT trial will take place in a high-acuity clinical care environment during delivery of a high-acuity procedure required for routine clinical care. During the time of the study intervention, the patient will have a critical care or emergency medicine nurse with a low patient-to-nurse staffing ratio, immediate access to a respiratory therapist, and a team of critical care physicians physically located on the study unit twenty-four hours a day. As a part of routine care all patients will be receiving continuous invasive or non-invasive monitoring of heart rate, blood pressure, respiratory rate, and oxygen saturation.

Study personnel will monitor compliance with the study inclusion and exclusion criteria, study protocol, and study safety measures daily. Study personnel will be readily available to answer questions at any time from patients, legally authorized representatives, or treating clinicians. If, at any point in a patient's clinical course, the treating clinicians believe an  $SpO_2$  target different from the assigned target is required for the safe treatment of the patient, the  $SpO_2$  target will be modified to the target the treating clinicians judge to be safest.

A structured plan for prospective collection of study outcomes has been specified, in addition to a process by which Adverse Events and Serious Adverse Events will be managed and reported as required to regulatory bodies.

A Data and Safety Monitoring Board (DSMB) will be appointed to oversee the study. The DSMB will be available throughout the trial to monitor enrollment, protocol compliance, safety, and adverse events. Additionally the DSMB will perform an interim analysis for safety and efficacy.

#### 9.2 Adverse Event Reporting

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

A system has been established to report and track clinical outcomes and adverse events (AEs). Study personnel will monitor the safety of subjects and follow AEs until the event resolves or is explained.

Clinical Outcomes (not considered Adverse Events). In this study of critically ill patients who are at high risk for death or other adverse outcomes due to their underlying critical illness, clinical outcomes, including death and organ dysfunction, will be systematically tracked (collected in the case report form) and will be included as part of the analyses for this study. For the purposes of reporting, death and organ dysfunction will not be recorded as AEs unless the investigator believes the event may have been caused by the study or is more severe or prolonged than expected given the underlying critical illness. This approach—considering death and organ dysfunction as outcomes rather than AEs and systemically tracking expected outcomes for analysis rather than solely recording individual AEs—is common in ICU trials because these outcomes/events occur commonly in the ICU and this system mandates that data regarding death, organ dysfunction, and expected outcomes be tracked systematically for all patients and analyzed appropriately. Clinical outcomes will be systemically tracked throughout the study period. Listed below are events that will be tracked as primary, secondary, or exploratory clinical outcomes and will not therefore be reported as AEs during this study (unless believed to be study related and more severe or prolonged than expected given the underlying critical illness):

- 1. Death (all deaths occurring prior to hospital discharge will be reported on the CRF in the vital status at hospital discharge section);
- 2. Recurrence of respiratory failure, including need for re-intubation or non-invasive mechanical ventilation, presence of acute respiratory distress syndrome, or presence of pneumothorax or pneumomediastinum;
- 3. Circulatory failure, including cardiac arrest or shock with or without receipt of vasopressors;
- 4. Incidence of sustained atrial and ventricular arrhythmias;
- 5. Acute kidney injury, including leading to increased creatinine or receipt of renal replacement therapy;
- 6. Hepatic injury or failure leading to increased bilirubin, AST, or ALT;
- 7. Coagulation derangements leading to elevated PT/INR or PTT, DIC, thrombocytopenia, or thrombocytosis;
- 8. Lactic acidosis;
- 9. Delirium, disability, and physical or cognitive impairment believed to be newly acquired;
- 10. All values for SpO<sub>2</sub>, SaO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, or PaO<sub>2</sub>/FiO<sub>2</sub> ratio;
- 11. All values for vital signs (e.g., temperature, respiratory rate, SpO<sub>2</sub>);
- 12. Receipt of co-interventions (e.g., number of arterial blood gasses, red cell transfusion)

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

13. Duration of ICU admission, ICU readmission;

- 14. Duration of hospitalization, hospital readmission;
- 15. Alterations in routine labs, including chemistries, complete blood counts, liver function tests, and hemostasis profiles.

Adverse Event Classifications. An Adverse Event (AE) will be any untoward medical occurrence for a patient enrolled in the trial that is not tracked as a clinical outcome, regardless of whether the event is considered study related or not. All AEs occurring during the observational study period will be recorded on the CRF. All AEs will then be assessed as to whether they are (1) related to study procedures, (2) serious, and/or (3) unexpected according to the following definitions:

- Related to study procedures. AEs that the investigator suspects are related to the study will be classified as study related. Certainty of relatedness is not required as long as a reasonable possibility exists that the AE is related to a study procedure.
- II. <u>Serious.</u> AEs that meet any of the criteria below will be considered Serious Adverse Events (SAEs):
  - a. Results in death
  - b. Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event and NOT an event that hypothetically might have caused death if it would have been more severe)
  - c. Prolongs an existing hospitalization
  - d. Results in persistent or significant disability or incapacity
  - e. Results in a congenital anomaly or birth defect
  - f. Important medical event that requires an intervention to prevent any of a-e above.
- III. <u>Unexpected.</u> AEs that are more severe or prolonged than expected based on the investigator's discretion will be considered Unexpected.

The PILOT trial will monitor, track, and report all Clinical Outcomes and AEs as required by regulatory bodies.

<u>Communication and Reporting of Adverse Events</u>. In order to ensure proper and timely reporting of all adverse events, there will be a clear communication plan for all study personnel to follow. AEs will be recorded in the AE CRF in the electronic database and reported to the PI within 5 days of occurrence. The PI will provide a report of all AEs annually to the IRB and DSMB as part of the annual review process as required. All SAEs will be reported to the PI within 72 hours of occurrence. The PI will, in turn, report all SAEs to the IRB, DSMB, and funding body within 7 calendar days of occurrence.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# 9.3 Frequency of Monitoring and Interim Analysis.

Study personnel will continuously monitor enrollment, protocol compliance, and AEs and SAEs throughout the course of the trial. Semi-annually, the DSMB will formally review enrollment, protocol compliance, and AEs and SAEs as part of a formal DSMB meeting. Additionally, the DSMB will be available to convene a meeting at any point in the course of the trial to review urgent issues related to AEs, protocol compliance, or unexpected adverse events. Study personnel and DSMB members will adhere to the expectations for reporting and managing AEs and unexpected adverse events outlined in the DSMB charter.

Interim Analysis. In addition to ongoing monitoring of safety throughout the trial, the DSMB will conduct a single interim analysis for efficacy and safety at the anticipated halfway point of the PILOT trial. The interim analysis will include patients enrolled during the first 18 months of the trial. The stopping boundary for efficacy will be met if the P value for the difference between groups is <0.001. Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05). Given the minimal risk nature of the study and current use of all SpO<sub>2</sub> target as a part of usual care, there will be no stopping boundary for futility. The DSMB will reserve the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety.

- **9.4 Data and Safety Monitoring Board (DSMB).** A formal independent DSMB will oversee the conduct of the trial and the planned interim analysis. The DSMB will be composed of at least one physician outside the study institution experienced in the conduct of critical care clinical trials and one biostatistical expert who will assist with study monitoring and performance of the interim analysis.
- **9.5 Data Monitoring Plan**. To ensure data are accurately and completely collected during the PILOT trial, the study team will follow a specific Data Monitoring Plan. All clinical outcomes will be collected in duplicate by both electronic data collection and by the study nurse. All study data from random sample of 10% of study records will be collected in duplicate by electronic data collection and by the study nurse. Each of these records will also be reviewed annually by the primary investigator to ensure data collection is accurate, complete, and current. The study biostatistician will run periodic data cleans throughout the study looking for outliers or overtly erroneous data. This Monitoring Plan will serve as a method for identifying and resolving systematic problems and therefore increase data quality. We will submit progress reports to the local IRB annually, or more frequently if requested.

# 10.0 Study Withdrawal/Discontinuation

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

Patients can be withdrawn from study participation in the following circumstances:

 The investigator decides that the patient should be withdrawn for safety considerations.

• There is a significant protocol violation in the judgment of the PI.

The reason and date of every withdrawal will be recorded in the patient study records. Follow-up will be performed for all patients who discontinue due to an adverse event or any other safety parameter. Follow-up will also be performed for all patients who end participation in the protocol for another reason, but who also have an adverse event or other safety parameter that could have led to discontinuation. Follow-up will be conducted until the condition has resolved, until diagnosis of the adverse event or safety parameter is deemed chronic and stable, or as long as clinically appropriate. This follow-up will be documented in the patient study record as well.

#### 11.0 Statistical Considerations

# Power calculation.

In a prior cluster-randomized cluster-crossover trial in the same ICU,<sup>51</sup> 880 mechanically ventilated adults were enrolled per year (73.3 per month), with a median of 22 VFDs [IQR 0-25 VFDs] and an intra-cluster intra-period correlation of 0.01. During the planned 36-month PILOT trial, we estimate 2,640 mechanically ventilated adults will be admitted to the study ICU, of whom 390 will be enrolled during washout periods and excluded from the primary analysis and 2,250 will be included in the primary analysis. With a total enrollment of 2,250 patients, a standard deviation in the primary outcome of VFDs of 11.4 days, and a two-sided alpha of 0.05, *the PILOT trial will have 92 percent statistical power to detect an absolute difference between groups in VFDs of 2.0 days* (similar to the numerical difference in VFDs between SpO<sub>2</sub> target groups reported in prior studies<sup>29,30</sup>).

#### <u>Primary analysis of the Primary Outcome</u>.

The primary analysis will be an intention-to-treat comparison of the primary outcome of VFDs between the higher, intermediate, and lower SpO2 target groups among all patients enrolled in the trial except [1] those admitted during one of the 7-day washout periods and [2] those with a laboratory-confirmed diagnosis of Coronavirus disease 2019 (COVID-19). We will use a proportional odds model with independent covariates of group assignment (higher, intermediate, or lower SpO2 target) and time. Time (in days) will be treated as a continuous variable with values ranging from 1 (first day of enrollment) to 1,097 (final day of enrollment) and will be analyzed using restricted cubic splines with multiple knots to allow for non-linearity resulting from seasonality or secular trends. For the purposes of declaring a statistically significant

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

difference between groups in the primary endpoint, we will consider the conditional effect from the proportional odds model and a two-sided P value of 0.05. In addition to the overall comparison of the three study groups, we will perform pair-wise comparisons between the lower and intermediate groups, lower and higher groups, and intermediate and higher groups using the same statistical approach.

# Sensitivity Analyses of the Primary Outcome

- We will repeat the primary analysis using alternative statistical approaches to comparing the VFDs outcome between groups. These statistical approaches will include:
  - o zero-inflated Poisson regression;
  - o zero-inflated negative binomial regression;
  - o global rank scale analysis (see Supplementary Appendix); and
  - Fine and Gray competing risk regression in which extubation from invasive mechanical ventilation is the event of interest and mortality is a competing event.
- We will repeat the primary analysis with adjustment for pre-specified baseline covariates.
- We will repeat the primary analysis replacing the continuous covariate of time with a categorical covariate of season defined as: winter (January, February, March); spring (April, May, June); summer (July, August, September); and fall (October, November, December).
- We will repeat the primary analysis among all patients enrolled in the trial, including [1] patients initiated on invasive mechanical ventilation in a study location during one of the pre-specified 7-day washout periods and [2] patients with a diagnosis of COVID-19 (estimated sample size of 3,000 patients).

# Analysis of Effect Modification for the Primary Outcome.

We will examine whether pre-specified baseline variables modify the effect of study group on the primary outcome using formal tests of statistical interaction in a proportional odds model. Independent variables will include study group assignment, the potential effect modifier of interest, and the interaction between the two (e.g., study group \* presence of sepsis or septic shock) and time. Significance will be determined by the P value for the interaction term, with values less than 0.10 considered to suggest a potential interaction and values less than 0.05 considered to confirm an interaction.

We will examine whether the following baseline variables modify the effect of study group on the primary outcome:

- Age (continuous variable);
- Race and ethnicity (Hispanic, Non-Hispanic Black, Non-Hispanic White, Other);
- Source of admission to the ICU (ED, hospital ward, another ICU in the study hospital, operating room, outside hospital);

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

• Duration of invasive mechanical ventilation prior to enrollment (0 minutes; 1 to 360 minutes; >360 minutes);

- Chronic comorbidities (categories are not mutually exclusive)
  - Receipt of supplemental oxygen at place of residence prior to hospital admission (yes, no);
  - Coronary artery disease or heart failure with reduced ejection fraction (yes, no);
- Acute diagnoses at enrollment (categories are not mutually exclusive)
  - cardiac arrest (yes, no);
  - acute myocardial infarction (yes, no);
  - sepsis or septic shock (yes, no);
  - acute respiratory distress syndrome (yes, no);
- Receipt of vasopressors at enrollment (yes, no);
- Non-respiratory SOFA score at enrollment (continuous variable);
- Time period (before the COVID-19 pandemic [July 2018 December 2019], during the COVID-19 pandemic [January 2020 – August 2021]).

#### Analysis of the Secondary Outcome

The sole pre-specified secondary outcome of 28-day in-hospital mortality will be compared between the three study groups in an intention-to-treat fashion in the primary analysis population using a logistic regression model with independent covariates of group assignment (higher, intermediate, or lower SpO2 target) and time. We also will perform pair-wise comparisons between the lower and intermediate groups, lower and higher groups, and intermediate and higher groups using the same statistical approach.

#### Analysis of the Exploratory Outcomes

Each of the exploratory outcomes will be compared between groups in an intention-to-treat fashion in the primary analysis population. Continuous outcomes will be compared between groups using a proportional odds model with independent covariates of group assignment (higher, intermediate, or lower SpO2 target) and time. Categorical outcomes will be compared between groups using a logistic regression model with independent covariates of group assignment (higher, intermediate, or lower SpO2 target) and time.

#### Corrections for multiple testing

We have pre-specified a single primary outcome and a single secondary outcome. Consistent with recommendations of the Food and Drug Administration and the European Medicines Association, each will be tested using a two-sided p-value with a significance level of 0.05. For all other analyses, emphasis will be placed on the estimate of effect size with 95% confidence intervals, as recommended by the

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

International Committee of Medical Journal Editors, and no corrections for multiple comparisons will be performed.

# Handling of missing data

The primary outcome of VFDs is not anticipated to be missing for any patients. Missing data will not be imputed for the primary outcome or any secondary or exploratory outcomes. In adjusted analyses, missing data for covariates will be imputed using multiple imputations.

# **Interim Analysis**

We will plan for the DSMB to conduct a single interim analysis for efficacy and safety at the anticipated halfway point of the trial. The interim analysis will include patients enrolled during the first 18 months of the trial. The stopping boundary for efficacy will be met if the P value for the difference between groups is <0.001 using a proportional odds model with independent covariates of group assignment (higher, intermediate, or lower SpO2 target) and time with regard to the primary outcome of VFDs. Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05). Given the minimal risk nature of the study and current use of all SpO2 target as a part of usual care, there will be no stopping boundary for futility. The DSMB will reserve the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety.

If the 18-month interim analysis reveals an enrollment indicative of <80% statistical power at completion, we will ask the DSMB to approve extending enrollment of the study to ensure the trial is not underpowered to detect the planned difference between groups in the primary outcome.

#### 12.0 Privacy/Confidentiality Issues

At no time during the course of this study, its analysis, or its publication will patient identities be revealed in any manner. The minimum necessary data containing patient or provider identities will be collected. All patients will be assigned a unique study ID number for tracking. Data collected from the medical record will be entered into the secure online database REDCap. Hard copies of the treating clinician modification of SpO<sub>2</sub> target sheet will be stored in a locked room until after the completion of enrollment and data cleaning. Once data are verified and the database is locked, all hard copies of data collection forms will be destroyed. All data will be maintained in the secure online database REDCap until the time of study publication. At the time of publication, a de-identified version of the database will be generated.

# 13.0 Follow-up and Record Retention

Patients will be followed after enrollment for 28 days or until hospital discharge, whichever occurs first. Data collected from the medical record will be entered into the

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

secure online database REDCap. Once data are verified and the database is locked, all hard copies of data collection forms will be destroyed. All data will be maintained in the secure online database REDCap until the time of study publication. At the time of publication, a de-identified version of the database will be generated.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

#### 14.0 References

1. Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med 2010;38(10):1947–53.

- 2. Wunsch H, Angus DC, Harrison DA, Linde-Zwirble WT, Rowan KM. Comparison of medical admissions to intensive care units in the United States and United Kingdom. Am J Respir Crit Care Med 2011;183(12):1666–73.
- 3. Adhikari NKJ, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet Lond Engl 2010;376(9749):1339–46.
- 4. Dasta JF, McLaughlin TP, Mody SH, Piech CT. Daily cost of an intensive care unit day: the contribution of mechanical ventilation. Crit Care Med 2005;33(6):1266–71.
- 5. Halpern NA, Pastores SM. Critical care medicine in the United States 2000-2005: an analysis of bed numbers, occupancy rates, payer mix, and costs. Crit Care Med 2010;38(1):65–71.
- 6. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. The Acute Respiratory Distress Syndrome Network. N Engl J Med 2000;342(18):1301–8.
- 7. Esteban A, Frutos-Vivar F, Muriel A, et al. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med 2013;188(2):220–30.
- 8. Herridge MS, Cheung AM, Tansey CM, et al. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med 2003;348(8):683–93.
- 9. Herridge MS, Tansey CM, Matté A, et al. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med 2011;364(14):1293–304.
- 10. Kahn JM, Benson NM, Appleby D, Carson SS, Iwashyna TJ. Long-term acute care hospital utilization after critical illness. JAMA 2010;303(22):2253–9.
- 11. Pandharipande PP, Girard TD, Jackson JC, et al. Long-term cognitive impairment after critical illness. N Engl J Med 2013;369(14):1306–16.
- 12. Fridovich I. Oxygen toxicity: a radical explanation. J Exp Biol 1998;201(Pt 8):1203–9.
- 13. Heffner JE, Repine JE. Pulmonary strategies of antioxidant defense. Am Rev Respir Dis 1989;140(2):531–54.
- 14. Freeman BA, Crapo JD. Hyperoxia increases oxygen radical production in rat lungs and lung mitochondria. J Biol Chem 1981;256(21):10986–92.
- 15. Waxman AB, Einarsson O, Seres T, et al. Targeted lung expression of interleukin-11 enhances murine tolerance of 100% oxygen and diminishes hyperoxia-induced DNA fragmentation. J Clin Invest 1998;101(9):1970–82.
- 16. Griffith DE, Garcia JG, James HL, Callahan KS, Iriana S, Holiday D. Hyperoxic exposure in humans. Effects of 50 percent oxygen on alveolar macrophage leukotriene B4 synthesis. Chest 1992;101(2):392–7.
- 17. Davis WB, Rennard SI, Bitterman PB, Crystal RG. Pulmonary oxygen toxicity. Early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med 1983;309(15):878–83.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

18. Aggarwal NR, Brower RG. Targeting normoxemia in acute respiratory distress syndrome may cause worse short-term outcomes because of oxygen toxicity. Ann Am Thorac Soc 2014;11(9):1449–53.

- 19. Meade MO, Cook DJ, Guyatt GH, et al. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA J Am Med Assoc 2008;299(6):637–45.
- 20. Eastwood G, Bellomo R, Bailey M, et al. Arterial oxygen tension and mortality in mechanically ventilated patients. Intensive Care Med 2012;38(1):91–8.
- 21. de Jonge E, Peelen L, Keijzers PJ, et al. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care Lond Engl 2008;12(6):R156.
- 22. National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network, Rice TW, Wheeler AP, et al. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA J Am Med Assoc 2012;307(8):795–803.
- 23. Rice TW, Wheeler AP, Thompson BT, et al. Enteral omega-3 fatty acid, gammalinolenic acid, and antioxidant supplementation in acute lung injury. JAMA J Am Med Assoc 2011;306(14):1574–81.
- 24. O'Driscoll BR, Howard LS, Earis J, Mak V, British Thoracic Society Emergency Oxygen Guideline Group, BTS Emergency Oxygen Guideline Development Group. BTS guideline for oxygen use in adults in healthcare and emergency settings. Thorax 2017;72(Suppl 1):ii1–90.
- 25. Supplemental Therapeutic Oxygen for Prethreshold Retinopathy Of Prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. Pediatrics 2000;105(2):295–310.
- 26. SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network, Carlo WA, Finer NN, et al. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med 2010;362(21):1959–69.
- 27. Schmidt B, Whyte RK, Asztalos EV, et al. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. JAMA 2013;309(20):2111–20.
- 28. BOOST II United Kingdom Collaborative Group, BOOST II Australia Collaborative Group, BOOST II New Zealand Collaborative Group, et al. Oxygen saturation and outcomes in preterm infants. N Engl J Med 2013;368(22):2094–104.
- 29. Panwar R, Hardie M, Bellomo R, et al. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med 2016;193(1):43–51.
- 30. Girardis M, Busani S, Damiani E, et al. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA 2016;316(15):1583–9.
- 31. Asfar P, Schortgen F, Boisramé-Helms J, et al. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med [Internet] 2017 [cited 2017 Feb 20]; Available from: http://linkinghub.elsevier.com/retrieve/pii/S2213260017300462

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

32. Panwar R, Capellier G, Schmutz N, et al. Current oxygenation practice in ventilated patients-an observational cohort study. Anaesth Intensive Care 2013;41(4):505–14.

- 33. Suzuki S, Eastwood GM, Peck L, Glassford NJ, Bellomo R. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care 2013;28(5):647–54.
- 34. Beasley R, Chien J, Douglas J, et al. Thoracic Society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: 'Swimming between the flags.' Respirol Carlton Vic 2015;20(8):1182–91.
- 35. Severinghaus JW. Simple, accurate equations for human blood O2 dissociation computations. J Appl Physiol 1979;46(3):599–602.
- 36. Stollings JL, Foss JJ, Ely EW, et al. Pharmacist leadership in ICU quality improvement: coordinating spontaneous awakening and breathing trials. Ann Pharmacother 2015;49(8):883–91.
- 37. Girard TD, Kress JP, Fuchs BD, et al. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet Lond Engl 2008;371(9607):126–34.
- 38. Semler MW, Noto MJ, Stollings J, et al. Effect Of Saline Versus Balanced Crystalloids On Major Adverse Kidney Events In The Medical Intensive Care Unit: The Salt Randomized Trial. Am J Respir Crit Care Med 2016;193:A4290.
- 39. Harris BU, Char DS, Feinstein JA, Verma A, Shiboski SC, Ramamoorthy C. Accuracy of Pulse Oximeters Intended for Hypoxemic Pediatric Patients. Pediatr Crit Care Med J Soc Crit Care Med World Fed Pediatr Intensive Crit Care Soc 2016;17(4):315–20.
- 40. Ehrenfeld JM, Funk LM, Van Schalkwyk J, Merry AF, Sandberg WS, Gawande A. The incidence of hypoxemia during surgery: evidence from two institutions. Can J Anaesth J Can Anesth 2010;57(10):888–97.
- 41. Lopez MG, Pretorius M, Shotwell MS, et al. The Risk of Oxygen during Cardiac Surgery (ROCS) trial: study protocol for a randomized clinical trial. Trials 2017;18(1):295.
- 42. Brower RG, Lanken PN, MacIntyre N, et al. Higher versus lower positive endexpiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med 2004;351(4):327–36.
- 43. Briel M, Meade M, Mercat A, et al. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA J Am Med Assoc 2010;303(9):865–73.
- 44. Barr J, Fraser GL, Puntillo K, et al. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med 2013;41(1):263–306.
- 45. Gélinas C, Fortier M, Viens C, Fillion L, Puntillo K. Pain assessment and management in critically ill intubated patients: a retrospective study. Am J Crit Care Off Publ Am Assoc Crit-Care Nurses 2004;13(2):126–35.
- 46. Sessler CN, Grap MJ, Brophy GM. Multidisciplinary management of sedation and analgesia in critical care. Semin Respir Crit Care Med 2001;22(2):211–26.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

47. Ely EW, Truman B, Shintani A, et al. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA 2003;289(22):2983–91.

- 48. Ely EW, Margolin R, Francis J, et al. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med 2001;29(7):1370–9.
- 49. Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med 1990;113(12):941–8.
- 50. Semler MW, Rice TW, Shaw AD, et al. Identification of Major Adverse Kidney Events Within the Electronic Health Record. J Med Syst 2016;40(7):167.
- 51. Semler MW, Self WH, Wang L, et al. Balanced crystalloids versus saline in the intensive care unit: study protocol for a cluster-randomized, multiple-crossover trial. Trials 2017;18(1).
- 52. Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med 1985;13(10):818–29.
- 53. Vincent JL, Moreno R, Takala J, et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med 1996;22(7):707–10.
- 54. Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet Lond Engl 1974;2(7872):81–4.
- 55. Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care 1998;36(1):8–27.
- 56. ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, et al. Acute respiratory distress syndrome: the Berlin Definition. JAMA J Am Med Assoc 2012;307(23):2526–33.
- 57. Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney inter 2012;2(Suppl):8.
- 58. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42(2):377–81.

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

# **Tracking of Protocol Versions:**

# Version 1.0 – Initial Protocol (5/1/2018)

# Version 1.1 – Revisions after initial meeting with DSMB (6/8/18)

- Updated protocol to specify that the primary analysis will use a proportional odd mixed effects model with a fixed effect of study group and a random effect of study period.
- Added sensitivity analyses using a zero-inflated Poisson model and a statetransitions model
- Specified the plan for sample size re-estimation at the interim analysis as follows: "If the 18-month interim analysis reveals an enrollment indicative of <80% statistical power at completion, we will ask the DSMB to approve extending enrollment of the study to ensure the trial is not underpowered to detect the planned difference between groups in the primary outcome."
- Specified that "Patients will be provided with an information sheet providing an IRB-approved lay language summary of the study activities. The information sheet will contain the contact information for the primary investigator who will remain available throughout the study period to provide additional information to patients and families upon request. All contact between patients, families, and surrogates and study personnel will be tracked in a case report form and available to investigators and the DSMB."

# <u>Version 1.2 – Protocol revisions during implementation (11/14/18)</u>

- Updated protocol to remove FiO2 and PEEP criteria from the SBT Safety Screen to allow patients who pass other elements of the SBT Safety Screen to attempt a daily SBT regardless of their current FiO2 or PEEP.
- Revised the Patient Information Sheet based on feedback from the Community-Engaged Research Core and patients on the Community Advisory Council to create a structured format with headers, make the narrative more conversational, and decrease the reading level.

# Version 1.3 – Protocol revisions prior to Continuing Review (6/19/19)

- Updated protocol to provide additional detail regarding (a) the process used to provide information about the study the patients, families, and surrogates in the study setting and (b) the documentation of this process.
- Updated the figures to match the changes to the SAT and SBT safety screen made during the 11/14/18 amendment.

#### Version 1.4 – Protocol revisions to incorporate final Statistical Analysis Plan (10/20/20)

- Revised trial name from "Preliminary Investigation of optimaL Oxygen Targets" to "Pragmatic Investigation of optimaL Oxygen Targets" to reflect the design
- Added details on the calculation of the primary outcome of VFDs to match SAP.
- Separated out the sole pre-specified secondary outcome of 28-day in-hospital

Study Title: Pragmatic Investigation of optimal Oxygen Targets (PILOT) Trial

Institution: Vanderbilt University Medical Center

mortality from the exploratory outcomes to match SAP.

- Added details on "Primary Analysis of the Primary Outcome", "Sensitivity Analyses of the Primary Outcome", "Analysis of Effect Modification for the Primary Outcome", "Analysis of the Secondary Outcome", "Analysis of the Exploratory Outcomes", "Corrections for multiple testing", and "Handling of missing data" to match the SAP.
- Updated figure with study group assignments to reflect paused enrollment in April and May of 2020 due to COVID-19.

# <u>Version 1.5 – Protocol revisions to incorporate updates to Statistical Analysis Plan during</u> peer review (4/7/2021)

- Revise statistical analysis plan to clarify how patients with a diagnosis of COVID-19 will be analyzed in the primary analysis, sensitivity analyses, and analyses of effect modification.
- Revise statistical analysis plan to define how race and ethnicity will be defined in the analysis of effect modification.

# Summary of Changes to the PILOT Trial Protocol

#### Version 1.0 – Initial Protocol (5/1/2018)

#### Version 1.1 – Revisions after initial meeting with DSMB (6/8/18)

- Updated protocol to specify that the primary analysis will use a proportional odd mixed effects model with a fixed effect of study group and a random effect of study period.
- · Added sensitivity analyses using a zero-inflated Poisson model and a state-transitions model
- Specified the plan for sample size re-estimation at the interim analysis as follows: "If the 18-month interim analysis reveals an enrollment indicative of <80% statistical power at completion, we will ask the DSMB to approve extending enrollment of the study to ensure the trial is not underpowered to detect the planned difference between groups in the primary outcome."
- Specified that "Patients will be provided with an information sheet providing an IRB-approved lay language summary of the study activities. The information sheet will contain the contact information for the primary investigator who will remain available throughout the study period to provide additional information to patients and families upon request. All contact between patients, families, and surrogates and study personnel will be tracked in a case report form and available to investigators and the DSMB."

#### <u>Version 1.2 – Protocol revisions during implementation (11/14/18)</u>

- Updated protocol to remove FiO2 and PEEP criteria from the SBT Safety Screen to allow patients who pass other elements of the SBT Safety Screen to attempt a daily SBT regardless of their current FiO2 or PEEP.
- Revised the Patient Information Sheet based on feedback from the Community-Engaged Research Core and patients on the Community Advisory Council to create a structured format with headers, make the narrative more conversational, and decrease the reading level.

#### Version 1.3 – Protocol revisions prior to Continuing Review (6/19/19)

- Updated protocol to provide additional detail regarding (a) the process used to provide information about the study the patients, families, and surrogates in the study setting and (b) the documentation of this process.
- Updated the figures to match the changes to the SAT and SBT safety screen made during the 11/14/18 amendment.

#### Version 1.4 – Protocol revisions to incorporate final Statistical Analysis Plan (10/20/20)

- Revised trial name from "Preliminary Investigation of optimaL Oxygen Targets" to "Pragmatic Investigation of optimaL Oxygen Targets" to reflect the design
- Added details on the calculation of the primary outcome of VFDs to match SAP.
- Separated out the sole pre-specified secondary outcome of 28-day in-hospital mortality from the exploratory outcomes to match SAP.
- Added details on "Primary Analysis of the Primary Outcome", "Sensitivity Analyses of the Primary Outcome", "Analysis of Effect Modification for the Primary Outcome", "Analysis of the Secondary Outcome", "Analysis of the Exploratory Outcomes", "Corrections for multiple testing", and "Handling of missing data" to match the SAP.
- Updated figure with study group assignments to reflect paused enrollment in April and May of 2020 due to COVID-19.

# <u>Version 1.5 – Protocol revisions to incorporate updates to Statistical Analysis Plan during peer review</u> (4/7/2021)

- Revise statistical analysis plan to clarify how patients with a diagnosis of COVID-19 will be analyzed in the primary analysis, sensitivity analyses, and analyses of effect modification.
- Revise statistical analysis plan to define how race and ethnicity will be defined in the analysis
  of effect modification.

Protocol and Statistical Analysis Plan for the Pragmatic Investigation of Optimal Oxygen Targets (PILOT) Clinical Trial

Matthew W. Semler, MD, MSc<sup>1</sup>, Jonathan D. Casey MD<sup>1</sup>, Bradley D. Lloyd RRT-ACCS<sup>2</sup>, Pamela G. Hastings RRT-ACCS<sup>2</sup>, Margaret A. Hays, RN<sup>1</sup>, Megan Roth, RN<sup>1</sup>, Joanna L. Stollings, PharmD, FCCM, FCCP<sup>3</sup>, John H. Brems, MD<sup>4</sup>; Kevin G. Buell MBBS<sup>4</sup>; Li Wang, MS<sup>5</sup>, Christopher J. Lindsell, PhD<sup>5</sup>; Robert E. Freundlich, MD<sup>6</sup>; Jonathan P. Wanderer, MD, MPhil<sup>6</sup>; Gordon R. Bernard MD<sup>1</sup>; Wesley H. Self MD, MPH<sup>7</sup>; Todd W. Rice, MD, MSc<sup>1</sup> for the PILOT Investigators\* and the Pragmatic Critical Care Research Group.

\* A full list of the PILOT Investigators may be found in supplemental file 1, section 1.

Affiliations: <sup>1</sup>Division of Allergy, Pulmonary, and Critical Care Medicine; <sup>2</sup>Division of Respiratory Care; <sup>3</sup>Department of Pharmaceutical Services; <sup>4</sup>Department of Medicine; <sup>5</sup>Department of Biostatistics; <sup>6</sup>Department of Anesthesiology and Department of Biomedical Informatics; <sup>7</sup>Department of Emergency Medicine – all at Vanderbilt University Medical Center, Nashville, TN

### Corresponding author:

Matthew W. Semler, MD, MSc

T-1210 MCN, 1161 21st Ave S., Nashville, TN 37232-2650

Fax: (615) 343-7448

Corresponding Author's Email Address: matthew.w.semler@vumc.org

Key words for indexing: Oxygen, Mechanical ventilation, Respiratory Failure

Subject Descriptor Number: 4.4 Clinical Trials in Critical Care Medicine

Manuscript Word Count (body only): 4,102

Abstract Word Count: 225 Version Date: April 2, 2021

#### ABSTRACT:

**Introduction:** Mechanical ventilation of intensive care unit (ICU) patients universally involves titration of the fraction of inspired oxygen (FiO<sub>2</sub>) to maintain arterial oxygen saturation (SpO<sub>2</sub>). However, the optimal SpO<sub>2</sub> target remains unknown.

Methods and Analysis: The Pragmatic Investigation of optimal Oxygen Targets (PILOT) trial is a prospective, unblinded, pragmatic, cluster-crossover trial being conducted in the emergency department and medical ICU at Vanderbilt University Medical Center in Nashville, TN, USA. PILOT compares use of a lower SpO2 target (target 90% and goal range 88-92%), an intermediate SpO2 target (target 94% and goal range 92-96%), and a higher SpO2 target (target 98% and goal range 96-100%). The study units are assigned to a single SpO2 target (cluster-level allocation) for each two-month study block, and the assigned SpO2 target switches every two months in a randomly generated sequence (cluster-level crossover). The primary outcome is ventilator-free days to study day 28, defined as the number of days alive and free of invasive mechanical ventilation from the final receipt of invasive mechanical ventilation through 28 days after enrollment.

**Ethics and dissemination:** The trial was approved by the Vanderbilt Institutional Review Board. The results will be submitted for publication in a peer-reviewed journal and presented at one or more scientific conferences.

**Trial Registration:** The trial protocol was registered with ClinicalTrials.gov on May 25, 2018 prior to initiation of patient enrollment (ClinicalTrials.gov identifier: NCT03537937).

# **ARTICLE SUMMARY**

Strengths and limitations of this study

- This ongoing pragmatic trial will provide information on the optimal oxygen saturation target during invasive mechanical ventilation of critically ill adults – informing a common therapy in current clinical practice for which there is limited available evidence on which to base care
- Broad inclusion criteria will increase generalizability and the sample size will allow examination of important patient subgroups
- The trial is being conducted at a single center
- The nature of the study intervention does not allow blinding
- Decisions regarding oxygen administration before and after invasive mechanical ventilation are deferred to treating clinicians

#### INTRODUCTION

Each year 2-3 million intensive care unit (ICU) patients receive invasive mechanical ventilation [1–3]. Despite recent advances in lung-protective ventilation [4], in-hospital mortality among mechanically ventilated ICU patients remains 25-35% [5].

Mechanical ventilation for ICU patients universally involves titrating the fraction of inspired oxygen (FiO<sub>2</sub>) to maintain arterial oxygen saturation (SpO<sub>2</sub>) within a goal range. Despite decades of ICU practice, however, the optimal SpO<sub>2</sub> target remains unknown. Higher SpO<sub>2</sub> targets (96-100%) provide a margin of safety against hypoxemia, but may increase exposure to excess FiO<sub>2</sub>, hyperoxemia, and tissue hyperoxia, causing oxidative damage [6–8], inflammation [9,10], and increased alveolar-capillary permeability [11]. Lower SpO<sub>2</sub> targets (88-92%) minimize exposure to excess FiO<sub>2</sub>, hyperoxemia, and tissue hyperoxia [4,12,13], but may increase the risk of hypoxemia and tissue hypoxia [14,15]. An intermediate SpO<sub>2</sub> target (92-96%) may avoid the risks of both hyperoxia and hypoxia or, conversely, may expose patients intermittently to both sets of risks [16,17].

The relative risks and benefits of different SpO<sub>2</sub> or PaO<sub>2</sub> targets have been extensively examined in the setting of the neonatal ICU [18–21] and have been examined among adult ICU patients in a series of recently-published clinical trials [22–27]. Together, these trials have suggested that both higher and lower oxygenation targets are safe – although some trials have potentially suggested better outcomes with higher targets[25] and other trials have suggested potentially better outcomes with lower targets[24].

Given the still incomplete evidence from randomized trials, current guidelines offer divergent recommendations – ranging from tolerating SpO<sub>2</sub> values as low as 88% [28–30] to pursuing SpO<sub>2</sub> values as high as 98% [31]. In clinical practice, hyperoxemia remains common [32,33], even among patients cared for by clinicians who self-identify as avoiding high oxygen levels [34].

The wide variation in current practice, conflicting guidelines, and conflicting data from some available trials indicate the need for further clinical trials to determine the effect of SpO<sub>2</sub> target on patient outcomes [12,35]. We designed the <u>Pragmatic Investigation of optimal Oxygen Targets</u> (PILOT) trial to examine the effects of higher, intermediate, and lower SpO<sub>2</sub> targets on the number of days alive and free of invasive mechanical ventilation among mechanically ventilated ICU patients.

#### **METHODS AND ANALYSIS**

This manuscript was prepared in accordance with Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines (Figure 1; SPIRIT checklist in online supplemental file 1, section 2). [36] This manuscript describes key elements of the trial protocol and statistical analysis plan. The Supplemental Methods in supplemental file 1 provide additional background on prior trials (section 3), rationale for design decisions (sections 4-5), SpO<sub>2</sub> monitoring and management (sections 6-8), institutional protocols for mechanical ventilation (sections 9-17), a complete list of data elements (section 18), definitions of exploratory outcomes and measures of separation between groups (sections 19-21), and details of the interim analysis (section 22) and secondary analyses (sections 23-25).

# Study Design

The PILOT trial is a prospective, unblinded, pragmatic, cluster-crossover trial being conducted in the emergency department and medical ICU at Vanderbilt University Medical Center in Nashville, TN, USA. PILOT compares use of a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%), an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%), and a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%) with regard to the number of days alive and free of invasive mechanical ventilation among mechanically ventilated ICU patients. Consistent with the concept of a pragmatic clinical trial [37], the eligibility criteria are broad, the delivery of the intervention is embedded in routine clinical care and executed by clinical personnel, and data collection prioritizes clinical outcomes over mechanistic evaluation. The trial was approved by the Vanderbilt University Medical Center Institutional Review Board (IRB) (IRB 171272). The trial is investigator-initiated with funding provided by the National Heart, Lung, and Blood Institute (K23HL143053). The trial protocol was registered with ClinicalTrials.gov on May 25, 2018 prior to initiation of patient enrollment on July 1, 2018 (ClinicalTrials.gov identifier: NCT03537937).

#### Patient and Public Involvement

Materials used to communicate about the study with patients and families were developed with input from the Vanderbilt Community Engaged Research Core and the Vanderbilt Community Advisory Council.

# Study Site and Population

The trial is being conducted in the adult emergency department (ED) and medical ICU at Vanderbilt University Medical Center.

### The inclusion criteria are:

- 1. Age ≥ 18 years
- 2. Receiving mechanical ventilation through an endotracheal tube or tracheostomy
- 3. Admitted to the study ICU or admission to the study ICU from the ED is planned

# The exclusion criteria are:

- Known pregnancy or beta hCG level greater than the laboratory upper limit of normal in a patient capable of becoming pregnant (if measured clinically)
- 2. Known to be a prisoner

Adults located in the study ICU or for whom admission to the study ICU from the ED is planned who meet inclusion criteria and do not meet exclusion criteria are enrolled immediately upon receipt of invasive mechanical ventilation in a study location. The time of enrollment for the trial ("time zero") is the time of first receipt of invasive mechanical ventilation in a participating study location.

#### Randomization and Treatment Allocation

For each of the 18 two-month blocks during the 36 months of enrollment in the PILOT trial, the medical ICU is assigned to a single SpO<sub>2</sub> target (cluster-level

allocation). Every two months, the ICU will switch between use of a lower SpO<sub>2</sub> target (target 90% and goal range 88-92%), use of an intermediate SpO<sub>2</sub> target (target 94% and goal range 92-96%), and use of a higher SpO<sub>2</sub> target (target 98% and goal range 96-100%) in a randomly generated sequence (cluster-level crossover) (Figure 2). The order of study group assignments for each two-month block was generated by computerized randomization using permuted blocks of 3 to minimize the impact of seasonal variation and temporal changes. For the 36 months of enrollment in the PILOT trial, patients receiving invasive mechanical ventilation in the ED for whom admission to the medical ICU is planned will receive the same SpO<sub>2</sub> target assigned to the medical ICU. The study did not enroll in April and May of 2020 due to disruptions in research and clinical care from the Coronavirus Infectious Disease 2019 (COVID-19) pandemic (Figure 2).

#### Washout Periods

The last 7 days of each two-month block are considered an analytic washout period during which the ICU continues to target the assigned SpO<sub>2</sub> but data from new patients are not included in the primary analysis. Assuming a median duration of mechanical ventilation of 3 [IQR 3-5] days, a 7-day washout period will ensure that 98% patients in the primary analysis do not experience a "crossover" from a period assigned to one assigned SpO<sub>2</sub> target to a period assigned to another SpO<sub>2</sub> target. Data from patients admitted during washout periods will be included in a pre-specified sensitivity analysis (see *Statistical Analysis* section). Any patient who does remain mechanically ventilated in the study ICU through a crossover from a period assigned to one SpO<sub>2</sub>

target to a period assigned to another SpO<sub>2</sub> target will be analyzed in the SpO<sub>2</sub> target group to which the ICU was assigned at the time of the patient's enrollment in the trial (intention-to-treat analysis).

# Study Interventions

# Choice of SpO<sub>2</sub> targets

In clinical practice, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adults fall between 88-100% [32,33]. Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: (1) allowing the lower end of the range of acceptable SpO<sub>2</sub> values to be as low as 88% [28,29] to avoid excess FiO<sub>2</sub>, hyperoxemia, and hyperoxia; (2) titrating within an intermediate range of SpO<sub>2</sub> values, such as 92-96% [38]; or (3) targeting higher SpO<sub>2</sub> to avoid the risks of hypoxemia and hypoxia [31]. The PILOT trial has three study groups, each emulating a different approach to SpO<sub>2</sub> targets represented in guidelines and clinical practice (Table 1).

# Oxygen Titration

In the study ED and ICU, titration of FiO<sub>2</sub> to maintain SpO<sub>2</sub> for mechanically ventilated adults is typically performed by respiratory therapists with input from nurses and physicians. In preparation for the PILOT trial, we collaborated with respiratory therapy leaders in the study ED and ICU to adapt existing ventilator management protocols to provide guidance for respiratory therapists in titrating FiO<sub>2</sub> to achieve each of the three study SpO<sub>2</sub> targets.

For patients enrolled in the study, respiratory therapists are instructed to begin titrating FiO<sub>2</sub> to the target SpO<sub>2</sub> value within 15 minutes of the initiation of mechanical ventilation. During the maintenance of invasive mechanical ventilation, SpO<sub>2</sub> is assessed by continuous pulse oximetry. The protocol directs the respiratory therapist managing the patient's ventilator to target an SpO<sub>2</sub> value of 90% in the lower SpO<sub>2</sub> target group, an SpO<sub>2</sub> value of 94% in the intermediate SpO<sub>2</sub> target group, and an SpO<sub>2</sub> value of 98% in the higher SpO<sub>2</sub> target group (Table 1). Respiratory therapists and other treating clinicians titrate FiO<sub>2</sub> when the SpO<sub>2</sub> out of the goal range, when the SpO<sub>2</sub> is within the goal range but closer alignment with the assigned SpO<sub>2</sub> target is desired, to facilitate weaning from mechanical ventilation, or for other clinical indications. SpO<sub>2</sub> is reassessed 5 minutes after each change in FiO<sub>2</sub> or sooner if clinically indicated.

The protocol determines the SpO<sub>2</sub> target from enrollment until the first of: (1) discontinuation of invasive mechanical ventilation, (2) transfer out of a participating study location, (3) completion of an SpO<sub>2</sub> target modification sheet by treating clinicians, or (4) end of the two-month study period. The protocol does not determine the SpO<sub>2</sub> target during time-periods in which the patient is not physically located in a study location (e.g., during transport) or when FiO<sub>2</sub> is being administered for purposes other than achieving a target SpO<sub>2</sub> (e.g., when an FiO<sub>2</sub> of 1.0 is being administered for a procedure).

At any time, if a treating clinician or a patient, family member, or surrogate feels that an SpO<sub>2</sub> target other than that assigned by the study would be best for the optimal treatment of the patient for any reason, the SpO<sub>2</sub> target for that patient is modified. To modify the target, the respiratory therapist and supervising physician complete a one-

page SpO<sub>2</sub> target modification sheet documenting the new SpO<sub>2</sub> target and the rationale for modifying the target. Examples of conditions for which the assigned SpO<sub>2</sub> target may be modified that were specified in the initial trial protocol included: pneumothorax; pneumomediastinum; carbon monoxide poisoning; decompression sickness; bleomycin toxicity; paraquat toxicity. Examples of conditions for which the assigned SpO<sub>2</sub> target may be modified that were not explicitly specified in the initial trial protocol include: severe chronic obstructive pulmonary disease; severe acute respiratory distress syndrome; severe anemia; status post lung transplantation; and receipt of extracorporeal membrane oxygenation support. Trial protocol directs only the titration of FiO<sub>2</sub> to the assigned SpO<sub>2</sub> target. Other aspects of invasive mechanical ventilation, such as tidal volume [4], positive end-expiratory pressure [39,40], and use of rescue therapies for hypoxemia, are determined by institutional protocols and treating clinicians (see sections 9-17 of supplemental file 1).

# Blinding

Similar to prior studies of SpO<sub>2</sub> targets among critically ill adults [22,24,26], patients and clinicians will not be blinded to study group assignment.

#### Data Collection

The PILOT trial uses data collected by two methods to minimize observer bias:

(1) manual data collection by study personnel and (2) automated collection of structured data recorded in routine clinical care, exported daily from the institution's electronic health record and patient registration, billing, and laboratory clinical information systems
into an Enterprise Data Warehouse. We have previously validated the quality of the automated method of data collection against the reference standard of two-physician manual chart review [41] and have employed this approach for the conduct of prior pragmatic trials [42,43]. Data are stored, curated, and secured in REDCap [44].

#### Outcomes

# **Primary Outcome**

The primary outcome is ventilator-free days (VFDs) to study day 28. VFDs will be defined as the number of whole calendar days alive and free of invasive mechanical ventilation beginning at midnight on the day of the final receipt of invasive mechanical ventilation through day 28 after enrollment [45,46]. Outcome ascertainment will cease at the time of hospital discharge or 28 days after enrollment, whichever occurs first. Receipt of invasive mechanical ventilation will be considered to end when patients undergo the final tracheal extubation or disconnection of the ventilator from the endotracheal tube or tracheostomy tube between enrollment and 28 days after enrollment. Patients whose final receipt of invasive mechanical ventilation occurs on the day of enrollment will receive 27 VFDs. Patients who continue to receive invasive mechanical ventilation 28 days after enrollment will receive 0 VFDs. Patient who die prior to day 28 will receive 0 VFDs. Patients who are discharged from the hospital prior to day 28 and are receiving invasive mechanical ventilation at the time of discharge will receive 0 VFDs. Patients who are removed from invasive mechanical ventilation and are discharged from the hospital without invasive mechanical ventilation prior to 28 days will be assumed to remain free of invasive mechanical ventilation between hospital

ventilation, return to invasive mechanical ventilation, and are subsequently removed again from invasive mechanical ventilation prior to day 28, VFDs will be counted from the final receipt of invasive mechanical ventilation prior to day 28.

# Secondary Outcome

The sole pre-specified secondary outcome is 28-day in-hospital mortality, defined as death from any cause between enrollment and the first of hospital discharge or 28 days after enrollment.

# **Exploratory Clinical Outcomes**

- ICU mortality death in the ICU between enrollment and the first of 28 days after enrollment or hospital discharge
- Free-day outcomes defined as whole calendar days from last receipt of therapy until 28 days (supplemental file 1, section 19)
  - a. Vasopressor-free days
  - b. Renal replacement therapy-free days
  - c. ICU-free days
  - d. Hospital-free days

# **Exploratory Organ Function Outcomes**

- 1. Daily non-respiratory SOFA score (Table S1) [47]
- 2. Plasma creatinine concentration (mg/dL)

- 3. Plasma lactate concentration (mmol/L)
- 4. Presence of acute respiratory distress syndrome by Berlin criteria [48]
- Stage II or greater AKI by Kidney Disease: Improving Global Outcomes
   (KDIGO) creatinine criteria [49]

# **Exploratory Safety Outcomes**

- 1. Atrial arrhythmia
- 2. Ventricular arrhythmia
- 3. Cardiac arrest with return of spontaneous circulation
- 4. Pneumothorax or pneumomediastinum
- 5. Ischemic stroke
- 6. Myocardial infarction [50]

# Additional Long-term Patient-Important Outcomes

The independently-funded Cognitive Outcomes in the Pragmatic Investigation of Optimal Oxygen Targets (CO-PILOT) study (R21AG063126) will assess cognitive, physical, and psychological outcomes at 12 months after enrollment in the PILOT trial. The protocol and statistical analysis plan for the CO-PILOT study will be published separately.

# **Statistical Analysis and Reporting**

Sample Size Estimation and Power Calculation

In a prior cluster-randomized cluster-crossover trial in the same ICU [51], 880 mechanically ventilated adults were enrolled per year (73.3 per month), with a median of 22 VFDs [IQR 0-25 VFDs] and an intra-cluster intra-period correlation of 0.01. We estimate 2,640 mechanically ventilated adults will be admitted to the study ICU during the 36-month PILOT trial, of whom 390 will be excluded from the primary analysis for initial receipt of invasive mechanical ventilation in a study location during a washout period and 2,250 will be enrolled and included in the primary analysis. With a total enrollment of 2,250 patients, a standard deviation in the primary outcome of VFDs of 11.4 days, and a two-sided alpha of 0.05, we calculated using a t-test that the PILOT trial will have 92 percent statistical power to detect an absolute reduction in VFDs of 2.0 days (similar to the numerical difference in VFDs between SpO<sub>2</sub> target groups reported in prior studies [22,24]).

# Data and Safety Monitoring Board and Interim Analysis

An independent Data and Safety Monitoring Board (DSMB) oversees the trial.

On March 23, 2020 the DSMB conducted a single, planned interim analysis at the anticipated halfway point of the trial and recommended the trial continue without modification (see DSMB charter in online supplemental file 2 and details of interim analysis in supplemental file 1, section 22). The DSMB is composed of two physicians outside the study institution with expertise in adult pulmonary and critical care medicine clinical practice and clinical research, one bioethicist, and one biostatistician.

# Statistical Analysis Principles

R (R Foundation for Statistical Computing, Vienna, Austria) will be used for analyses. Analyses will be conducted at the level of an individual patient during an individual hospitalization in an intent-to-treat fashion, unless otherwise specified. Continuous variables will be reported as mean  $\pm$  SD or median and IQR; categorical variables will be reported as frequencies and proportions.

#### Main Analysis of the Primary Outcome

The main analysis will be an intention-to-treat comparison of the primary outcome of VFDs between the higher, intermediate, and lower SpO<sub>2</sub> target groups among all patients enrolled in the trial except [1] those admitted during one of the 7-day washout periods and [2] those with a laboratory-confirmed diagnosis of COVID-19.

Patients with a diagnosis of COVID-19 will be excluded from the main analysis for two reasons. First, the majority of the PILOT trial occurred prior the COVID-19 pandemic, with too few two-month study blocks occurring during the pandemic to ensure balance in the number of patients with COVID-19 between trial groups. Second, at the study hospital, ICU patients diagnosed with COVID-19 are transferred to a separate, dedicated COVID-19 ICU that was not participating in the PILOT trial. Thus, patients with COVID-19 are unlikely to have received significant exposure to the SpO<sub>2</sub> target intervention in the PILOT trial. Patients enrolled during washout periods and patients diagnosed with COVID-19 will be included in sensitivity analyses (see *Sensitivity Analyses* below).

It is possible to estimate a conditional effect, which is interpreted as the effect of a given SpO<sub>2</sub> target on an individual patient given the values of the covariates for that

patient, or a marginal effect, which is interpreted as the population effect of implementing a given SpO<sub>2</sub> target as a general policy [52]. Since an SpO<sub>2</sub> target intervention may be applied both at the patient level as an individual intervention and at the unit level as a general policy, both may be of interest.

To estimate the conditional effect, we will use a proportional odds model with independent covariates of group assignment (higher, intermediate, or lower SpO<sub>2</sub> target) and time [53,54]. Time (in days) will be treated as a continuous variable with values ranging from 1 (first day of enrollment) to 1,097 (final day of enrollment) and will be analyzed using restricted cubic splines with multiple knots to allow for non-linearity resulting from seasonality or secular trends. For the purposes of declaring a statistically significant difference between groups in the primary endpoint, we will consider the conditional effect from the proportional odds model and a two-sided P value of 0.05.

To estimate the marginal effect, we will use generalized estimating equations (GEE) with study period as the cluster and an independent variable for group assignment (higher, intermediate, or lower SpO<sub>2</sub> target).

For both approaches, in addition to assessing for an overall group effect within the model, we will estimate the differences between each pair of SpO<sub>2</sub> targets by extracting 95% confidence intervals from the model.

#### Sensitivity Analyses of the Primary Outcome

 We will repeat the primary analysis using alternative statistical approaches to comparing the VFDs outcome between groups such as zero-inflated Poisson

- regression or zero-inflated negative binomial regression, global rank scale analysis [55], and Fine and Gray competing risk regression.
- We will repeat the primary analysis with adjustment for pre-specified baseline covariates of age, sex, race and ethnicity, source of ICU admission, vasopressor receipt, and acute diagnoses at enrollment, and severity of illness as assessed by the non-respiratory SOFA score.
- We will repeat the primary analysis replacing the continuous covariate of time
  with a categorical covariate of season defined as: winter (January, February,
  March); spring (April, May, June); summer (July, August, September); and fall
  (October, November, December).
- We will repeat the primary analysis among all patients enrolled in the trial, including [1] patients initiated on invasive mechanical ventilation in a study location during one of the pre-specified 7-day washout periods and [2] patients with a diagnosis of COVID-19.

# Analysis of Effect Modification for the Primary Outcome

We will examine whether pre-specified baseline variables modify the effect of study group on the primary outcome using formal tests of statistical interaction in a proportional odds model. Independent variables will include study group assignment, the potential effect modifier of interest, and the interaction between the two (e.g., study group \* presence of sepsis or septic shock) and time. Significance will be determined by the P value for the interaction term, with values less than 0.10 considered to suggest a potential interaction and values less than 0.05 considered to confirm an interaction.

We will examine whether the following baseline variables modify the effect of study group on the primary outcome:

- 1. Age;
- 2. Race and ethnicity (Hispanic, Non-Hispanic Black, Non-Hispanic White, Other);
- Source of admission to the ICU (ED, hospital ward, another ICU in the study hospital, operating room, outside hospital);
- 4. Duration of invasive mechanical ventilation prior to enrollment;
- 5. Chronic comorbidities (categories are not mutually exclusive)
  - a. Receipt of supplemental oxygen at place of residence prior to hospital admission (yes, no);
  - b. Coronary artery disease or heart failure with reduced ejection fraction (yes, no);
- 6. Acute diagnoses at enrollment (categories are not mutually exclusive) [56]
  - a. cardiac arrest (yes, no);
  - b. acute myocardial infarction (yes, no);
  - c. sepsis or septic shock (yes, no);
  - d. acute respiratory distress syndrome (yes, no);
- 7. Receipt of vasopressors at enrollment (yes, no);
- 8. Non-respiratory SOFA score at enrollment;
- 9. Time period (before the COVID-19 pandemic [July 2018 December 2019], during the COVID-19 pandemic [January 2020 August 2021]).

The sole pre-specified secondary outcome of 28-day in-hospital mortality will be compared between the three study groups in an intention-to-treat fashion in the main analysis population using a logistic regression model with independent covariates of group assignment (higher, intermediate, or lower SpO<sub>2</sub> target) and time. In addition to assessing for an overall group effect within the model, we will estimate the differences between each pair of SpO<sub>2</sub> targets by extracting 95% confidence intervals from the model.

# Analysis of the Exploratory Outcomes

Each of the exploratory outcomes will be compared between groups in an intention-to-treat fashion in the main analysis population. Exploratory outcomes will be compared between study groups in a similar manner as for primary and secondary outcomes. A logistic model will be used for binary outcomes, a multinomial model for categorical outcomes, and a proportional odds model will be used for ordinal and continuous outcomes.

# Trial Status

PILOT is an ongoing pragmatic trial comparing higher, intermediate, and lower SpO<sub>2</sub> targets for mechanically ventilated critically ill adults. Patient enrollment began on July 1, 2018 and is anticipated to conclude on August 31, 2021.

# **Ethics and dissemination**

IRB Approval

The trial was approved by the Institutional Review Board (IRB) of Vanderbilt University Medical Center with a waiver of informed consent (IRB# 171272), details of which are provided in supplemental file 1, section 26. Participants who regain capacity to provide informed consent, or legally authorized surrogate decision-makers for those patients who do not regain the capacity to provide informed consent, are approached to provide informed consent for assessment of long-term outcomes as a part of the independently-funded Cognitive Outcomes in the Pragmatic Investigation of Optimal Oxygen Targets (CO-PILOT) study (R21AG063126).

#### Information for Patients and Families

An information sheet providing an IRB-approved lay language summary of the study and containing the contact information for investigators (who remain available throughout the study period to provide additional information to patients and families upon request) is made available throughout the study period in glass display cases near the public entrance to the ICU and near the center of the ICU, in the 'welcome packet' of information about the ICU, which is distributed at the time of ICU admission to patients, families, and surrogates by the medical receptionist or charge nurse as a part of routine admission processes, in a brochure holder in the family waiting room for the study ICU, and by treating physicians and respiratory therapist to any patients, families, or surrogates with questions or concerns about the study.

# Protocol Changes

Any changes to the trial protocol will be recorded on ClinicalTrials.Gov as per SPIRIT guidelines (see section 27 of supplemental file 1).

# Data Handling and Sharing

For details of privacy, data handling, and data sharing, see sections 28-29 of supplemental file 1.

#### Dissemination Plan

Trial results will be submitted to a peer-reviewed journal for consideration of publication and will be presented at scientific conferences. The results of the study will be disseminated to patients and the public at the completion of the trial.

Contributorship statement: Study concept and design: M.W.S., J.D.C., C.J.L., G.R.B., W.H.S., T.W.R.; Drafting of the manuscript: M.W.S., L.W., C.J.L.; Critical revision of the manuscript for important intellectual content: M.W.S., J.D.C., B.D.L., P.G.H., M.A.H., M.R., J.L.S., J.H.B., K.G.B., L.W., C.J.L., R.E.F., J.P.W., G.R.B., W.H.S., T.W.R; Statistical analysis: L.W., C.J.L.; Study supervision: G.R.B., W.H.S., T.W.R.

**Conflicts of Interest:** All authors completed and submitted the ICMJE Form for Disclosure of Potential Conflicts of Interest. R.E.F. reported receiving grant funding and consulting fees from Medtronic and stock from 3M outside the current work. T.W.R.

reported receiving consulting fees from Cumberland Pharmaceuticals outside the current work. The authors declared no potential conflicts of interest with the current work.

Funding: This study was supported in part by a grant from the National Heart Lung and Blood Institute (K23HL143053). J.D.C was supported in part by the NIH (K23HL153584). R.E.F. was supported in part by the NIH (1KL2TR002245, 1K23HL148640). T.W.R. was supported in part by the NIH (U01HL123033, UL1TR002244). Data collection used the Research Electronic Data Capture (REDCap) tool developed and maintained with Vanderbilt Institute for Clinical and Translational Research grant support (UL1 TR000445 from the National Center for Advancing Translational Sciences). The funding institutions had no role in (1) conception, design, or conduct of the study, (2) collection, management, analysis, interpretation, or presentation of the data, or (3) preparation, review, or approval of the manuscript.

#### **REFERENCES**

- 1 Wunsch H, Linde-Zwirble WT, Angus DC, et al. The epidemiology of mechanical ventilation use in the United States. Crit Care Med 2010;38:1947–53. doi:10.1097/CCM.0b013e3181ef4460
- Wunsch H, Angus DC, Harrison DA, et al. Comparison of medical admissions to intensive care units in the United States and United Kingdom. Am J Respir Crit Care Med 2011;183:1666–73. doi:10.1164/rccm.201012-1961OC
- Adhikari NKJ, Fowler RA, Bhagwanjee S, et al. Critical care and the global burden of critical illness in adults. Lancet Lond Engl 2010;376:1339–46. doi:10.1016/S0140-6736(10)60446-1
- 4 Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. The Acute Respiratory Distress Syndrome Network. *N Engl J Med* 2000;**342**:1301–8. doi:10.1056/NEJM200005043421801
- Esteban A, Frutos-Vivar F, Muriel A, et al. Evolution of mortality over time in patients receiving mechanical ventilation. *Am J Respir Crit Care Med* 2013;**188**:220–30. doi:10.1164/rccm.201212-2169OC
- 6 Fridovich I. Oxygen toxicity: a radical explanation. *J Exp Biol* 1998;**201**:1203–9.
- Heffner JE, Repine JE. Pulmonary strategies of antioxidant defense. *Am Rev Respir Dis* 1989;**140**:531–54. doi:10.1164/ajrccm/140.2.531
- 8 Freeman BA, Crapo JD. Hyperoxia increases oxygen radical production in rat lungs and lung mitochondria. *J Biol Chem* 1981;**256**:10986–92.
- 9 Waxman AB, Einarsson O, Seres T, et al. Targeted lung expression of interleukin-11 enhances murine tolerance of 100% oxygen and diminishes hyperoxia-induced DNA fragmentation. *J Clin Invest* 1998;**101**:1970–82. doi:10.1172/JCl1337
- 10 Griffith DE, Garcia JG, James HL, et al. Hyperoxic exposure in humans. Effects of 50 percent oxygen on alveolar macrophage leukotriene B4 synthesis. *Chest* 1992;**101**:392–7.
- 11 Davis WB, Rennard SI, Bitterman PB, et al. Pulmonary oxygen toxicity. Early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med 1983;309:878–83. doi:10.1056/NEJM198310133091502
- 12 Aggarwal NR, Brower RG. Targeting normoxemia in acute respiratory distress syndrome may cause worse short-term outcomes because of oxygen toxicity. *Ann Am Thorac Soc* 2014;**11**:1449–53. doi:10.1513/AnnalsATS.201407-297PS
- 13 Meade MO, Cook DJ, Guyatt GH, et al. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. *JAMA J Am Med Assoc* 2008;**299**:637–45. doi:10.1001/jama.299.6.637

- 14 Eastwood G, Bellomo R, Bailey M, et al. Arterial oxygen tension and mortality in mechanically ventilated patients. *Intensive Care Med* 2012;**38**:91–8. doi:10.1007/s00134-011-2419-6
- de Jonge E, Peelen L, Keijzers PJ, *et al.* Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. *Crit Care Lond Engl* 2008;**12**:R156. doi:10.1186/cc7150
- Allen BS, Ilbawi MN. Hypoxia, reoxygenation and the role of systemic leukodepletion in pediatric heart surgery. *Perfusion* 2001;**16 Suppl**:19–29. doi:10.1177/026765910101600i104
- 17 Allen BS. The reoxygenation injury: is it clinically important? *J Thorac Cardiovasc Surg* 2002;**124**:16–9.
- 18 Supplemental Therapeutic Oxygen for Prethreshold Retinopathy Of Prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. *Pediatrics* 2000;**105**:295–310.
- 19 SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network, Carlo WA, Finer NN, et al. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med 2010;**362**:1959–69. doi:10.1056/NEJMoa0911781
- 20 Schmidt B, Whyte RK, Asztalos EV, et al. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. *JAMA* 2013;**309**:2111–20. doi:10.1001/jama.2013.5555
- 21 BOOST II United Kingdom Collaborative Group, BOOST II Australia Collaborative Group, BOOST II New Zealand Collaborative Group, *et al.* Oxygen saturation and outcomes in preterm infants. *N Engl J Med* 2013;**368**:2094–104. doi:10.1056/NEJMoa1302298
- 22 Panwar R, Hardie M, Bellomo R, *et al.* Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. *Am J Respir Crit Care Med* 2016;**193**:43–51. doi:10.1164/rccm.201505-10190C
- 23 Asfar P, Schortgen F, Boisramé-Helms J, et al. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med Published Online First: February 2017. doi:10.1016/S2213-2600(17)30046-2
- 24 Girardis M, Busani S, Damiani E, *et al.* Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. *JAMA* 2016;**316**:1583–9. doi:10.1001/jama.2016.11993
- 25 Barrot L, Asfar P, Mauny F, et al. Liberal or Conservative Oxygen Therapy for Acute Respiratory Distress Syndrome. *N Engl J Med* 2020;**382**:999–1008. doi:10.1056/NEJMoa1916431
- 26 ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group, Mackle D, Bellomo R, *et al.* Conservative Oxygen Therapy during Mechanical Ventilation in the ICU. *N Engl J Med* Published Online First: 14 October 2019. doi:10.1056/NEJMoa1903297

- 27 Schjørring OL, Klitgaard TL, Perner A, et al. Lower or Higher Oxygenation Targets for Acute Hypoxemic Respiratory Failure. N Engl J Med Published Online First: 20 January 2021. doi:10.1056/NEJMoa2032510
- 28 Siemieniuk RAC, Chu DK, Kim LH-Y, *et al.* Oxygen therapy for acutely ill medical patients: a clinical practice guideline. *BMJ* 2018;**363**:k4169. doi:10.1136/bmj.k4169
- 29 National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network, Rice TW, Wheeler AP, et al. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. *JAMA J Am Med Assoc* 2012;**307**:795–803. doi:10.1001/jama.2012.137
- 30 Rice TW, Wheeler AP, Thompson BT, et al. Enteral omega-3 fatty acid, gamma-linolenic acid, and antioxidant supplementation in acute lung injury. *JAMA J Am Med Assoc* 2011;**306**:1574–81. doi:10.1001/jama.2011.1435
- 31 O'Driscoll BR, Howard LS, Earis J, *et al.* BTS guideline for oxygen use in adults in healthcare and emergency settings. *Thorax* 2017;**72**:ii1–90. doi:10.1136/thoraxjnl-2016-209729
- 32 Panwar R, Capellier G, Schmutz N, et al. Current oxygenation practice in ventilated patients-an observational cohort study. *Anaesth Intensive Care* 2013;**41**:505–14.
- 33 Suzuki S, Eastwood GM, Peck L, *et al.* Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. *J Crit Care* 2013;**28**:647–54. doi:10.1016/j.jcrc.2013.03.010
- 34 Helmerhorst HJ, Schultz MJ, van der Voort PH, *et al.* Self-reported attitudes versus actual practice of oxygen therapy by ICU physicians and nurses. *Ann Intensive Care* 2014;**4**:23. doi:10.1186/s13613-014-0023-y
- 35 Self WH, Semler MW, Rice TW. Oxygen Targets for Patients Who Are Critically III: Emerging Data and State of Equipoise. *Chest* 2020;**157**:487–8. doi:10.1016/j.chest.2019.12.010
- 36 SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. PubMed NCBI. https://www.ncbi.nlm.nih.gov/pubmed/23303884 (accessed 8 Jan 2018).
- 37 Ware JH, Hamel MB. Pragmatic Trials Guides to Better Patient Care? *N Engl J Med* 2011;**364**:1685–7. doi:10.1056/NEJMp1103502
- 38 Beasley R, Chien J, Douglas J, *et al.* Thoracic Society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: 'Swimming between the flags.' *Respirol Carlton Vic* 2015;**20**:1182–91. doi:10.1111/resp.12620
- 39 Brower RG, Lanken PN, MacIntyre N, et al. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med 2004;**351**:327–36. doi:10.1056/NEJMoa032193

- 40 Briel M, Meade M, Mercat A, *et al.* Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. *JAMA J Am Med Assoc* 2010;**303**:865–73. doi:10.1001/jama.2010.218
- 41 Semler MW, Rice TW, Shaw AD, et al. Identification of Major Adverse Kidney Events Within the Electronic Health Record. *J Med Syst* 2016;**40**:167. doi:10.1007/s10916-016-0528-z
- 42 Semler MW, Noto MJ, Stollings J, et al. Effect Of Saline Versus Balanced Crystalloids On Major Adverse Kidney Events In The Medical Intensive Care Unit: The Salt Randomized Trial. Am J Respir Crit Care Med 2016;**193**:A4290.
- 43 Semler MW, Self WH, Wang L, et al. Balanced crystalloids versus saline in the intensive care unit: study protocol for a cluster-randomized, multiple-crossover trial. *Trials* 2017;**18**. doi:10.1186/s13063-017-1871-1
- 44 Harris PA, Taylor R, Thielke R, et al. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. *J Biomed Inform* 2009;**42**:377–81. doi:10.1016/j.jbi.2008.08.010
- 45 Schoenfeld DA, Bernard GR. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. *Crit Care Med* 2002;**30**:1772–7.
- 46 Harhay MO, Wagner J, Ratcliffe SJ, et al. Outcomes and statistical power in adult critical care randomized trials. Am J Respir Crit Care Med 2014;**189**:1469–78. doi:10.1164/rccm.201401-0056CP
- 47 Vincent JL, Moreno R, Takala J, et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. *Intensive Care Med* 1996;**22**:707–10.
- 48 ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, *et al.* Acute respiratory distress syndrome: the Berlin Definition. *JAMA J Am Med Assoc* 2012;**307**:2526–33. doi:10.1001/jama.2012.5669
- 49 Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury. *Kidney inter* 2012;**2(Suppl)**:8.
- 50 Thygesen K, Alpert JS, Jaffe AS, et al. Fourth Universal Definition of Myocardial Infarction (2018). *J Am Coll Cardiol* 2018;**72**:2231–64. doi:10.1016/j.jacc.2018.08.1038
- 51 Semler MW, Self WH, Wanderer JP, et al. Balanced Crystalloids versus Saline in Critically III Adults. *N Engl J Med* 2018;**378**:829–39. doi:10.1056/NEJMoa1711584
- 52 Zeger SL, Liang KY, Albert PS. Models for longitudinal data: a generalized estimating equation approach. *Biometrics* 1988;**44**:1049–60.
- 53 Turner RM, White IR, Croudace T, et al. Analysis of cluster randomized cross-over trial data: a comparison of methods. *Stat Med* 2007;**26**:274–89. doi:10.1002/sim.2537

- Parienti J-J, Kuss O. Cluster-crossover design: a method for limiting clusters level effect in community-intervention studies. *Contemp Clin Trials* 2007;**28**:316–23. doi:10.1016/j.cct.2006.10.004
- 55 Beitler JR, Sarge T, Banner-Goodspeed VM, et al. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. *JAMA* Published Online First: 18 2019. doi:10.1001/jama.2019.0555
- 56 Munshi L, Ferguson ND. Evolving Issues in Oxygen Therapy in Acute Care Medicine. *JAMA* Published Online First: 24 January 2020. doi:10.1001/jama.2019.22029

# **FIGURES**

Figure 1. Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) checklist. Enrollment, Interventions, and Assessments.

Figure 2. Group assignment during the trial. For each of the 18 two-month study periods, the study ICU is randomly assigned to a higher, intermediate, or lower SpO<sub>2</sub> target. In this figure, the letters "A", "B", and "C" each correspond to one of the three possible SpO<sub>2</sub> targets, the allocation sequence of which remains concealed until the start of each two-month study period. The study did not enroll in April and May of 2020 due to disruptions in research and clinical care from the Coronavirus Infectious Disease 2019 (COVID-19) pandemic. As a result, March and June of 2020 represent a single-two-month block assigned to one SpO<sub>2</sub> target.

# **TABLES**

Table 1. SpO<sub>2</sub> and PaO<sub>2</sub> targets and goal ranges by study group.

| Study Group | SpO <sub>2</sub> target | SpO <sub>2</sub> goal range | PaO <sub>2</sub> target | PaO <sub>2</sub> goal range |
|---|---|---|---|---|
| Lower SpO <sub>2</sub> target | 90% | 88-92% | 60 mm Hg | 55-65 mm Hg |
| Intermediate SpO <sub>2</sub> target | 94% | 92-96% | 70 mm Hg | 65-80 mm Hg |
| Higher SpO <sub>2</sub> target | 98% | 96-100% | 110 mm Hg | > 80 mm Hg |

For each study group, the SpO<sub>2</sub> target and goal range are displayed. PaO<sub>2</sub> is used to guide titration of FiO<sub>2</sub> for participants without functioning pulse oximetry monitoring.

# BMJ Open Protocol and statistical analysis plan for the Pragmatic Investigation of optimaL Oxygen Targets (PILOT) clinical trial

Matthew W Semler , 1 Jonathan D Casey, 1 Bradley D. Lloyd, 2 Pamela G. Hastings,<sup>2</sup> Margaret Hays,<sup>1</sup> Megan Roth,<sup>1</sup> Joanna Stollings,<sup>3</sup> John Brems,<sup>4</sup> Kevin George Buell,<sup>4</sup> Li Wang,<sup>5</sup> Christopher J. Lindsell,<sup>5</sup> Robert E. Freundlich,<sup>6</sup> Jonathan P. Wanderer,<sup>6</sup> Gordon R. Bernard,<sup>1</sup> Wesley H. Self,<sup>7</sup> Todd W. Rice. The PILOT Investigators and the Pragmatic Critical Care Research Group

To cite: Semler MW. Casev JD. Lloyd BD, et al. Protocol and statistical analysis plan for the Pragmatic Investigation of optimaL Oxygen Targets (PILOT) clinical trial. BMJ Open 2021;11:e052013. doi:10.1136/ bmjopen-2021-052013

Prepublication history and additional supplemental material for this paper are available online. To view these files, please visit the journal online (http://dx.doi.org/10.1136/ bmjopen-2021-052013).

Received 05 April 2021 Accepted 12 October 2021

# **ABSTRACT**

Introduction Mechanical ventilation of intensive care unit (ICU) patients universally involves titration of the fraction of inspired oxygen to maintain arterial oxygen saturation (SpO<sub>2</sub>). However, the optimal SpO<sub>2</sub> target remains unknown.

Methods and analysis The Pragmatic Investigation of optimaL Oxygen Targets (PILOT) trial is a prospective, unblinded, pragmatic, cluster-crossover trial being conducted in the emergency department (ED) and medical ICU at Vanderbilt University Medical Center in Nashville. Tennessee, USA. PILOT compares use of a lower SpO. target (target 90% and goal range: 88%-92%), an intermediate SpO<sub>2</sub> target (target 94% and goal range: 92%-96%) and a higher SpO<sub>2</sub> target (target 98% and goal range: 96%-100%). The study units are assigned to a single SpO<sub>2</sub> target (cluster-level allocation) for each 2-month study block, and the assigned SpO<sub>2</sub> target switches every 2 months in a randomly generated sequence (cluster-level crossover). The primary outcome is ventilator-free days (VFDs) to study day 28, defined as the number of days alive and free of invasive mechanical ventilation from the final receipt of invasive mechanical ventilation through 28 days after enrolment.

Ethics and dissemination The trial was approved by the Vanderbilt Institutional Review Board. The results will be submitted for publication in a peer-reviewed journal and presented at one or more scientific conferences.

Trial registration number The trial protocol was registered with ClinicalTrials.gov on 25 May 2018 prior to initiation of patient enrolment (ClinicalTrials.gov identifier: NCT03537937).

# Check for updates

@ Author(s) (or their employer(s)) 2021. Re-use permitted under CC BY-NC. No commercial re-use. See rights and permissions. Published by

For numbered affiliations see end of article.

#### **Correspondence to**

Dr Matthew W Semler: matthew.w.semler@vumc.org

# INTRODUCTION

Each year 2-3 million intensive care unit (ICU) patients receive invasive mechanical ventilation. 1-3 Despite recent advances in lung-protective ventilation,4 in-hospital mortality among mechanically ventilated ICU patients remains 25%-35%.5

Mechanical ventilation for ICU patients universally involves titrating the fraction of

### Strengths and limitations of this study

- ► This ongoing pragmatic trial will provide information on the optimal oxygen saturation target during invasive mechanical ventilation of critically ill adultsinforming a common therapy in current clinical practice for which there is limited available evidence on which to base care.
- Broad inclusion criteria will increase generalisability and the sample size will allow examination of important patient subgroups.
- The trial is being conducted at a single centre.
- The nature of the study intervention does not allow
- Decisions regarding oxygen administration before and after invasive mechanical ventilation are deferred to treating clinicians.

inspired oxygen (FiO<sub>9</sub>) to maintain arterial oxygen saturation (SpO<sub>9</sub>) within a goal range. Despite decades of ICU practice, however, the optimal SpO<sub>9</sub> target remains unknown. Higher SpO<sub>9</sub> targets (96%–100%) provide a margin of safety against hypoxaemia, but may increase exposure to excess FiO<sub>9</sub>, hyperoxaemia, and tissue hyperoxia, causing oxidative damage, 6-8 inflammation 9 10 and increased alveolar-capillary permeability.<sup>11</sup> Lower SpO<sub>9</sub> targets (88%–92%) minimise exposure to excess FiO<sub>2</sub>, hyperoxaemia and tissue hyperoxia, 4 12 13 but may increase the risk of hypoxaemia and tissue hypoxia. 14 15 An intermediate SpO<sub>9</sub> target (92%-96%) may avoid the risks of both hyperoxia and hypoxia or, conversely, may expose patients intermittently to both sets of risks. 16 17

The relative risks and benefits of different SpO<sub>9</sub> or PaO<sub>9</sub> targets have been extensively examined in the setting of the neonatal ICU<sup>18-21</sup> and have been examined among



adult ICU patients in a series of recently published clinical trials. Together, these trials have suggested that both higher and lower oxygenation targets are safe—although some trials have potentially suggested better outcomes with higher targets and other trials have suggested potentially better outcomes with lower targets.

Given the still incomplete evidence from randomised trials, current guidelines offer divergent recommendations—ranging from tolerating  ${\rm SpO_2}$  values as low as  $88\%^{28-30}$  to pursuing  ${\rm SpO_2}$  values as high as  $98\%.^{31}$  In clinical practice, hyperoxaemia remains common,  $^{32}$   $^{33}$  even among patients cared for by clinicians who self-identify as avoiding high oxygen levels.  $^{34}$ 

The wide variation in current practice, conflicting guidelines and conflicting data from some available trials indicate the need for further clinical trials to determine the effect of  $\mathrm{SpO}_2$  target on patient outcomes. <sup>12 35</sup> We designed the Pragmatic Investigation of optimaL Oxygen Targets (PILOT) trial to examine the effects of higher, intermediate and lower  $\mathrm{SpO}_2$  targets on the number of days alive and free of invasive mechanical ventilation among mechanically ventilated ICU patients.

#### **METHODS AND ANALYSIS**

This manuscript was prepared by the PILOT investigators (online supplemental file 1, section 1) in accordance with Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines (figure 1; SPIRIT checklist in online supplemental file 1, section 2). 36 This manuscript describes key elements of the trial protocol and statistical analysis plan. The supplemental methods in online supplemental file 1 provide additional background on prior trials (section 3), rationale for design decisions (sections 4–5), SpO<sub>0</sub> monitoring and management (sections 6-8), institutional protocols for mechanical ventilation (sections 9-17), a complete list of data elements (section 18), definitions of exploratory outcomes and measures of separation between groups (sections 19-21), and details of the interim analysis (section 22) and secondary analyses (sections 23–25).

#### Study design

The PILOT trial is a prospective, unblinded, pragmatic, cluster-crossover trial being conducted in the ED and medical ICU at Vanderbilt University Medical Center in Nashville, Tennessee, USA. PILOT compares use of a

| | STUDY PERIOD | | | |
|---|---|---|---|---|
| | Allocation and<br>Enrollment | On-S | Study<br>Termination | |
| TIMEPOINT | First receipt of<br>invasive mechanical<br>ventilation in a<br>study location | Receiving<br>invasive<br>mechanical<br>ventilation in<br>study location | Hospitalized but<br>not receiving<br>invasive<br>mechanical<br>ventilation in a<br>study location | Discharge or 28<br>days after<br>enrolment |
| ENROLMENT: | X | | | |
| Eligibility screen | X | | | |
| Allocation | Х | | | |
| INTERVENTIONS: | | | | |
| Higher SpO2 Target Titrating FiO2 to SpO2 96-100% | Х | X | | |
| Intermediate SpO2 Target<br>Titrating FiO2 to SpO2 92-96% | X | X | | |
| Lower SpO2 Target Titrating FiO2 to SpO2 88-92% | X | X | | |
| Screening for indications for<br>SpO2 target modification | X | X | | |
| ASSESSMENTS: | | | | |
| Baseline Variables | Х | | | |
| On-study Variables | Х | Х | Х | |
| Clinical Outcomes | | | | Х |

**Figure 1** Standard Protocol Items: Recommendations for Interventional Trials checklist. Enrolment, interventions and assessments. FiO<sub>2</sub>, fraction of inspired oxygen; SpO<sub>2</sub>, arterial oxygen saturation.

lower SpO<sub>9</sub> target (target 90% and goal range: 88%–92%), an intermediate SpO<sub>9</sub> target (target 94% and goal range: 92%–96%) and a higher SpO<sub>9</sub> target (target 98% and goal range: 96%-100%) with regard to the number of days alive and free of invasive mechanical ventilation among mechanically ventilated ICU patients. Consistent with the concept of a pragmatic clinical trial,<sup>37</sup> the eligibility criteria are broad, the delivery of the intervention is embedded in routine clinical care and executed by clinical personnel, and data collection prioritises clinical outcomes over mechanistic evaluation. The trial was approved by the Vanderbilt University Medical Center Institutional Review Board (IRB 171272). The trial is investigator initiated with funding provided by the National Heart, Lung, and Blood Institute (K23HL143053). The trial protocol was registered with ClinicalTrials.gov on 25 May 2018 prior to initiation of patient enrolment on 1 July 2018 (ClinicalTrials.gov identifier: NCT03537937).

#### Patient and public involvement

Materials used to communicate about the study with patients and families were developed with input from the Vanderbilt Community Engaged Research Core and the Vanderbilt Community Advisory Council.

#### Study site and population

The trial is being conducted in the adult ED and medical ICU at Vanderbilt University Medical Center.

#### The inclusion criteria are

- 1. Age ≥18 years.
- 2. Receiving mechanical ventilation through an endotracheal tube or tracheostomy.
- 3. Admitted to the study ICU or admission to the study ICU from the ED is planned.

#### The exclusion criteria are

- 1. Known pregnancy or beta-human chorionic gonadotropin level greater than the laboratory upper limit of normal in a patient capable of becoming pregnant (if measured clinically).
- 2. Known to be a prisoner.

Adults located in the study ICU or for whom admission to the study ICU from the ED is planned who meet inclusion criteria and do not meet exclusion criteria are enrolled immediately on receipt of invasive mechanical

ventilation in a study location. The time of enrolment for the trial ('time zero') is the time of first receipt of invasive mechanical ventilation in a participating study location.

#### **Randomisation and treatment allocation**

For each of the 18 2-month blocks during the 36 months of enrolment in the PILOT trial, the medical ICU is assigned to a single SpO<sub>9</sub> target (cluster-level allocation). Every 2 months, the ICU will switch between use of a lower SpO<sub>9</sub> target (target 90% and goal range: 88%–92%), use of an intermediate SpO<sub>2</sub> target (target 94% and goal range: 92%-96%) and use of a higher SpO<sub>9</sub> target (target 98% and goal range: 96%–100%) in a randomly generated sequence (cluster-level crossover) (figure 2). The order of study group assignments for each 2-month block was generated by computerised randomisation using permuted blocks of three to minimise the impact of seasonal variation and temporal changes. For the 36 months of enrolment in the PILOT trial, patients receiving invasive mechanical ventilation in the ED for whom admission to the medical ICU is planned will receive the same SpO<sub>9</sub> target assigned to the medical ICU. The study did not enrol in April and May of 2020 due to disruptions in research and clinical care from the COVID-19 pandemic (figure 2).

#### **Washout periods**

The last 7 days of each 2-month block are considered an analytic washout period during which the ICU continues to target the assigned SpO<sub>9</sub>, but data from new patients are not included in the primary analysis. Assuming a median duration of mechanical ventilation of 3 (IQR: 3–5) days, a 7-day washout period will ensure that 98% patients in the primary analysis do not experience a 'crossover' from a period assigned to one assigned SpO<sub>9</sub> target to a period assigned to another SpO<sub>9</sub> target. Data from patients admitted during washout periods will be included in a prespecified sensitivity analysis (see Statistical analysis section). Any patient who does remain mechanically ventilated in the study ICU through a crossover from a period assigned to one SpO<sub>9</sub> target to a period assigned to another SpO<sub>9</sub> target will be analysed in the SpO<sub>9</sub> target group to which the ICU was assigned at the time of the patient's enrolment in the trial (intentionto-treat analysis).

| Study Year 1 | | | | | Study Year 2 | | | | Study Year 3 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug | Sep-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar<br>& Jun | Jul-<br>Aug | Sept-<br>Oct | Nov-<br>Dec | Jan-<br>Feb | Mar-<br>Apr | May-<br>Jun | Jul-<br>Aug |
| | 2018 20 | | | 19 | | | 2020 | | | | | | 20 | 21 | | | |
| А | В | С | В | С | Α | С | В | Α | Α | В | С | В | Α | С | В | Α | С |

Figure 2 Group assignment during the trial. For each of the 18 2-month study periods, the study intensive care unit is randomly assigned to a higher, intermediate or lower SpO<sub>2</sub> target. in this figure, The letters 'A', 'B' and 'C' each correspond to one of the three possible SpO2 targets, the allocation sequence of which remains concealed until the start of each 2-month study period. The study did not enrol in April and May of 2020 due to disruptions in research and clinical care from the COVID-19 pandemic. As a result, March and June of 2020 represent a single 2-month block assigned to one SpO, target. SpO, arterial oxygen saturation.

Table 1 SpO<sub>2</sub> and PaO<sub>3</sub> targets and goal ranges by study group

| Study group | SpO <sub>2</sub> target | SpO <sub>2</sub> goal range | PaO <sub>2</sub> target (mm<br>Hg) | PaO <sub>2</sub> goal range<br>(mm Hg) |
|---|---|---|---|---|
| Lower SpO <sub>2</sub> target | 90% | 88%-92% | 60 | 55–65 |
| Intermediate SpO <sub>2</sub> target | 94% | 92%-96% | 70 | 65–8 |
| Higher SpO <sub>2</sub> target | 98% | 96%-100% | 110 | >80 |

For each study group, the  $SpO_2$  target and goal range are displayed.  $PaO_2$  is used to guide titration of  $FiO_2$  for participants without reliable pulse oximetry monitoring.

FiO,, fraction of inspired oxygen; PaO,, arterial oxygen tension; SpO,, arterial oxygen saturation.

#### **Study interventions**

#### Choice of SpO<sub>2</sub> targets

In clinical practice, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adults fall between 88% and 100%. <sup>32</sup> <sup>33</sup> Within this range, current guidelines for oxygen therapy in mechanically ventilated adults outline three contrasting approaches: (1) allowing the lower end of the range of acceptable SpO<sub>2</sub> values to be as low as 88% <sup>28</sup> <sup>29</sup> to avoid excess FiO<sub>2</sub>, hyperoxaemia and hyperoxia; (2) titrating within an intermediate range of SpO<sub>2</sub> values, such as 92%–96% <sup>38</sup>; or (3) targeting higher SpO<sub>2</sub> to avoid the risks of hypoxaemia and hypoxia. <sup>31</sup> The PILOT trial has three study groups, each emulating a different approach to SpO<sub>2</sub> targets represented in guidelines and clinical practice (table 1).

#### Oxygen titration

In the study ED and ICU, titration of  $\mathrm{FiO}_2$  to maintain  $\mathrm{SpO}_2$  for mechanically ventilated adults is typically performed by respiratory therapists with input from nurses and physicians. In preparation for the PILOT trial, we collaborated with respiratory therapy leaders in the study ED and ICU to adapt existing ventilator management protocols to provide guidance for respiratory therapists in titrating  $\mathrm{FiO}_2$  to achieve each of the three study  $\mathrm{SpO}_2$  targets.

For patients enrolled in the study, respiratory therapists are instructed to begin titrating FiO<sub>9</sub> to the target SpO<sub>9</sub> value within 15 min of the initiation of mechanical ventilation. During the maintenance of invasive mechanical ventilation, SpO<sub>9</sub> is assessed by continuous pulse oximetry. The protocol directs the respiratory therapist managing the patient's ventilator to target an SpO<sub>9</sub> value of 90% in the lower SpO<sub>9</sub> target group, an SpO<sub>9</sub> value of 94% in the intermediate SpO<sub>9</sub> target group and an SpO<sub>9</sub> value of 98% in the higher SpO<sub>9</sub> target group (table 1). Respiratory therapists and other treating clinicians titrate FiO, when the SpO, is out of the goal range, when the SpO<sub>9</sub> is within the goal range but closer alignment with the assigned SpO<sub>9</sub> target is desired, to facilitate weaning from mechanical ventilation, or for other clinical indications. SpO<sub>9</sub> is reassessed 5 min after each change in FiO<sub>9</sub> or sooner if clinically indicated.

The protocol determines the  $SpO_2$  target from enrolment until the first of: (1) discontinuation of invasive mechanical ventilation, (2) transfer out of a participating

study location, (3) completion of an  $SpO_2$  target modification sheet by treating clinicians or (4) end of the 2-month study period. The protocol does not determine the  $SpO_2$  target during time periods in which the patient is not physically located in a study location (eg, during transport) or when  $FiO_2$  is being administered for purposes other than achieving a target  $SpO_2$  (eg, when an  $FiO_2$  of 1.0 is being administered for a procedure).

At any time, if a treating clinician or a patient, family member or surrogate feels that an SpO<sub>9</sub> target other than that assigned by the study would be best for the optimal treatment of the patient for any reason, the SpO<sub>9</sub> target for that patient is modified. To modify the target, the respiratory therapist and supervising physician complete a one-page SpO<sub>o</sub> target modification sheet documenting the new SpO<sub>9</sub> target and the rationale for modifying the target. Examples of conditions for which the assigned SpO<sub>9</sub> target may be modified that were specified in the initial trial protocol included pneumothorax, pneumomediastinum, carbon monoxide poisoning, decompression sickness, bleomycin toxicity and paraquat toxicity. Examples of conditions for which the assigned SpO<sub>9</sub> target may be modified that were not explicitly specified in the initial trial protocol include severe chronic obstructive pulmonary disease, severe acute respiratory distress syndrome, severe anaemia, status post lung transplantation and receipt of extracorporeal membrane oxygenation support. Trial protocol directs only the titration of FiO<sub>9</sub> to the assigned SpO<sub>9</sub> target. Other aspects of invasive mechanical ventilation, such as tidal volume, <sup>4</sup> positive end-expiratory pressure<sup>39 40</sup> and use of rescue therapies for hypoxaemia, are determined by institutional protocols and treating clinicians (see sections 9-17 of online supplemental file 1).

#### **Blinding**

Similar to prior studies of  ${\rm SpO_2}$  targets among critically ill adults, <sup>22 24 26</sup> patients and clinicians will not be blinded to study group assignment.

#### **Data collection**

The PILOT trial uses data collected by two methods to minimise observer bias: (1) manual data collection by study personnel and (2) automated collection of structured data recorded in routine clinical care, exported daily from the institution's electronic health record and patient registration, billing and laboratory clinical information systems into an Enterprise Data Warehouse. We have previously validated the quality of the automated method of data collection against the reference standard of two-physician manual chart review<sup>41</sup> and have employed this approach for the conduct of prior pragmatic trials. Data are stored, curated and secured in REDCap. EDCap.

# **Outcomes**

#### Primary outcome

The primary outcome is VFDs to study day 28. VFDs will be defined as the number of whole calendar days alive and free of invasive mechanical ventilation beginning at midnight on the day of the final receipt of invasive mechanical ventilation through day 28 after enrolment. 45 46 Outcome ascertainment will cease at the time of hospital discharge or 28 days after enrolment, whichever occurs first. Receipt of invasive mechanical ventilation will be considered to end when patients undergo the final tracheal extubation or disconnection of the ventilator from the endotracheal tube or tracheostomy tube between enrolment and 28 days after enrolment. Patients whose final receipt of invasive mechanical ventilation occurs on the day of enrolment will receive 27 VFDs. Patients who continue to receive invasive mechanical ventilation 28 days after enrolment will receive 0 VFDs. Patients who die prior to day 28 will receive 0 VFDs. Patients who are discharged from the hospital prior to day 28 and are receiving invasive mechanical ventilation at the time of discharge will receive 0 VFDs. Patients who are removed from invasive mechanical ventilation and are discharged from the hospital without invasive mechanical ventilation prior to 28 days will be assumed to remain free of invasive mechanical ventilation between hospital discharge and day 28. For patients who are removed from invasive mechanical ventilation, return to invasive mechanical ventilation, and are subsequently removed again from invasive mechanical ventilation prior to day 28, VFDs will be counted from the final receipt of invasive mechanical ventilation prior to day 28.

#### Secondary outcome

The sole prespecified secondary outcome is 28-day in-hospital mortality, defined as death from any cause between enrolment and the first of hospital discharge or 28 days after enrollment.

#### **Exploratory clinical outcomes**

- 1. ICU mortality—death in the ICU between enrolment and the first of 28 days after enrolment or hospital discharge
- 2. Free-day outcomes—defined as whole calendar days from last receipt of therapy until 28 days (online supplemental file 1, section 19)
  - i. Vasopressor-free days
  - ii. Renal replacement therapy-free days
  - iii. ICU-free days

#### v. Hospital-free days

#### Exploratory organ function outcomes

- Daily non-respiratory Sequential Organ Failure Assessment (SOFA) score (online supplemental table S1)<sup>47</sup>
- 2. Plasma creatinine concentration (mg/dL)
- 3. Plasma lactate concentration (mmol/L)
- 4. Presence of a cute respiratory distress syndrome by Berlin criteria  $^{48}\,$
- Stage II or greater acute kidney injury (AKI) by Kidney Disease: Improving Global Outcomes creatinine criteria.<sup>49</sup>

#### **Exploratory safety outcomes**

- 1. Atrial arrhythmia
- 2. Ventricular arrhythmia
- 3. Cardiac arrest with return of spontaneous circulation
- 4. Pneumothorax or pneumomediastinum
- 5. Ischaemic stroke
- 6. Myocardial infarction<sup>50</sup>

#### Additional long-term patientimportant outcomes

The independently funded Cognitive Outcomes in the Pragmatic Investigation of Optimal Oxygen Targets (CO-PILOT) study (R21AG063126) will assess cognitive, physical and psychological outcomes at 12 months after enrolment in the PILOT trial. The protocol and statistical analysis plan for the CO-PILOT study will be published separately.

#### Statistical analysis and reporting

#### Sample size estimation and power calculation

In a prior cluster-randomised cluster-crossover trial in the same ICU,<sup>51</sup> 880 mechanically ventilated adults were enrolled per year (73.3 per month), with a median of 22 VFDs (IQR: 0-25 VFDs) and an intracluster intraperiod correlation of 0.01. We estimate 2640 mechanically ventilated adults will be admitted to the study ICU during the 36-month PILOT trial, of whom 390 will be excluded from the primary analysis for initial receipt of invasive mechanical ventilation in a study location during a washout period and 2250 will be enrolled and included in the primary analysis. With a total enrolment of 2250 patients, a SD in the primary outcome of VFDs of 11.4 days, and a two-sided alpha of 0.05, we calculated using a t-test that the PILOT trial will have 92% statistical power to detect an absolute reduction in VFDs of 2.0 days (similar to the numerical difference in VFDs between SpO<sub>9</sub> target groups reported in prior studies<sup>22 24</sup>).

# DSMB and interim analysis

An independent Data and Safety Monitoring Board (DSMB) oversees the trial. On 23 March 2020 the DSMB conducted a single, planned interim analysis at the anticipated halfway point of the trial and recommended the trial to continue without modification (see DSMB charter in online supplemental file 2) and details of interim analysis in online supplemental file 1, section 22). The

DSMB is composed of two physicians outside the study institution with expertise in adult pulmonary and critical care medicine clinical practice and clinical research, one bioethicist and one biostatistician.

#### Statistical analysis principles

R (R Foundation for Statistical Computing, Vienna, Austria) will be used for analyses. Analyses will be conducted at the level of an individual patient during an individual hospitalisation in an intent-to-treat fashion, unless otherwise specified. Continuous variables will be reported as mean±SD or median and IQR; categorical variables will be reported as frequencies and proportions.

#### Main analysis of the primary outcome

The main analysis will be an intention-to-treat comparison of the primary outcome of VFDs between the higher, intermediate and lower SpO<sub>9</sub> target groups among all patients enrolled in the trial except<sup>1</sup> those admitted during one of the 7-day washout periods and those with a laboratory-confirmed diagnosis of COVID-19. Patients with a diagnosis of COVID-19 will be excluded from the main analysis for two reasons. First, the majority of the PILOT trial occurred prior the COVID-19 pandemic, with too few 2-month study blocks occurring during the pandemic to ensure balance in the number of patients with COVID-19 between trial groups. Second, at the study hospital, ICU patients diagnosed with COVID-19 are transferred to a separate, dedicated COVID-19 ICU that was not participating in the PILOT trial. Thus, patients with COVID-19 are unlikely to have received significant exposure to the SpO<sub>9</sub> target intervention in the PILOT trial. Patients enrolled during washout periods and patients diagnosed with COVID-19 will be included in sensitivity analyses (see Sensitivity analyses below).

It is possible to estimate a conditional effect, which is interpreted as the effect of a given SpO<sub>2</sub> target on an individual patient given the values of the covariates for that patient, or a marginal effect, which is interpreted as the population effect of implementing a given SpO<sub>2</sub> target as a general policy.<sup>52</sup> Since an SpO<sub>2</sub> target intervention may be applied both at the patient level as an individual intervention and at the unit level as a general policy, both may be of interest.

To estimate the conditional effect, we will use a proportional odds model with independent covariates of group assignment (higher, intermediate or lower  ${\rm SpO_2}$  target) and time.  $^{53}$  Time (in days) will be treated as a continuous variable with values ranging from 1 (first day of enrolment) to 1097 (final day of enrolment) and will be analysed using restricted cubic splines with multiple knots to allow for non-linearity resulting from seasonality or secular trends. For the purposes of declaring a statistically significant difference between groups in the primary endpoint, we will consider the conditional effect from the proportional odds model and a two-sided p value of 0.05.

To estimate the marginal effect, we will use generalised estimating equations with study period as the cluster and an independent variable for group assignment (higher, intermediate or lower SpO<sub>9</sub> target).

For both approaches, in addition to assessing for an overall group effect within the model, we will estimate the differences between each pair of  ${\rm SpO_2}$  targets by extracting 95% CIs from the model.

#### Sensitivity analyses of the primary outcome

- ▶ We will repeat the primary analysis using alternative statistical approaches to comparing the VFDs outcome between groups such as zero-inflated Poisson regression or zero-inflated negative binomial regression, global rank scale analysis and Fine and Gray competing risk regression.
- We will repeat the primary analysis with adjustment for prespecified baseline covariates of age, sex, race and ethnicity, source of ICU admission, vasopressor receipt, acute diagnoses at enrolment, and severity of illness as assessed by the non-respiratory SOFA score.
- ▶ We will repeat the primary analysis replacing the continuous covariate of time with a categorical covariate of season defined as: winter (January, February, March); spring (April, May, June); summer (July, August, September); and fall (October, November, December).
- ▶ We will repeat the primary analysis among all patients enrolled in the trial, including¹ patients initiated on invasive mechanical ventilation in a study location during one of the prespecified 7-day washout periods and² patients with a diagnosis of COVID-19.

#### Analysis of effect modification for the primary outcome

We will examine whether prespecified baseline variables modify the effect of study group on the primary outcome using formal tests of statistical interaction in a proportional odds model. Independent variables will include study group assignment, the potential effect modifier of interest and the interaction between the two (eg, study group × presence of sepsis or septic shock) and time. Significance will be determined by the p value for the interaction term, with values <0.10 considered to suggest a potential interaction and values <0.05 considered to confirm an interaction.

We will examine whether the following baseline variables modify the effect of study group on the primary outcome:

- 1. Age;
- 2. Race and ethnicity (Hispanic, non-Hispanic Black, non-Hispanic white, Other);
- 3. Source of admission to the ICU (ED, hospital ward, another ICU in the study hospital, operating room, outside hospital);
- 4. Duration of invasive mechanical ventilation prior to enrollment;
- 5. Chronic comorbidities (categories are not mutually exclusive)
  - Receipt of supplemental oxygen at place of residence prior to hospital admission (yes, no);



- ii. Coronary artery disease or heart failure with reduced ejection fraction (yes, no);
- 6. Acute diagnoses at enrollment (categories are not mutually exclusive) 56
  - i. cardiac arrest (yes, no);
  - ii. acute myocardial infarction (yes, no);
  - iii. sepsis or septic shock (yes, no);
  - iv. acute respiratory distress syndrome (yes, no);
- 7. Receipt of vasopressors at enrollment (yes, no);
- 8. Non-respiratory SOFA score at enrollment;
- 9. Time period before the COVID-19 pandemic (July 2018 to December 2019), and during the COVID-19 pandemic (January 2020 to August 2021).

#### Analysis of the secondary outcome

The sole prespecified secondary outcome of 28-day in-hospital mortality will be compared between the three study groups in an intention-to-treat fashion in the main analysis population using a logistic regression model with independent covariates of group assignment (higher, intermediate or lower  ${\rm SpO_2}$  target) and time. In addition to assessing for an overall group effect within the model, we will estimate the differences between each pair of  ${\rm SpO_2}$  targets by extracting 95% CIs from the model.

#### Analysis of the exploratory outcomes

Each of the exploratory outcomes will be compared between groups in an intention-to-treat fashion in the main analysis population. Exploratory outcomes will be compared between study groups in a similar manner as for primary and secondary outcomes. A logistic model will be used for binary outcomes, a multinomial model for categorical outcomes, and a proportional odds model will be used for ordinal and continuous outcomes.

#### Trial status

PILOT is an ongoing pragmatic trial comparing higher, intermediate and lower  ${\rm SpO_2}$  targets for mechanically ventilated critically ill adults. Patient enrolment began on 1 July 2018 and is anticipated to conclude on 31 August 2021.

#### **Ethics and dissemination**

#### IRB approval

The trial was approved by the IRB of Vanderbilt University Medical Center with a waiver of informed consent (IRB# 171272), details of which are provided in (online supplemental file 1, section 26). Participants who regain capacity to provide informed consent, or legally authorised surrogate decision-makers for those patients who do not regain the capacity to provide informed consent, are approached to provide informed consent for assessment of long-term outcomes as a part of the independently funded CO-PILOT study (R21AG063126).

#### Information for patients and families

An information sheet providing an IRB approved lay language summary of the study and containing the contact information for investigators (who remain available throughout the study period to provide additional information to patients and families on request) is made available throughout the study period in glass display cases near the public entrance to the ICU and near the centre of the ICU, in the 'welcome packet' of information about the ICU, which is distributed at the time of ICU admission to patients, families and surrogates by the medical receptionist or charge nurse as a part of routine admission processes, in a brochure holder in the family waiting room for the study ICU, and by treating physicians and respiratory therapist to any patients, families, or surrogates with questions or concerns about the study.

#### Protocol changes

Any changes to the trial protocol will be recorded on ClinicalTrials.Gov as per SPIRIT guidelines (see section 27 of online supplemental file 1).

#### Data handling and sharing

For details of privacy, data handling and data sharing, see sections 28–29 of online supplemental file 1.

#### Dissemination plan

Trial results will be submitted to a peer-reviewed journal for consideration of publication and will be presented at scientific conferences. The results of the study will be disseminated to patients and the public at the completion of the trial.

The full list of the PILOT investigators may be found in (online supplemental file 1, section 1).

#### **Author affiliations**

<sup>1</sup>Department of Medicine, Division of Allergy, Pulmonary and Critical Care Medicine, Vanderbilt University School of Medicine, Nashville, Tennessee, USA <sup>2</sup>Division of Respiratory Care, Vanderbilt University Medical Center, Nashville, Tennessee, USA

<sup>3</sup>Department of Pharmaceutical Services, Vanderbilt University Medical Center, Nashville, Tennessee, USA

<sup>4</sup>Department of Medicine, Vanderbilt University Medical Center, Nashville, Tennessee. USA

<sup>5</sup>Department of Biostatistics, Vanderbilt University Schoool of Medicine, Nashville, TN. USA

<sup>6</sup>Department of Anesthesiology, Vanderbilt University Medical Center, Nashville, Tennessee. USA

<sup>7</sup>Department of Emergency Medicine, Vanderbilt University Medical Center, Nashville, Tennessee, USA

#### Twitter Bradley D. Lloyd @BradLloydVFL

Collaborators PILOT Investigators Department of Anesthesiology – Robert E Freundlich\*, Jonathan P Wanderer\* Department of Biostatistics – Christopher J Lindsell\*, Li Wang\* Department of Emergency Medicine – Jin H Han, Wesley H Self\* Department of Internal Medicine – John H Brems\*, Kevin G Buell\* Department of Pharmaceutical Services – Sneha Patel, Joanna L Stollings \*Division of Allergy, Pulmonary, and Critical Care Medicine – Gordon R. Bernard\*, Jonathan D Casey\*, Christina Cleveland, Margaret A Hays\*, Luis E Huerta, Karen Jackson, Todd W Rice\*, Megan Roth\*, Matthew W Semler\* Division of Respiratory Care – Pamela G Hastings\*, Bradley D Lloyd\*, Roger K Richardson, J Craig Rooks All at Vanderbilt University Medical Center in Nashville, Tennessee. Asterisk (\*) denotes members of the writing committee.

Contributors Study concept and design was done by MWS, JDC, CJL, GB, WHS and TWR. Drafting of the manuscript was done by MWS, LW and CJL. Critical revision of the manuscript for important intellectual content was performd by MWS, JDC, BDL, PH, MH, MR, JS, JB, KGB, LW, CJL, RF, JPW, GB, WHS and TWR. LW and



CJL were responsible for statistical analysis. Study supervision was done by GB, WHS and TWR.

Funding This study was supported in part by a grant from the National Heart Lung and Blood Institute (K23HL143053). JDC was supported in part by the NIH (K23HL153584). REF was supported in part by the NIH (1KL2TR002245, 1K23HL148640). TWR was supported in part by the NIH (U01HL123033, UL1TR002244). Data collection used the Research Electronic Data Capture (REDCap) tool developed and maintained with Vanderbilt Institute for Clinical and Translational Research grant support (UL1 TR000445 from the National CenterCentre for Advancing Translational Sciences). The funding institutions had no role in (1) conception, design or conduct of the study, (2) collection, management, analysis, interpretation or presentation of the data or (3) preparation, review or approval of the manuscript.

Competing interests All authors completed and submitted the ICMJE Form for Disclosure of Potential Conflicts of Interest. RF reported receiving grant funding and consulting fees from Medtronic and stock from 3M outside the current work. TWR reported receiving consulting fees from Cumberland Pharmaceuticals outside the current work. The authors declared no potential conflicts of interest with the current work.

Patient consent for publication Not applicable.

Provenance and peer review Not commissioned; externally peer reviewed.

Supplemental material This content has been supplied by the author(s). It has not been vetted by BMJ Publishing Group Limited (BMJ) and may not have been peer-reviewed. Any opinions or recommendations discussed are solely those of the author(s) and are not endorsed by BMJ. BMJ disclaims all liability and responsibility arising from any reliance placed on the content. Where the content includes any translated material, BMJ does not warrant the accuracy and reliability of the translations (including but not limited to local regulations, clinical guidelines, terminology, drug names and drug dosages), and is not responsible for any error and/or omissions arising from translation and adaptation or otherwise.

Open access This is an open access article distributed in accordance with the Creative Commons Attribution Non Commercial (CC BY-NC 4.0) license, which permits others to distribute, remix, adapt, build upon this work non-commercially, and license their derivative works on different terms, provided the original work is properly cited, appropriate credit is given, any changes made indicated, and the use is non-commercial. See: http://creativecommons.org/licenses/by-nc/4.0/.

#### **ORCID ID**

Matthew W Semler http://orcid.org/0000-0002-7664-8263

#### **REFERENCES**

- Wunsch H, Linde-Zwirble WT, Angus DC, et al. The epidemiology of mechanical ventilation use in the United States. Crit Care Med 2010;38:1947–53.
- Wunsch H, Angus DC, Harrison DA, et al. Comparison of medical admissions to intensive care units in the United States and United Kingdom. Am J Respir Crit Care Med 2011;183:1666–73.
- 3 Adhikari NKJ, Fowler RA, Bhagwanjee S, et al. Critical care and the global burden of critical illness in adults. Lancet 2010;376:1339–46.
- 4 , Brower RG, Matthay MA, et al, Acute Respiratory Distress Syndrome Network. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med 2000;342:1301–8.
- 5 Esteban A, Frutos-Vivar F, Muriel A, et al. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med 2013;188:220–30.
- 6 Fridovich I. Oxygen toxicity: a radical explanation. J Exp Biol 1998;201:1203–9.
- 7 Heffner JE, Repine JE. Pulmonary strategies of antioxidant defense. Am Rev Respir Dis 1989;140:531–54.
- 8 Freeman BA, Crapo JD. Hyperoxia increases oxygen radical production in rat lungs and lung mitochondria. *J Biol Chem* 1981;256:10986–92.
- 9 Waxman AB, Einarsson O, Seres T, et al. Targeted lung expression of interleukin-11 enhances murine tolerance of 100% oxygen and diminishes hyperoxia-induced DNA fragmentation. J Clin Invest 1998;101:1970–82.
- 10 Griffith DE, Garcia JG, James HL, et al. Hyperoxic exposure in humans. Effects of 50 percent oxygen on alveolar macrophage leukotriene B4 synthesis. Chest 1992;101:392–7.

- 1 Davis WB, Rennard SI, Bitterman PB, et al. Pulmonary oxygen toxicity. early reversible changes in human alveolar structures induced by hyperoxia. N Engl J Med 1983;309:878–83.
- 12 Aggarwal NR, Brower RG. Targeting normoxemia in acute respiratory distress syndrome may cause worse short-term outcomes because of oxygen toxicity. *Ann Am Thorac Soc* 2014;11:1449–53.
- 13 Meade MO, Cook DJ, Guyatt GH, et al. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA 2008;299:637–45.
- 14 Eastwood G, Bellomo R, Bailey M, et al. Arterial oxygen tension and mortality in mechanically ventilated patients. *Intensive Care Med* 2012;38:91–8.
- 15 de Jonge E, Peelen L, Keijzers PJ, et al. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care 2008;12:R156.
- 16 Allen BS, Ilbawi MN. Hypoxia, reoxygenation and the role of systemic leukodepletion in pediatric heart surgery. *Perfusion* 2001;16 Suppl:19–29.
- 17 Allen BS. The reoxygenation injury: is it clinically important? *J Thorac Cardiovasc Surg* 2002;124:16–19.
- 18 Supplemental therapeutic oxygen for prethreshold retinopathy of prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. *Pediatrics* 2000;105:295–310.
- 19 SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network, Carlo WA, Finer NN, et al. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med 2010;362:1959–69.
- 20 Schmidt B, Whyte RK, Asztalos EV, et al. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. JAMA 2013:309:2111–20.
- 21 BOOST II United Kingdom Collaborative Group, BOOST II Australia Collaborative Group, BOOST II New Zealand Collaborative Group, et al. Oxygen saturation and outcomes in preterm infants. N Engl J Med 2013;368:2094–104.
- 22 Panwar R, Hardie M, Bellomo R, et al. Conservative versus liberal oxygenation targets for mechanically ventilated patients. a pilot multicenter randomized controlled trial. Am J Respir Crit Care Med 2016;193:43–51.
- 23 Asfar P, Schortgen F, Boisramé-Helms J, et al. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a twoby-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med 2017;5:180–90.
- 24 Girardis M, Busani S, Damiani E, et al. Effect of conservative vs conventional oxygen therapy on mortality among patients in an intensive care unit: the oxygen-ICU randomized clinical trial. JAMA 2016;316:1583–9.
- 25 Barrot L, Asfar P, Mauny F, et al. Liberal or conservative oxygen therapy for acute respiratory distress syndrome. N Engl J Med 2020;382:999–1008.
- 26 ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group, Mackle D, Bellomo R, et al. Conservative oxygen therapy during mechanical ventilation in the ICU. N Engl J Med 2020;382:989-998.
- 27 Schjørring OL, Klitgaard TL, Perner A, et al. Lower or higher oxygenation targets for acute hypoxemic respiratory failure. N Engl J Med Overseas Ed 2021;384:1301–11.
- 28 Siemieniuk RAC, Chu DK, Kim LH-Y, et al. Oxygen therapy for acutely ill medical patients: a clinical practice guideline. BMJ 2018;363:k4169.
- 29 National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network, Rice TW, Wheeler AP, et al. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA 2012;307:795–803.
- 30 Rice TW, Wheeler AP, Thompson BT, et al. Enteral omega-3 fatty acid, gamma-linolenic acid, and antioxidant supplementation in acute lung injury. JAMA 2011;306:1574–81.
- 31 O'Driscoll BR, Howard LS, Earis J, et al. Bts guideline for oxygen use in adults in healthcare and emergency settings. *Thorax* 2017;72:ii1–90.
- 32 Panwar R, Capellier G, Schmutz N, et al. Current oxygenation practice in ventilated patients-an observational cohort study. *Anaesth Intensive Care* 2013;41:505–14.
- 33 Suzuki S, Eastwood GM, Peck L, et al. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care 2013;28:647–54.



- 34 Helmerhorst HJ, Schultz MJ, van der Voort PH, et al. Self-reported attitudes versus actual practice of oxygen therapy by ICU physicians and nurses. Ann Intensive Care 2014;4:23.
- 35 Self WH, Semler MW, Rice TW. Oxygen targets for patients who are critically ill: emerging data and state of equipoise. *Chest* 2020;157:487–8.
- 36 SPIRIT. Explanation and elaboration: guidance for protocols of clinical trials. - PubMed - NCBI, 2013. Available: https://www.ncbi. nlm.nih.gov/pubmed/23303884 [Accessed 08 Jan 2018].
- 37 Ware JH, Hamel MB. Pragmatic trials--guides to better patient care? N Engl J Med 2011;364:1685–7.
- 38 Beasley R, Chien J, Douglas J, et al. Thoracic society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: 'swimming between the flags'. Respirology 2015;20:1182–91.
- 39 Brower RG, Lanken PN, MacIntyre N, et al. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med 2004;351:327–36.
- 40 Briel M, Meade M, Mercat A, et al. Higher vs lower positive endexpiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA 2010;303:865–73.
- 41 Semler MW, Rice TW, Shaw AD, et al. Identification of major adverse kidney events within the electronic health record. J Med Syst 2016;40:167.
- 42 Semler MW, Noto MJ, Stollings J. Effect of saline versus balanced crystalloids on major adverse kidney events in the medical intensive care unit: the salt randomized trial. Am J Respir Crit Care Med 2016;193:A4290.
- 43 Semler MW, Self WH, Wang L, et al. Balanced crystalloids versus saline in the intensive care unit: study protocol for a clusterrandomized, multiple-crossover trial. *Trials* 2017;18.
- 44 Harris PA, Taylor R, Thielke R, et al. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42:377–81.
- 45 Schoenfeld DA, Bernard GR, ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of

- treatments for acute respiratory distress syndrome. Crit Care Med 2002;30:1772–7.
- 46 Harhay MO, Wagner J, Ratcliffe SJ, et al. Outcomes and statistical power in adult critical care randomized trials. Am J Respir Crit Care Med 2014;189:1469–78.
- 47 Vincent JL, Moreno R, Takala J, et al. The SOFA (sepsis-related organ failure assessment) score to describe organ dysfunction/ failure. on behalf of the Working group on sepsis-related problems of the European Society of intensive care medicine. *Intensive Care Med* 1996;22:707–10.
- 48 , Ranieri VM, Rubenfeld GD, et al, ARDS Definition Task Force. Acute respiratory distress syndrome: the Berlin definition. JAMA 2012;307:2526–33.
- 49 Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO clinical practice guideline for acute kidney injury. Kidney inter 2012;2:8 https://kdigo.org/guidelines/acutekidney-injury/
- 50 Thygesen K, Alpert JS, Jaffe AS, et al. Fourth universal definition of myocardial infarction (2018). J Am Coll Cardiol 2018;72:2231–64.
- 51 Semler MW, Self WH, Wanderer JP, et al. Balanced crystalloids versus saline in critically ill adults. N Engl J Med 2018;378:829–39.
- 52 Zeger SL, Liang KY, Albert PS. Models for longitudinal data: a generalized estimating equation approach. *Biometrics* 1988:44:1049–60.
- 53 Turner RM, White IR, Croudace T, et al. Analysis of cluster randomized cross-over trial data: a comparison of methods. Stat Med 2007;26:274–89.
- 54 Parienti J-J, Kuss O. Cluster-crossover design: a method for limiting clusters level effect in community-intervention studies. *Contemp Clin Trials* 2007;28:316–23.
- 55 Beitler JR, Sarge T, Banner-Goodspeed VM, et al. Effect of titrating positive end-expiratory pressure (PEEP) with an esophageal pressure-guided strategy vs an empirical high PEEP-Fio2 strategy on death and days free from mechanical ventilation among patients with acute respiratory distress syndrome: a randomized clinical trial. JAMA 2019;321:846.
- 56 Munshi L, Ferguson ND. Evolving issues in oxygen therapy in acute care medicine. JAMA 2020;323:607.

# **ONLINE SUPPLEMENT TO:**

# Protocol and Statistical Analysis Plan for the Pragmatic Investigation of Optimal Oxygen Targets (PILOT) Clinical Trial

# **Contents**

| 6 | UPPLEMENTAL METHODS | 3 |
|---|---|---|
| | 1. List of PILOT Investigators | 3 |
| | 2. SPIRIT 2013 Checklist | 4 |
| | 3. Prior Clinical Trials of Oxygen Targets for Adult ICU Patients | 11 |
| | 4. Rationale for Cluster-level Allocation | 13 |
| | 5. Rationale for Targeting SpO <sub>2</sub> versus PaO <sub>2</sub> | 15 |
| | 6. Approach to Monitoring SpO <sub>2</sub> | 16 |
| | 7. Feedback on SpO <sub>2</sub> Target Adherence | 17 |
| | 8. SpO <sub>2</sub> Targets in Patients who return to Invasive Mechanical Ventilation | 18 |
| | 9. Liberation from Mechanical Ventilation | 19 |
| | 10. Protocol for Ventilator Management in the Study ICU | 20 |
| | 11. Protocol for Assessment of Pain (CPOT score) in the Study ICU | 21 |
| | 12. Protocol for Assessment of Agitation (RASS score) in the Study ICU | 22 |
| | 13. Protocol for Delirium Assessment (CAM-ICU score) in the Study ICU | 23 |
| | 14. Protocol for Management of Pain, Agitation, and Delirium in the Study ICU | 24 |
| | 15. Protocol for Daily Spontaneous Awakening Trial (SAT) Safety Screen, SAT Performance Spontaneous Breathing Trial (SBT) Safety Screen, and SBT Performance | |
| | 16. Protocol for Early Mobility in the Study ICU | 26 |
| | 17. Treatment Decisions Determined by Treating Clinicians during the Study | 27 |
| | 18. Data Collected at Each Timepoint | 28 |
| | 19. Definition of Days Alive and Free of a Supportive Therapy | 30 |
| | 20. Measures of Separation between Groups and Processes of Care | 31 |
| | 21. Assessment of Compliance with the Assigned SpO <sub>2</sub> Target | 32 |
| | 22. Interim Analysis | 33 |
| | 23. Pre-specified Baseline Co-variates | 34 |
| | 24. Corrections for Multiple Testing | 35 |
| | 25. Handling of Missing Data | 36 |

| 26. Rationale for Waiver of Informed Consent | 37 |
|------------------------------------------------|----|
| 27. Plan for Communication of Protocol Changes | 39 |
| 28. Patient Privacy and Data Storage | |
| 29. Data Sharing Plan | |
| SUPPLEMENTAL TABLES | 42 |
| Table S1. Modified Non-respiratory SOFA Score | 42 |
| SUPPLEMENTAL REFERENCES | |

#### SUPPLEMENTAL METHODS

# 1. List of PILOT Investigators

Department of Anesthesiology - Robert E. Freundlich\*, Jonathan P. Wanderer\*

Department of Biostatistics – Christopher J. Lindsell\*, Li Wang\*

Department of Emergency Medicine - Jin H. Han, Wesley H. Self\*

Department of Internal Medicine - John H. Brems\*, Kevin G. Buell\*

Department of Pharmaceutical Services - Sneha Patel, Joanna L. Stollings\*

Division of Allergy, Pulmonary, and Critical Care Medicine – Gordon R. Bernard\*,

Jonathan D. Casey\*, Christina Cleveland, Margaret A. Hays\*, Luis E. Huerta, Karen

Jackson, Todd W. Rice\*, Megan Roth\*, Matthew W. Semler\*

Division of Respiratory Care – Pamela G. Hastings\*, Bradley D. Lloyd\*, Roger K.

Richardson, J. Craig Rooks

All at Vanderbilt University Medical Center in Nashville, TN

<sup>\*</sup>denotes members of the writing committee

# 2. SPIRIT 2013 Checklist



# SPIRIT 2013 Checklist:

Recommended items to address in a clinical trial protocol and related documents\*

| Section/item | Item<br>No | Description | Addressed<br>on page<br>number |
|---|---|---|---|
| Administrative | infor | mation | |
| Title | 1 | Descriptive title identifying the study design, population, interventions, and, if applicable, trial acronym | 1 |
| Trial | 2a | Trial identifier and registry name. If not yet registered, name of intended registry | 3 |
| registration | 2b | All items from the World Health Organization Trial Registration Data Set | 3 |
| Protocol version | 3 | Date and version identifier | 2 |
| Funding | 4 | Sources and types of financial, material, and other support | |
| Roles and | 5a | Names, affiliations, and roles of protocol contributors | 1, sup 2_ |
| responsibilities | 5b | Name and contact information for the trial sponsor | 1 |
| | 5c | Role of study sponsor and funders, if any, in study design; collection, management, analysis, and interpretation of data; writing of the report; and the decision to submit the report for publication, including whether they will have ultimate authority over any of these activities | 1-2 |

| | 5d | Composition, roles, and responsibilities of the coordinating center, steering committee, endpoint adjudication committee, data management team, and other individuals or groups overseeing the trial, if applicable (see Item 21a for data monitoring committee) | 1 |
|---|---|---|---|
| Introduction | | | |
| Background<br>and rationale | 6a | Description of research question and justification for undertaking the trial, including summary of relevant studies (published and unpublished) examining benefits and harms for each intervention | <u>5-6</u> |
| | 6b | Explanation for choice of comparators | 5,6, 9 |
| Objectives | 7 | Specific objectives or hypotheses | 6 |
| Trial design | 8 | Description of trial design including type of trial (eg, parallel group, crossover, factorial, single group), allocation ratio, and framework (eg, superiority, equivalence, noninferiority, exploratory) | 6-7 |
| Methods: Part | icipan | ts, interventions, and outcomes | |
| Study setting | 9 | Description of study settings (eg, community clinic, academic hospital) and list of countries where data will be collected. Reference to where list of study sites can be obtained | 7 |
| Eligibility<br>criteria | 10 | Inclusion and exclusion criteria for participants. If applicable, eligibility criteria for study centers and individuals who will perform the interventions (eg, surgeons, psychotherapists) | 7-8 |
| Interventions | 11a | Interventions for each group with sufficient detail to allow replication, including how and when they will be administered | 9-11 |

| | 11b | Criteria for discontinuing or modifying allocated interventions for a given trial | 11-12 |
|---|---|---|---|
| | | participant (eg, drug dose change in response to harms, participant request, or improving/worsening disease) | |
| | 11c | Strategies to improve adherence to intervention protocols, and any procedures for monitoring adherence (eg, drug tablet return, laboratory tests) | Sup 17 |
| | 11d | Relevant concomitant care and interventions that are permitted or prohibited during the trial | 12-13 |
| Outcomes | 12 | Primary, secondary, and other outcomes, including the specific measurement variable (eg, systolic blood pressure), analysis metric (eg, change from baseline, final value, time to event), method of aggregation (eg, median, proportion), and time point for each outcome. Explanation of the clinical relevance of chosen efficacy and harm outcomes is strongly recommended | 14-17 |
| Participant<br>timeline | 13 | Time schedule of enrolment, interventions (including any run-ins and washouts), assessments, and visits for participants. A schematic diagram is highly recommended (see Figure) | Fig 1 |
| Sample size | 14 | Estimated number of participants needed to achieve study objectives and how it was determined, including clinical and statistical assumptions supporting any sample size calculations | 15-16 |
| Recruitment | 15 | Strategies for achieving adequate participant enrollment to reach target sample size | 15 |

**Methods: Assignment of interventions (for controlled trials)** 

Allocation:

| Sequence<br>generation | 16a | Method of generating the allocation sequence (eg, computer-generated random numbers), and list of any factors for stratification. To reduce predictability of a random sequence, details of any planned restriction (eg, blocking) should be provided in a separate document that is unavailable to those who enroll participants or assign interventions | _8-9 |
|---|---|---|---|
| Allocation concealment mechanism | 16b | Mechanism of implementing the allocation sequence (eg, central telephone; sequentially numbered, opaque, sealed envelopes), describing any steps to conceal the sequence until interventions are assigned | _8-9, Fig 2 |
| Implementati<br>on | 16c | Who will generate the allocation sequence, who will enroll participants, and who will assign participants to interventions | _8-10 |
| Blinding<br>(masking) | 17a | Who will be blinded after assignment to interventions (eg, trial participants, care providers, outcome assessors, data analysts), and how | _12 |
| | 17b | If blinded, circumstances under which unblinding is permissible, and procedure for revealing a participant's allocated intervention during the trial | _NA |
| Methods: Data | colle | ction, management, and analysis | |
| Data collection methods | 18a | Plans for assessment and collection of outcome, baseline, and other trial data, including any related processes to promote data quality (eg, duplicate measurements, training of assessors) and a description of study instruments (eg, questionnaires, laboratory tests) along with their reliability and validity, if known. Reference to where data collection forms can be found, if not in the protocol | _13-14_ |
| | 18b | Plans to promote participant retention and complete follow-up, including list of any outcome data to be collected for participants who discontinue or deviate from intervention protocols | 13 |

| Data<br>management | 19 | Plans for data entry, coding, security, and storage, including any related processes to promote data quality (eg, double data entry; range checks for data values). Reference to where details of data management procedures can be found, if not in the protocol | 13 |
|---|---|---|---|
| Statistical methods | 20a | Statistical methods for analyzing primary and secondary outcomes. Reference to where other details of the statistical analysis plan can be found, if not in the protocol | 16-21 |
| | 20b | Methods for any additional analyses (eg, subgroup and adjusted analyses) | 16-21 |
| | 20c | Definition of analysis population relating to protocol non-adherence (eg, as randomized analysis), and any statistical methods to handle missing data (eg, multiple imputation) | 16,21 |
| Methods: Mon | itoring | g | |
| Data<br>monitoring | 21a | Composition of data monitoring committee (DMC); summary of its role and reporting structure; statement of whether it is independent from the sponsor and competing interests; and reference to where further details about its charter can be found, if not in the protocol. Alternatively, an explanation of why a DMC is not needed | 16 |
| | 21b | Description of any interim analyses and stopping guidelines, including who will have access to these interim results and make the final decision to terminate the trial | <u>Sup 34</u> |
| Harms | 22 | Plans for collecting, assessing, reporting, and managing solicited and spontaneously reported adverse events and other unintended effects of trial interventions or trial conduct | _Sup 17,34 |
| Auditing | 23 | Frequency and procedures for auditing trial conduct, if any, and whether the process will be independent from investigators and the sponsor | Sup 17 |
# **Ethics and dissemination**

| Research ethics approval | 24 | Plans for seeking research ethics committee/institutional review board (REC/IRB) approval | <u>22</u> |
|---|---|---|---|
| Protocol amendments | 25 | Plans for communicating important protocol modifications (eg, changes to eligibility criteria, outcomes, analyses) to relevant parties (eg, investigators, REC/IRBs, trial participants, trial registries, journals, regulators) | Sup 40 |
| Consent or assent | 26a | Who will obtain informed consent or assent from potential trial participants or authorized surrogates, and how (see Item 32) | 22 |
| | 26b | Additional consent provisions for collection and use of participant data and biological specimens in ancillary studies, if applicable | 22 |
| Confidentiality | 27 | How personal information about potential and enrolled participants will be collected, shared, and maintained in order to protect confidentiality before, during, and after the trial | Sup 40 |
| Declaration of interests | 28 | Financial and other competing interests for principal investigators for the overall trial and each study site | 2 |
| Access to data | 29 | Statement of who will have access to the final trial dataset, and disclosure of contractual agreements that limit such access for investigators | _Sup 40-42_ |
| Ancillary and post-trial care | 30 | Provisions, if any, for ancillary and post-trial care, and for compensation to those who suffer harm from trial participation | NA |
| Dissemination policy | 31a | Plans for investigators and sponsor to communicate trial results to participants, healthcare professionals, the public, and other relevant groups (eg, via publication, reporting in results databases, or other data sharing arrangements), including any publication restrictions | 23 |
| | 31b | Authorship eligibility guidelines and any intended use of professional writers | Sup 2 |

| | 31c | Plans, if any, for granting public access to the full protocol, participant-levelSup 42_ dataset, and statistical code |
|---|---|---|
| Appendices | | |
| Informed consent materials | 32 | Model consent form and other related documentation given to participants andNA_ authorized surrogates |
| Biological<br>specimens | 33 | Plans for collection, laboratory evaluation, and storage of biological specimens forNA_ genetic or molecular analysis in the current trial and for future use in ancillary studies, if applicable |

<sup>\*</sup>It is strongly recommended that this checklist be read in conjunction with the SPIRIT 2013 Explanation & Elaboration for important clarification on the items. Amendments to the protocol should be tracked and dated. The SPIRIT checklist is copyrighted by the SPIRIT Group under the Creative Commons "Attribution-NonCommercial-NoDerivs 3.0 Unported" license.

# 3. Prior Clinical Trials of Oxygen Targets for Adult ICU Patients

To date, five small-to-moderate sized clinical trials have examined SpO2 targets among adult ICU patients [1–6]. The first trial compared a lower SpO<sub>2</sub> target (88-92%) with a higher SpO<sub>2</sub> target (96-100%) among 103 mechanically ventilated patients [1]. Targeting these SpO<sub>2</sub> ranges produced adequate separation between groups in SpO<sub>2</sub>, PaO<sub>2</sub>, and FiO<sub>2</sub> without any concern for safety, but the trial was not powered to detect differences in clinical outcomes. The second trial enrolled mechanically ventilated adults with septic shock and reported a numerically higher mortality for those randomized to an FiO<sub>2</sub> of 1.0 compared with those randomized to an SpO<sub>2</sub> target of 88-95% [2]. The third trial reported an 8% absolute reduction in mortality with use of an SpO<sub>2</sub> target of 94-98% compared to 97-100% among 434 patients in a single ICU [3]. These findings were limited by early study termination and the authors concluded that a larger trial was needed [3]. The fourth trial compared use of an SpO<sub>2</sub> target of 88-92% versus 96-100% among 205 mechanically ventilated adults with acute respiratory distress syndrome [4]. No statistically significant difference was observed between groups. Although outcomes appeared to numerically favor the higher SpO<sub>2</sub> target group, interpretation was limited by early study termination. The fifth trial enrolled 1000 ICU patients within 2 hours of the initiation of mechanical ventilation [5]. Patients in the intervention group received the lowest FiO<sub>2</sub> that maintained SpO<sub>2</sub> > 90%. Patients in the control group received oxygen therapy at the discretion of treating clinicians targeting SpO2 values between 91-100%. No difference between groups in clinical outcomes was observed, although modest separation between groups and sample size may have limited power to detect differences in patient-centered outcomes. The sixth trial randomized 2,928 adult ICU

patients with acute hypoxemic respiratory failure on at least 10 liters of oxygen per minute or a fraction of inspired oxygen of at least 0.5 to a PaO<sub>2</sub> target of either 60 mm Hg or 90 mm Hg. The trial reported no significant differences between groups in 90-day mortality, ventilator-free days, or new episodes of shock, myocardial ischemia, ischemic stroke, or intestinal ischemia.

#### 4. Rationale for Cluster-level Allocation

Group assignment in the PILOT trial occurs at the level of the ICU (cluster) for several reasons. In routine clinical care in the study ICU, titration of FiO<sub>2</sub> to maintain SpO<sub>2</sub> for all mechanically ventilated adults is performed by 2 to 4 respiratory therapists, with input from nurses and physicians. The management of mechanical ventilation (selection of tidal volume, titration of positive end-expiratory pressure, screening for and performance of spontaneous breathing trials) is governed by unit-wide protocols implemented by the 2 to 4 respiratory therapists for all patients in the unit. Assigning the entire unit to a single SpO<sub>2</sub> target emulates the way mechanical ventilation is managed during clinical care and limits contamination that might result from a respiratory therapist managing multiple patients assigned to different SpO<sub>2</sub> targets.

Additionally, exposure to excess FiO<sub>2</sub>, hyperoxemia, and hyperoxia is most common in the minutes-to-hours immediately following initiation of invasive mechanical ventilation [7,8]. In a recent randomized trial examining tracheal intubation of critically ill adults, the median values for lowest SpO<sub>2</sub> and highest FiO<sub>2</sub> were 97% and 1.0, respectively, in the first hour of invasive mechanical ventilation, compared with 96% and 0.6 between 1 hour and 6 hours and 94% and 0.5 between 6 hours and 24 hours [9]. Even brief periods of early hyperoxia or hypoxia may affect organ function [10–12] and clinical outcomes [13–16]. Enrollment immediately after initiation of invasive mechanical ventilation minimizes pre-study exposure to excess FiO<sub>2</sub>, hyperoxemia, and hyperoxia and facilitates on-study separation between groups. Multiple prior trials examining SpO<sub>2</sub> targets have aimed to enroll patients shortly after the initiation of invasive mechanical ventilation [5,17]. In these patient-level parallel-group trials,

however, the logistical challenges of performing screening, enrollment, randomization, and study group assignment immediately following initiation of invasive mechanical ventilation resulted in the exclusion of 60-90% of eligible patients – raising concern for systematic exclusion of important patient groups (e.g., patients with higher acuity of illness). In PILOT, group assignment at the cluster level allows enrollment immediately on initiation of invasive mechanical ventilation in the ED or ICU. This approach emulates the manner in which oxygen therapy is managed in practice, precludes systematic exclusion of important patient groups, decreases pre-study exposure to hyperoxia and hypoxia, and facilitates early separation in oxygen therapy between groups.

# 5. Rationale for Targeting SpO<sub>2</sub> versus PaO<sub>2</sub>

SpO<sub>2</sub> is measured continuously via non-invasive pulse oximetry for nearly all mechanically ventilated ICU patients. In contrast, PaO<sub>2</sub> is assessed via arterial puncture intermittently and selectively, with most measurements occurring early in the admission of severely ill patients. Similar to prior clinical trials of oxygen therapy during mechanical ventilation [1,5], the PILOT trial targets SpO<sub>2</sub> rather than PaO<sub>2</sub> for patients with functioning non-invasive pulse oximetry monitoring. For patients in the PILOT trial for whom non-invasive pulse oximetry monitoring is unavailable or inaccurate (e.g., inadequate plethysmography signal due to hypoperfusion), PaO<sub>2</sub> values corresponding to the assigned SpO<sub>2</sub> target are used to guide oxygen therapy [18].

# 6. Approach to Monitoring SpO<sub>2</sub>

For all mechanically ventilated patients in the study ED and ICU, SpO₂ is continuously monitored using Nellcor™ SpO₂ Adhesive Sensors (Medtronic, Minneapolis, MN), which measure changes in red and infrared light absorption in an arteriolar bed throughout the pulse cycle to report a non-normalized real-time plethysmographic waveform and arterial hemoglobin saturation values averaged over the prior 6 seconds with a mean difference between SpO₂ and SaO₂ < 2% for SpO₂ values 80-100% [19]. Plethysmography and SpO₂ values are displayed [1] on IntelliVue MP90 bedside patient monitors (PHILIPS, Amsterdam, Netherlands) in each ED and ICU room, [2] on telemetry monitors located at ED and ICU nursing stations and adjacent to the respiratory therapy office, and [3] in real-time in the institutional electronic health record, available from any physical location. SpO₂ values are archived every 60 seconds into an Enterprise Data Warehouse [20–22].

# 7. Feedback on SpO<sub>2</sub> Target Adherence

During the study, the IntelliVue MP90 bedside patient monitors in each room are set to generate an alarm for  $SpO_2$  values outside the range considered to be at goal for the assigned  $SpO_2$  target group. For example, for patients in the intermediate  $SpO_2$  target group,  $SpO_2$  values 92-96% generate no alarm, whereas  $SpO_2$  values  $\leq 91\%$  or  $\geq 97\%$  generate an alarm alerting nursing staff and respiratory therapy to the out-of-range value.

Study personnel remotely monitor SpO<sub>2</sub> values every four hours from 4 AM through 10 PM Monday through Friday and during a 10% sample of night and weekend hours to identify instances of lag between out-of-range SpO<sub>2</sub> values and FiO<sub>2</sub> titration, provide feedback and support to respiratory therapists and bedside nurses, and identify barriers to achieving the assigned SpO<sub>2</sub> target.

Prior to the trial, all respiratory therapists, nurses, and supervising physicians who practice in the study ICU received formal training in the study protocol. Throughout the duration of the study, study personnel attend respiratory therapy group meetings, nursing unit board meetings, and ICU physician leadership meetings to provide continuing education about the study, reinforce elements of the study protocol including the process for SpO<sub>2</sub> target modification by treating clinicians, screen for safety concerns or potential adverse events, and identify and address barriers to achieving the SpO<sub>2</sub> targets.

# 8. SpO<sub>2</sub> Targets in Patients who return to Invasive Mechanical Ventilation

Patients who discontinue invasive mechanical ventilation and return to invasive mechanical ventilation in a study location during the same two-month study period continue to be managed using the same assigned SpO<sub>2</sub> target. Similarly, patients who are transferred out from a study location and return to receiving invasive mechanical ventilation in a study location during the same two-month study period continue to be managed using the same assigned SpO<sub>2</sub> target. Patients who remain on invasive mechanical ventilation in a study location through the end of a two-month study period receive the SpO<sub>2</sub> target assigned by the study until midnight on the night that the two-month study period ends, after which time treating clinicians determine the SpO<sub>2</sub> target with which the patient is managed. Similarly, for patients who are enrolled during one two-month study period, discontinue invasive mechanical ventilation or transferred out of the study location, and return to receiving invasive mechanical ventilation during a subsequent two-month study period, treating clinicians determine the SpO<sub>2</sub> target with which the patient is managed during the subsequent episode of invasive mechanical ventilation.

#### 9. Liberation from Mechanical Ventilation

Each day of mechanical ventilation, all patients in the study ICU are assessed for safety of a spontaneous awakening trial (SAT) and spontaneous breathing trial (SBT) [23] using the SAT and SBT safety criteria from the Awakening and Breathing Controlled trial [24]. To prevent patients in the higher SpO<sub>2</sub> target group from experiencing delays in qualifying for an SBT based on receipt of higher FiO<sub>2</sub> to achieve the higher SpO<sub>2</sub> target, patients in all groups are allowed to qualify for an SAT and SBT regardless of their current FiO<sub>2</sub> or PEEP settings, as long as the other SAT and SBT Safety Screen criteria are met and treating clinicians feel performance of an SAT and SBT is safe. Definitions of SAT and SBT failure and the ventilator settings and duration of the SBT are the same as those used in the ABC trial and during clinical care in the study ICU. For patients who have passed an SBT, the decision to discontinue invasive mechanical ventilation is made by the treating clinicians.

#### 10. Protocol for Ventilator Management in the Study ICU

# **Predicted Body Weight (PBW) Calculation:**

Males: PBW (kg) = (height in inches -60)\*2.3+50 Females: PBW (kg) = (height in inches -60)\*2.3+45.5

Mode: Assist Control

Tidal volume: 6 ml/kg PBW

**Respiratory rate**: Set to maintain 60-70% minute ventilation prior to tracheal intubation. Adjust rate to maintain pH 7.30-7.45, NOT TO EXCEED 35 bpm or PC02 < 25.

**I:E Ratio**: Avoid inverse ratio ventilation

#### PEEP titration:

| FiO2 | 0.3-0.4 | 0.4 | 0.5 | 0.5 | 0.6 | 0.7 | 0.7 | 0.7 | 8.0 | 0.9 | 0.9 | 0.9 | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PEEP | 5 | 8 | 8 | 10 | 10 | 10 | 12 | 14 | 14 | 14 | 16 | 18 | 18-25 |

Wean patient to the lowest level of FiO2 & PEEP while maintaining goal SpO2.

#### **Acidosis Management:**

- 1. If pH <7.30, increase RR to 35 as needed.
- 2. If pH remains <7.3 with RR = 35 call House Officer
- 3. If pH <7.15, consider bicarbonate administration, may increase TV by 1 ml/kg PBW increments until pH is >7.15 or TV = 8 ml/kg PBW (under these conditions Pplat targets [see below] may be exceeded).

**Alkalosis Management:** If pH >7.45, decrease RR.

#### **Management of Tidal Volume:**

- 1. Titrate TV by 1ml/kg increments (minimum of 4ml/kg PBW) to maintain a Pplat below 30cm H2O.
- 2. Measure & record Pplat (0.5 sec inspiratory pause), SpO2, Total RR, TV and pH (if available) at least every 4 hours AND after each change in PEEP or TV.

# 11. Protocol for Assessment of Pain (CPOT score) in the Study ICU

| Indicator | Assessment | Score | Description |
|---|---|---|---|
| Facial expressions | Relaxed, neutral | 0 | No muscle tension observed |
| | Tense | 1 | Presence of frowning, brow lowering, orbit<br>tightening and levator contraction or any other<br>change (e.g. opening eyes or tearing during<br>nociceptive procedures) |
| | Grimacing | 2 | All previous facial movements plus eyelid tightly closed (the patient may present with mouth open or biting the endotracheal tube) |
| Body movements | Absence of movements or normal position | 0 | Does not move at all (doesn't necessarily mean<br>absence of pain) or normal position (movements not<br>aimed toward the pain site or not made for the<br>purpose of protection) |
| | Protection | 1 | Slow, cautious movements, touching or rubbing the pain site, seeking attention through movements |
| | Restlessness/Agitation | 2 | Pulling tube, attempting to sit up, moving limbs/thrashing, not following commands, striking at staff, trying to climb out of bed |
| Compliance with the ventilator (intubated patients) | Tolerating ventilator or movement | 0 | Alarms not activated, easy ventilation |
| • | Coughing but tolerating | 1 | Coughing, alarms may be activated but stop spontaneously |
| OR | Fighting ventilator | 2 | Asynchrony: blocking ventilation, alarms frequently activated |
| Vocalizations (extubated patients) | Talking in normal tone or no sound | 0 | Talking in normal tone or no sound |
| | Sighing, moaning | 1 | Sighing, moaning |
| | Crying out, sobbing | 2 | Crying out, sobbing |
| Muscle tension | Relaxed | 0 | No resistance to passive movements |
| | Tense, rigid | 1 | Resistance to passive movements |
| Evaluate by passive flexion and extension of the upper limbs when patient is at rest or evaluation when | Very tense or rigid | 2 | Strong resistance to passive movements or incapacity to complete them |
| TOTAL | | /8 | |

Adapted from: https://www.icudelirium.org/medical-professionals/assess-prevent-and-manage-pain

Gélinas, C. (2010). Nurses' Evaluations of the Feasibility and the Clinical Utility of the Critical-Care Pain Observation Tool. Pain Management Nursing, 11(2), 115-125.

Arbour, C., & Gélinas, C. (2011). Ask the Experts. Setting Goals for Pain Management When Using a Behavioral Scale: Example With the Critical-Care Pain Observation Tool. Critical Care Nurse, 31, 66-68.

## 12. Protocol for Assessment of Agitation (RASS score) in the Study ICU



Reproduced with permission from:

https://www.icudelirium.org/medical-professionals/delirium/monitoring-delirium-in-the-icu

# 13. Protocol for Delirium Assessment (CAM-ICU score) in the Study ICU

#### Confusion Assessment Method for the ICU (CAM-ICU) Flowsheet 1. Acute Change or Fluctuating Course of Mental Status: **CAM-ICU** negative Is there an acute change from mental status baseline? <u>OR</u> **NO DELIRIUM** Has the patient's mental status fluctuated during the past 24 hours? YES 2. Inattention: Squeeze my hand when I say the letter 'A'." CAM-ICU negative 0 - 2 Read the following sequence of letters: SAVEAHAART or CASABLANCA or ABADBADAAY **NO DELIRIUM Errors** ERRORS: No squeeze with 'A' & Squeeze on letter other than 'A' If unable to complete Letters → Pictures , > 2 Errors **RASS** other 3. Altered Level of Consciousness CAM-ICU positive **Current RASS level** than zero DELIRIUM Present RASS = zero 4. Disorganized Thinking: > 1 Error 1. Will a stone float on water? 2. Are there fish in the sea? 3. Does one pound weigh more than two? 4. Can you use a hammer to pound a nail? 0 - 1 Command: "Hold up this many fingers" (Hold up 2 fingers) Error CAM-ICU negative "Now do the same thing with the other hand" (Do not demonstrate) **NO DELIRIUM** "Add one more finger" (If patient unable to move both arms)

Copyright © 2002, E. Wesley Ely, MD, MPH and Vanderbilt University, all rights reserved

#### Reproduced with permission from:

https://www.icudelirium.org/medical-professionals/delirium/monitoring-delirium-in-the-icu

# 14. Protocol for Management of Pain, Agitation, and Delirium in the Study ICU



Reproduced with permission from:

https://www.icudelirium.org/medical-professionals/delirium/monitoring-delirium-in-the-icu

# 15. Protocol for Daily Spontaneous Awakening Trial (SAT) Safety Screen, SAT Performance, Spontaneous Breathing Trial (SBT) Safety Screen, and SBT Performance



Adapted for the PILOT trial from the "Wake Up and Breathe Flowchart", found at: https://www.icudelirium.org/medical-professionals/both-sat-and-sbt

# 16. Protocol for Early Mobility in the Study ICU



# 17. Treatment Decisions Determined by Treating Clinicians during the Study

All treatment decisions except choice of SpO<sub>2</sub> target during invasive mechanical ventilation of are made by treating clinicians, including: approach to oxygen therapy before invasive mechanical ventilation; use of non-invasive ventilation before invasive mechanical ventilation; choice of ventilator mode during invasive mechanical ventilation; approach to positive end-expiratory pressure during invasive mechanical ventilation; administration of neuromuscular blocking agents, inhaled epoprostenol, prone positioning, or extracorporeal membrane oxygenation; administration of vasopressors or ionotropes, antimicrobial medications, diuretics, intravenous fluid, or blood products; arterial or venous blood gas measurement, measurement of lactate concentration, measurement of central or mixed venous oxygen saturation.

# 18. Data Collected at Each Timepoint

### Enrollment (Day 0)

- Data collected by both manual and automated methods: age; sex; race; ethnicity; height, weight; time from presentation to the study hospital to enrollment; time from ICU admission to enrollment; time from first receipt of invasive mechanical ventilation to enrollment; study location at enrollment; source of admission to the ICU;
- Data collected only by manual method: baseline comorbidities; acute illnesses at enrollment; indication for invasive mechanical ventilation
- 3. Data collected only by automated method: non-respiratory Sequential Organ Failure Assessment (SOFA) score [25] (see supplemental appendix); Elixhauser Comorbidity Index [26]; Glasgow Coma Scale score [27]; vital signs (temperature, heart rate, systolic blood pressure, diastolic blood pressure, SpO<sub>2</sub>); mechanical ventilator settings (mode, set and exhaled tidal volume, set and actual respiratory rate, positive end-expiratory pressure, peak pressure, FiO<sub>2</sub>); serum laboratory values (white blood cell count, hemoglobin, platelet count, sodium, potassium, bicarbonate, creatinine, bilirubin, alanine aminotransferase, aspartate aminotransferase, lactate, arterial pH, PaO<sub>2</sub>, SaO<sub>2</sub>).

#### On-Study (Days 0-28)

- 1. Data collected only by manual method:
  - a. For the subset of all patient enrolled during the first 12 months of the trial,
     physician manual review blinded to study group assignment will determine

- whether each patient experienced acute respiratory distress syndrome (ARDS) by Berlin criteria [28], atrial arrhythmia, ventricular arrhythmia, cardiac arrest, pneumothorax or pneumomediastinum, ischemic stroke, or myocardial infarction.
- b. For the full duration of the trial, each time treating clinicians, patients, or families elect to modify the assigned SpO<sub>2</sub> target, study personnel will record the date and time of the modification, the SpO<sub>2</sub> range to which the target was modified, and the rationale for modifying the SpO<sub>2</sub> target.
- c. Each weekday, study personnel will record for each patient the results of the SAT Safety Screen, SAT, SBT Safety Screen, and SBT.
- 2. Data collected only by automated method: vital signs, ventilator settings, and serum laboratory values (as above); receipt of extracorporeal membrane oxygenation; receipt of neuromuscular blockade; receipt of inhaled epoprostenol; receipt of red cell transfusion; number of arterial blood gases; non-respiratory SOFA score; Richmond Agitation and Sedation Score [29]; Confusion Assessment Method for the ICU (CAM-ICU) score [30].

#### Termination (Day 28)

Data collected by both manual and automated methods: death prior to hospital discharge; time from enrollment to death; duration of ICU admission; duration of hospital admission; duration of invasive mechanical ventilation; receipt of vasopressors; duration of vasopressor receipt; receipt of renal replacement therapy; duration of renal replacement therapy receipt.

# 19. Definition of Days Alive and Free of a Supportive Therapy

Each of the outcomes related to the number of days alive and free of a specific supportive therapy (e.g., vasopressor-free days, renal replacement therapy-free days, ICU-free days, and hospital-free days) will be defined using the same approach as the primary outcome of ventilator-free days.

Days alive and free of the supportive therapy will be defined as the number of calendar days alive and free of the supportive therapy from the final receipt of the supportive therapy through 28 days after enrollment [67,68]. The day of enrollment will be considered to be day 0. Outcome ascertainment will cease at the time of hospital discharge or 28 days after enrollment, whichever occurs first.

Receipt of the supportive therapy will be considered to end at the time of the patient's final receipt of the supportive therapy between enrollment and 28 days after enrollment. Patients who continue to receive the supportive therapy at day 28 will receive a value of zero. Patients who die prior to day 28 will receive a value of zero. Patients who are discharged from the hospital prior to day 28 and are receiving the supportive therapy at the time of discharge will receive a value of zero. Patients who are removed from the supportive therapy and are discharged from the hospital without the supportive therapy prior to 28 days will be assumed to remain free of the supportive therapy between hospital discharge and day 28. For patients who are removed from the supportive therapy, return to receiving the supportive therapy, and are subsequently removed again from the supportive therapy prior to day 28, days alive and free of the supportive therapy will be counted from the final receipt of the supportive therapy prior to day 28.

# 20. Measures of Separation between Groups and Processes of Care

#### Measures of Separation between Groups

- 1. SpO<sub>2</sub> during invasive mechanical ventilation
- 2. SaO<sub>2</sub> during invasive mechanical ventilation
- 3. FiO<sub>2</sub> during invasive mechanical ventilation
- 4. PaO<sub>2</sub> during invasive mechanical ventilation
- 5. Episodes of hypoxemia, including:
  - a.  $SpO_2 < 85\%$  for  $\geq 5$  minutes
  - b.  $SpO_2 < 80\%$  for  $\ge 5$  minutes
  - c.  $SpO_2 < 70\%$  for  $\ge 2$  minutes
- 6. Episodes of hyperoxemia, including:
  - a.  $SpO_2 > 98\%$  for  $\geq 5$  minutes
  - b.  $SpO_2 > 98\%$  for  $\ge 30$  minutes
- 7. Proportion of patients with a value for PaO<sub>2</sub> < 55 mm Hg
- 8. Proportion of patients with a value for PaO<sub>2</sub> > 120 mm Hg

#### Measures of Processes of Care

- 1. Tidal volume
- 2. Positive end-expiratory pressure
- 3. Peak airway pressure
- 4. Receipt of mandatory ventilator mode
- 5. Number of arterial blood gasses
- 6. Hemoglobin
- 7. Red cell transfusion

# 21. Assessment of Compliance with the Assigned SpO<sub>2</sub> Target

All SpO<sub>2</sub> values measured during invasive mechanical ventilation are assessed for compliance with the assigned SpO<sub>2</sub> target. An SpO<sub>2</sub> value is considered compliant with the trial protocol if any of the following conditions are met:

- 1. Measured SpO<sub>2</sub> is within the target range
- 2. Measured SpO<sub>2</sub> is above the target range and the FiO<sub>2</sub> is 21%
- 3. Measured SpO<sub>2</sub> is below the target range and the FiO<sub>2</sub> is 100%
- 4. Measured SpO<sub>2</sub> occurs after treating clinicians have completed an SpO<sub>2</sub> target modification sheet

# 22. Interim Analysis

On March 23, 2020, the DSMB conducted a single, planned interim analysis for efficacy and safety at the anticipated halfway point of the trial. The interim analysis included data from patients enrolled during the first 18 months of the trial. According to the criteria specified in the trial protocol, the stopping boundary for efficacy would have been met if the P value for the difference between groups was <0.001 using a proportional odds model with independent covariates of group assignment (higher, intermediate, or lower SpO<sub>2</sub> target) and time. A stopping boundary for futility was not pre-specified. After conducting the planned interim analysis, the DSMB recommended the study continue without modification.

The DSMB reserves the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety.

Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05).

# 23. Pre-specified Baseline Co-variates

We will repeat the primary analysis with adjustment for the following pre-specified baseline covariates: age (continuous), sex (male, female), race and ethnicity (Hispanic, Non-Hispanic Black, Non-Hispanic White, Other), source of ICU admission (ED, hospital ward, another ICU in the study hospital, operating room, outside hospital), vasopressor receipt (yes, no), and acute diagnoses at enrollment (cardiac arrest, acute myocardial infarction, sepsis or septic shock, acute respiratory distress syndrome), and severity of illness as assessed by the non-respiratory SOFA score.

To account for non-linear relationships, continuous variables will be analyzed using restricted cubic splines with between 3 and 5 knots.

# 24. Corrections for Multiple Testing

We have pre-specified a single primary outcome and a single secondary outcome. Consistent with recommendations of the Food and Drug Administration [65] and the European Medicines Association [66], each will be tested using a two-sided p-value with a significance level of 0.05. For all other analyses, emphasis will be placed on the estimate of effect size with 95% confidence intervals, as recommended by the *International Committee of Medical Journal Editors* [67], and no corrections for multiple comparisons will be performed.

# 25. Handling of Missing Data

The primary outcome of VFDs is not anticipated to be missing for any patients. Missing data will not be imputed for the primary outcome or any secondary or exploratory outcomes. None of the covariates pre-specified for the adjusted analysis are anticipated to be missing for any patients. In additional adjusted analyses, any missing data for covariates will be imputed using multiple imputations.

#### 26. Rationale for Waiver of Informed Consent

For all mechanically ventilated ICU patients, FiO<sub>2</sub> is titrated to maintain SpO<sub>2</sub> as a part of clinical care. In current clinical care, 98% of SpO<sub>2</sub> values experienced by mechanically ventilated adult ICU patients fall between 88-100% [31,32]. Within this range, current guidelines for oxygen therapy in mechanically ventilated adults advocate contrasting approaches: [1] tolerating SpO<sub>2</sub> values as low as 88% (NIH/NHLBI ARDS Network) [33], [2] titrating within the range 92-96% (Thoracic Society of Australia and New Zealand) [34], or [3] allowing SpO<sub>2</sub> values above 96% (British Thoracic Society) [35]. The lower SpO<sub>2</sub> target, intermediate SpO<sub>2</sub> target, and higher SpO<sub>2</sub> target examined in this study are all intermittently used in routine clinical care in the study ICU and are all within the range recommended by at least one international guideline. No high-quality data suggest that one SpO2 target is better than the others for patient outcomes. During the PILOT trial, whenever treating clinicians feel that the optimal SpO<sub>2</sub> target for a specific patient is known, that SpO<sub>2</sub> target is used. Thus, the PILOT trial only determines the SpO<sub>2</sub> target for patients whose treating clinicians are uncertain which SpO<sub>2</sub> target would be optimal for the patient and feel all three targets represent comparable and reasonable approaches.

Because the SpO<sub>2</sub> targets being compared in the study [1] are common approaches to managing a universal supportive therapy to which patients would be exposed as a part of clinical care if not participating in the study, [2] have no high-quality data suggesting the superiority of one approach over the others, and [3] are all comparable approaches for the patient from the perspective of the treating clinician,

participation in the study presents minimal incremental risk compared to clinical care for mechanically ventilated ICU patients outside of the study.

Initiation of mechanical ventilation for critically ill patients is frequently a time-sensitive procedure. Despite the availability of a formal informed consent document for tracheal intubation and initiation of mechanical ventilation, time allows for discussion of risks and benefits of these clinical procedures in less than 10% of cases during clinical care in the study ICU. Titration of FiO<sub>2</sub> to target SpO<sub>2</sub> in PILOT begins within 15 minutes of the initiation of mechanical ventilation with a goal of intervening during the period with the highest prevalence of excess FiO<sub>2</sub>, hyperoxemia, and hyperoxia. Moreover, in this cluster-randomized trial, the entire ICU is assigned to a single SpO<sub>2</sub> target delivered by the unit's respiratory therapists through a unit-wide oxygen titration protocol. Obtaining informed consent from every patient receiving invasive mechanical ventilation in the study ED and ICU prior to the initiation of invasive mechanical ventilation would be impracticable and would potentially delay delivery of a time-sensitive intervention.

Because the study presents minimal incremental risk, the study does not adversely affect the welfare or privacy rights of the participants, and obtaining informed consent prior to enrollment is impracticable, the study is being conducted with a waiver of informed consent.

# 27. Plan for Communication of Protocol Changes

Any changes to the trial protocol (e.g., changes to eligibility criteria, outcomes, analyses) will require a new version of the full trial protocol which will be tracked with the date of the update and the version number of the trial protocol. A list summarizing the changes that are made with each protocol revision will be included at the end of each protocol. The updated protocol will be sent to the Vanderbilt IRB for approval prior to implementation of the protocol change. At the time of publication, the original trial protocol and the final trial protocol, including the summary of changes made with each protocol change, will be included in the supplementary material for publication.

# 28. Patient Privacy and Data Storage

All patients are assigned a unique study ID number for tracking. Data collected from the medical record is entered into the secure online database REDCap. All data is maintained in the secure online database REDCap until the time of study publication. At the time of publication, a de-identified database will be generated.

# 29. Data Sharing Plan

Upon reasonable request, a completely de-identified data set may be provided by the authors. Request to share data from the PILOT trial should be sent to the principal investigator, Matthew W. Semler, at matthew.w.semler@vumc.org. The dataset will be provided to researchers whose proposed use of the data has been approved by the PILOT steering committee and an Institutional Review Board and is accompanied by an executed Data Use Agreement.

#### **SUPPLEMENTAL TABLES**

Table S1. Modified Non-respiratory SOFA Score.

| | 0 | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|
| Coagulation | > 150 | 101-150 | 51-100 | 21-50 | ≤ 20 |
| Platelets (x10 <sup>3</sup> /mm <sup>3</sup> ) | | | | | |
| Liver | < 1.2 | 1.2-1.9 | 2.0-5.9 | 6.0-11.9 | ≥ 12 |
| Bilirubin (mg/dL) | | | | | |
| Cardiovascular | Mean arterial | Mean arterial | On dopamine | On dopamine | On dopamine |
| Blood pressure | pressure ≥ 70 | pressure < 70 | ≤ <b>5</b> | > 5 | > 15 |
| _ | mmHg and no | mmHg and no | mcg/kg/min or | mcg/kg/min, | mcg/kg/min, |
| | receipt of | receipt of | any | epinephrine ≤ | epinephrine > |
| | dopamine, | dopamine, | dobutamine | 0.1 | 0.1 |
| | dobutamine, | dobutamine, | | mcg/kg/min, | mcg/kg/min, |
| | epinephrine, or | epinephrine, or | | or | or |
| | norepinephrine | norepinephrine | | norepinephrine | norepinephrine |
| | | | | $\leq 0.1$ | > 0.1 |
| | | | | mcg/kg/min | mcg/kg/min |
| Brain | 15 | 13-14 | 10-12 | 6-9 | < 6 |
| Glascow coma score | | | | | |
| Kidney | Creatinine | Creatinine 1.2- | Creatinine 2.0- | Creatinine 3.5- | Creatinine > 5 |
| Renal function | <1.2 mg/dL | 1.9 mg/dL | 3.4 mg/dL | 4.9 mg/dL | mg/dL |

The Sequential Organ Failure Assessment (SOFA) score (Vincent et al Critical Care Medicine 1998) is composed of scores from six organ systems, graded from 0 to 4 according to the degree of dysfunction or failure. Scores range from 0 (no evidence of organ dysfunction or failure) to 24 (evidence of severe dysfunction failure in each of the six organ systems). The modified non-respiratory SOFA score is composed of scores from five of the six organ systems included in the complete SOFA score (excluding the respiratory system), graded on the same scale as the complete SOFA score. Scores range from 0 (no evidence of organ dysfunction or failure) to 20 (evidence of severe organ dysfunction or failure in each of the five organ systems assessed).

#### SUPPLEMENTAL REFERENCES

- 1 Panwar R, Hardie M, Bellomo R, *et al.* Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. *Am J Respir Crit Care Med* 2016;**193**:43–51. doi:10.1164/rccm.201505-1019OC
- 2 Asfar P, Schortgen F, Boisramé-Helms J, et al. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. The Lancet Respiratory Medicine Published Online First: February 2017. doi:10.1016/S2213-2600(17)30046-2
- 3 Girardis M, Busani S, Damiani E, et al. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA 2016;316:1583–9. doi:10.1001/jama.2016.11993
- 4 Barrot L, Asfar P, Mauny F, *et al.* Liberal or Conservative Oxygen Therapy for Acute Respiratory Distress Syndrome. *N Engl J Med* 2020;**382**:999–1008. doi:10.1056/NEJMoa1916431
- 5 ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group, Mackle D, Bellomo R, et al. Conservative Oxygen Therapy during Mechanical Ventilation in the ICU. N Engl J Med Published Online First: 14 October 2019. doi:10.1056/NEJMoa1903297
- 6 Schjørring OL, Klitgaard TL, Perner A, et al. Lower or Higher Oxygenation Targets for Acute Hypoxemic Respiratory Failure. N Engl J Med Published Online First: 20 January 2021. doi:10.1056/NEJMoa2032510
- 7 Kraft F, Andel H, Gamper J, *et al.* Incidence of hyperoxia and related in-hospital mortality in critically ill patients: a retrospective data analysis. *Acta Anaesthesiol Scand* 2018;**62**:347–56. doi:10.1111/aas.13047
- 8 Palmer E, Post B, Klapaukh R, et al. The Association between Supraphysiologic Arterial Oxygen Levels and Mortality in Critically III Patients. A Multicenter Observational Cohort Study. Am J Respir Crit Care Med 2019;200:1373–80. doi:10.1164/rccm.201904-0849OC
- 9 Casey JD, Janz DR, Russell DW, et al. Bag-Mask Ventilation during Tracheal Intubation of Critically Ill Adults. N Engl J Med 2019;380:811–21. doi:10.1056/NEJMoa1812405
- 10 Brenner M, Stein D, Hu P, *et al.* Association between early hyperoxia and worse outcomes after traumatic brain injury. *Arch Surg* 2012;**147**:1042–6. doi:10.1001/archsurg.2012.1560
- 11 Stub D, Smith K, Bernard S, et al. Air Versus Oxygen in ST-Segment-Elevation Myocardial Infarction. Circulation 2015:**131**:2143–50. doi:10.1161/CIRCULATIONAHA.114.014494
- 12 Fessel JP, Flynn CR, Robinson LJ, et al. Hyperoxia synergizes with mutant bone morphogenic protein receptor 2 to cause metabolic stress, oxidant injury, and pulmonary hypertension. Am J Respir Cell Mol Biol 2013;49:778–87. doi:10.1165/rcmb.2012-0463OC
- 13 Page D, Ablordeppey E, Wessman BT, *et al.* Emergency department hyperoxia is associated with increased mortality in mechanically ventilated patients: a cohort study. *Critical Care* 2018;**22**:9. doi:10.1186/s13054-017-1926-4
- 14 Roberts BW, Kilgannon JH, Hunter BR, et al. Association Between Early Hyperoxia Exposure After Resuscitation From Cardiac Arrest and Neurological Disability: Prospective Multicenter Protocol-Directed Cohort Study. Circulation 2018:137:2114–24. doi:10.1161/CIRCULATIONAHA.117.032054

- Kilgannon JH, Jones AE, Shapiro NI, et al. Association between arterial hyperoxia following resuscitation from cardiac arrest and in-hospital mortality. JAMA 2010;303:2165–71. doi:10.1001/jama.2010.707
- 16 Austin MA, Wills KE, Blizzard L, et al. Effect of high flow oxygen on mortality in chronic obstructive pulmonary disease patients in prehospital setting: randomised controlled trial. BMJ 2010;341:c5462. doi:10.1136/bmj.c5462
- 17 Young P, Bailey M, Bellomo R, *et al.* HyperOxic Therapy OR NormOxic Therapy after out-of-hospital cardiac arrest (HOT OR NOT): a randomised controlled feasibility trial. *Resuscitation* 2014;**85**:1686–91. doi:10.1016/j.resuscitation.2014.09.011
- 18 Severinghaus JW. Simple, accurate equations for human blood O2 dissociation computations. *J Appl Physiol Respir Environ Exerc Physiol* 1979;**46**:599–602.
- Harris BU, Char DS, Feinstein JA, et al. Accuracy of Pulse Oximeters Intended for Hypoxemic Pediatric Patients. Pediatr Crit Care Med 2016;17:315–20. doi:10.1097/PCC.0000000000000660
- 20 Buell KG, Casey JD, Wang L, et al. Big Data for Clinical Trials: Automated Collection of SpO2 for a Trial of Oxygen Targets during Mechanical Ventilation. Journal of Medical Systems 2020;44:153. doi:10.1007/s10916-020-01632-4
- 21 Ehrenfeld JM, Funk LM, Van Schalkwyk J, et al. The incidence of hypoxemia during surgery: evidence from two institutions. Can J Anaesth 2010;57:888–97. doi:10.1007/s12630-010-9366-5
- 22 Lopez MG, Pretorius M, Shotwell MS, *et al.* The Risk of Oxygen during Cardiac Surgery (ROCS) trial: study protocol for a randomized clinical trial. *Trials* 2017;**18**:295. doi:10.1186/s13063-017-2021-5
- 23 Stollings JL, Foss JJ, Ely EW, et al. Pharmacist leadership in ICU quality improvement: coordinating spontaneous awakening and breathing trials. Ann Pharmacother 2015;49:883–91. doi:10.1177/1060028015582050
- 24 Girard TD, Kress JP, Fuchs BD, *et al.* Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. *Lancet* 2008;**371**:126–34. doi:10.1016/S0140-6736(08)60105-1
- 25 Vincent JL, Moreno R, Takala J, *et al.* The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. *Intensive Care Med* 1996;**22**:707–10.
- 26 Elixhauser A, Steiner C, Harris DR, et al. Comorbidity measures for use with administrative data. *Med Care* 1998:**36**:8–27.
- 27 Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. *Lancet* 1974;**2**:81–4.
- 28 ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, *et al.* Acute respiratory distress syndrome: the Berlin Definition. *JAMA* 2012;**307**:2526–33. doi:10.1001/jama.2012.5669
- 29 Sessler CN, Gosnell MS, Grap MJ, et al. The Richmond Agitation–Sedation Scale. Am J Respir Crit Care Med 2002;166:1338–44. doi:10.1164/rccm.2107138
- 30 Ely EW, Margolin R, Francis J, et al. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med 2001;29:1370– 9.

- 31 Panwar R, Capellier G, Schmutz N, et al. Current oxygenation practice in ventilated patients-an observational cohort study. *Anaesth Intensive Care* 2013;**41**:505–14.
- 32 Suzuki S, Eastwood GM, Peck L, *et al.* Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. *J Crit Care* 2013;**28**:647–54. doi:10.1016/j.jcrc.2013.03.010
- 33 National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network, Rice TW, Wheeler AP, et al. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. *JAMA* 2012;**307**:795–803. doi:10.1001/jama.2012.137
- 34 Beasley R, Chien J, Douglas J, *et al.* Thoracic Society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: 'Swimming between the flags.' *Respirology* 2015;**20**:1182–91. doi:10.1111/resp.12620
- 35 O'Driscoll BR, Howard LS, Earis J, et al. BTS guideline for oxygen use in adults in healthcare and emergency settings. *Thorax* 2017;**72**:ii1–90. doi:10.1136/thoraxjnl-2016-209729

# DATA AND SAFETY MONITORING BOARD CHARTER

Charter, Data and Safety Monitoring Board for "Preliminary Investigation of optimaL Oxygen Targets (PILOT) trial"

> Matthew W. Semler MD, MSc Li Wang, MS Jonathan D. Casey, MD Todd W. Rice, MD, MSc Wesley H. Self, MD, MPH Gordon R. Bernard, MD

Confidential Information
The information contained within this Charter is confidential and intended for the use of the DSMB members.

| DSMB Member Printed Name | |
|--------------------------|----------|
| DSMB Member Signature | <br>Date |

# Charter, Data and Safety Monitoring Board for the Preliminary Investigation of optimaL Oxygen Targets (PILOT) trial

Version 1.2 6/29/2018

#### 1. Introduction

This Charter is for the Data and Safety Monitoring Board (DSMB) for the <u>Preliminary Investigation of optimal Oxygen Targets</u> (PILOT) trial.

The Charter is intended to be a living document. The DSMB and investigators will review it at regular intervals to determine whether any changes in procedure are needed.

#### 2. Responsibilities of the DSMB

The DSMB is responsible for safeguarding the interests of study participants, assessing the safety and efficacy of study procedures, and for monitoring the overall conduct of the study.

The DSMB is an independent group advisory to the investigators and affiliated institution, and is required to provide recommendations about starting, continuing, and stopping the study. The DSMB makes recommendations about:

- Participant safety and risk/benefit ratio of study procedures and interventions, including whether new data from other sources affects the study
- Initial approval of the protocol and subsequent amendments (with specific attention to study population, intervention, and study procedures)
- Adherence to the protocol requirements
- Completeness, quality, and planned analysis of data
- Ancillary study burden on participants and main study

#### 3. Communication Plan

Communication with DSMB members will be primarily through the DSMB Chair and the primary investigator (Dr. Semler) or study biostatistician (Ms. Wang). Study investigators will not communicate about the study with DSMB members outside of DSMB meetings. The primary investigator may contact the DSMB Chair when needed for urgent concerns or clarifications of recommendations.

#### 4. DSMB Members and Research Staff

DSMB members and their expertise are listed in Appendix A. The DSMB Chair will perform the functions of the Executive Secretary (ES). He will draft meeting summaries, compose final recommendations, and assure the accurate and timely transmission of the final recommendations to the investigators. The primary investigator (Dr. Semler) will be responsible for timely notification of co-investigators of all DSMB recommendations. *Ad hoc* members may be added to supplement expertise for single or multiple meetings.

#### 5. Scheduling, Timing, and Organization of Meetings

DSMB meetings will be held by teleconference. The purpose of the first meeting is to review and discuss this Charter, provide an overview of study activities, review the trial protocol, review the DSMB data reporting template, and finalize the Data and Safety Monitoring Plan. Each DSMB member will sign and return this Charter to the primary investigator (Dr. Semler) to

indicate recommendation for approval. Enrollment in the trial will not begin until the DSMB has recommended approval and IRB approval has been obtained.

- Meetings by teleconference will be held twice a year, with additional meetings scheduled as needed. Conference calls will be scheduled by the primary investigator (Dr. Semler) in collaboration with the DSMB members.
- A single interim analysis will be performed in the 30 days after data on the primary outcome is available for patients enrolled in the first 18 months of the trial.
- The DSMB will conclude its operations when all study procedures, follow up, analysis, and publication of the primary results have been completed.

The agenda for DSMB meetings will be drafted by the primary investigator (Dr. Semler) and study biostatistician (Ms. Wang), and finalized in consultation with the DSMB Chair. The agenda and meeting materials will be distributed by the primary investigator (Dr. Semler) or his appointee, two (2) weeks before each meeting. The NHLBI Program Office will receive this material at the same time as DSMB members.

When the agenda is distributed, DSMB members will be asked to report any new conflicts of interest since the last DSMB meeting. New conflicts will be reviewed by the Chair and study staff to determine if the conflict limits the ability of the DSMB member to participate in the discussion according to conflict of interest policy at the study institution.

To ensure proper trial conduct, at each meeting the DSMB will review the following data:

- adverse events and other safety data,
- quality and completeness of study data, and
- enrollment data

At the single pre-planned interim analysis after 18 months of enrollment, the DSMB will review a formal interim analysis for efficacy by the primary endpoint (as outlined below in the stopping guidelines).

It is expected that all DSMB members will attend every meeting. For the purposes of voting on recommendations, a quorum is three (3) members of the Board. All standing Monitoring Board members are voting members. The Board may also decide in advance whether *ad hoc* members can vote.

#### 6. Organization of Meetings

Meetings are organized into open, closed, and executive sessions.

- Open session information is presented to the DSMB by the study investigators, with time for discussion.
- Closed session the DSMB and blinded study staff (NHLBI program staff may be invited to attend at the Chair's discretion) discuss confidential data (any study data grouped by treatment arm), including information on efficacy and safety. The DSMB can decide to be unblinded to treatment assignments by the study statistician. The principal investigator and staff involved in subject enrollment and treatment may not be present or review grouped data.

- Executive session (optional) DSMB members (and NHLBI program staff at the Chair's discretion) may elect to convene to discuss study issues independently. If the executive session occurs on a conference call, steps will be taken to ensure that only the appropriate participants are on the call, and to invite others to re-join the call only at the conclusion of the executive session.
- Recommendations (optional) Meeting attendees may be reconvened to receive the DSMB's recommendations.

At the conclusion of the closed and executive sessions, the participants will be re-convened so that the DSMB Chair can provide a summary of the DSMB's recommendations. This provides an opportunity for study investigators to ask questions to clarify the recommendations. The meeting is then adjourned.

#### 7. Expedited Safety Reporting

A system has been established to track and report adverse events (AEs). Study personnel will monitor the safety of subjects and follow AEs until the event resolves or is explained.

<u>Clinical Outcomes</u> (not considered Adverse Events). In this study of critically ill patients who are at high risk for death or other adverse outcomes due to their underlying critical illness, clinical outcomes, including death and organ dysfunction, will be systematically tracked (collected in the case report form) and will be included as part of the analyses for this study. For the purposes of reporting, death and organ dysfunction will not be recorded as AEs unless the investigator believes the event may have been caused by the study or is more severe or prolonged than expected given the underlying critical illness. Listed below are events that will be tracked as primary or secondary clinical outcomes and will not therefore be reported as AEs (unless believed to be study related and more severe or prolonged than expected given the underlying critical illness):

- 1. Death (all deaths occurring prior to hospital discharge will be reported on the CRF in the vital status at hospital discharge section);
- 2. Recurrence of respiratory failure, including need for re-intubation or non-invasive mechanical ventilation, presence of acute respiratory distress syndrome, or presence of pneumothorax;
- 3. Circulatory failure, including cardiac arrest or shock with or without receipt of vasopressors;
- 4. Incidence of sustained atrial and ventricular arrhythmias:
- 5. Acute kidney injury, including leading to increased creatinine or receipt of renal replacement therapy;
- 6. Hepatic injury or failure leading to increased bilirubin, AST, or ALT;
- Coagulation derangements leading to elevated PT/INR or PTT, DIC, thrombocytopenia, or thrombocytosis;
- 8. Lactic acidosis;
- 9. Delirium, disability, and physical or cognitive impairment believed to be newly acquired;
- 10. All values for SpO<sub>2</sub>, SaO<sub>2</sub>, FiO<sub>2</sub>, PaO<sub>2</sub>, or PaO<sub>2</sub>/FiO<sub>2</sub> ratio;
- 11. All values for vital signs (e.g., temperature, respiratory rate, SpO2);
- 12. Receipt of co-interventions (e.g., net fluid balance, number of arterial blood gasses, red cell transfusion)
- 13. Duration of ICU admission, ICU readmission;

- 14. Duration of hospitalization, hospital readmission;
- 15. Alterations in routine labs, including chemistries, complete blood counts, liver function tests, and hemostasis profiles.

Adverse Event Classifications. An Adverse Event (AE) will be defined as any untoward medical occurrence for a patient enrolled in the trial that is not tracked as a clinical outcome, regardless of whether the event is considered study related or not. All AEs occurring during the observational study period will be recorded on the CRF. All AEs will then be assessed as to whether they are (1) related to study procedures, (2) serious, and/or (3) unexpected according to the following definitions:

- I. <u>Related to study procedures.</u> AEs that the investigator suspects are related to the study will be classified as study related. Certainty of relatedness is not required as long as a reasonable possibility exists that the AE is related to a study procedure.
- II. <u>Serious.</u> AEs that meet any of the criteria below will be considered Serious Adverse Events (SAEs):
  - a. Results in death
  - b. Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event and NOT an event that hypothetically might have caused death if it would have been more severe)
  - c. Prolongs an existing hospitalization
  - d. Results in persistent or significant disability or incapacity
  - e. Results in a congenital anomaly or birth defect
- f. Important medical event that requires an intervention to prevent any of a-e above.
- III. <u>Unexpected.</u> AEs that are more severe or prolonged than expected based on the investigator's discretion will be considered Unexpected.

Communication and Reporting of Adverse Events. AEs will be recorded in the AE CRF in the electronic database and reported to the primary investigator (Dr. Semler) within 5 calendar days of occurrence. The primary investigator will provide a report of all AEs annually to the IRB, and semi-annually to the DSMB as part of the semi-annual DSMB meetings. All SAEs will be reported to the primary investigator within 72 hours of occurrence. The primary investigator will, in turn, report all SAEs to the IRB, DSMB, and funding body within 7 calendar days of occurrence. Consistent with NHLBI policy, unanticipated problems that do not qualify as an SAE will be reported by the investigator to the IRB, DSMB, and NHLBI within 14 calendar days of the investigator becoming aware of the problem.

Review by the DSMB. All AEs will be reviewed by the DSMB at the scheduled semi-annual DSMB meetings. All SAEs will be reviewed by the DSMB Chair within three (3) days of notification. The DSMB Chair will respond to the primary investigator (Dr. Semler) and NHLBI program office with recommendations within seven (7) days.

#### 8. Reports to the DSMB

For each meeting, the study biostatistician (Ms. Wang) will prepare summary reports and tables to facilitate the oversight role of the DSMB. The DSMB will discuss at the first and subsequent meetings what data they wish to review and how it should be presented (Appendix B).

## 9. Reports of DSMB Deliberations

• Full Summary and Recommendations: The DSMB Chair/ES is responsible for sending the DSMB meeting summary to the Board within seven (7) calendar days of the meeting. The summary should be signed by the DSMB Chair and include key topics discussed, the response of the investigators to previous recommendations, and the recommendations of the DSMB. The study statistician may receive the full summary as decided by the DSMB chair on a meeting by meeting basis.

Voting on recommendations will follow Roberts' Rules of Order (Robert's Rules of Order Newly Revised (11th Edition) RONR.

Board Recommendations - signed by the DSMB Chair, will be sent to the investigators within fourteen (14) calendar days after the meeting. Recommendations should include a statement as to whether the study is approved to continue as planned, should continue with specified changes, or should be stopped. Requests for additional data from the investigators or DCC/statistician should include an expected due date. In addition to recommendations memos issued to investigators (for review and IRB distribution), recommendations related to blinded data or data analysis issues may be issued separately for DCCs or statisticians.

The recommendations will be distributed by the principal investigator to co-investigators, to the local IRB, and to the NHLBI Program Office.

Action plan: This lists the DSMB's recommendations and the primary investigator's
action plan outlining the steps required to implement the DSMB recommendations. It is
submitted to the NHLBI Program Office and DSMB within fourteen (14) calendar days
after the DSMB meeting.

#### 10. Statistical Monitoring Guidelines

In addition to ongoing monitoring of safety throughout the trial, the DSMB will conduct a single interim analysis for efficacy and safety at the anticipated halfway point of the trial. The interim analysis will include patients enrolled during the first 18 months of the trial. The stopping boundary for efficacy will be met if the P value for the difference between groups is <0.001 using a proportional odds mixed effects model accounting for fixed effects (group) and random effects (period) with regard to the primary outcome of VFDs. Use of the conservative Haybittle-Peto boundary (P < 0.001) will allow the final analysis to be performed using an unchanged level of significance (P = 0.05). There will be no stopping boundary for futility. The DSMB will reserve the right to stop the trial at any point, request additional data or interim analyses, or request modifications of the study protocol as required to protect patient safety. If the 18-month interim analysis reveals an enrollment indicative of <80% statistical power at completion, we will ask the DSMB to approve extending enrollment of the study to ensure the trial is not underpowered to detect the planned difference between groups in the primary outcome.

# **PILOT Trial Statistical Analysis Plan Revision Sequence**

| April 2, 2021 | Original Statistical Analysis Plan completed |
|---|---|
| April 5, 2021 | Original Statistical Analysis Plan submitted for publication |
| August 25, 2021 | Statistical Analysis Plan submission completed peer review |
| August 31, 2021 | Final patient enrolled |

October 28, 2021 Final Statistical Analysis Plan\* published:

Semler MW, Casey JD, Lloyd BD, Hastings PG, Hays M, Roth M, Stollings J, Brems J, Buell KG, Wang L, Lindsell CJ, Freundlich RE, Wanderer JP, Bernard GR, Self WH, Rice TW; PILOT Investigators and the Pragmatic Critical Care Research Group. Protocol and statistical analysis plan for the Pragmatic Investigation of optimal Oxygen Targets (PILOT) clinical trial. *BMJ Open.* 2021 Oct 28;11(10):e052013. PMID: 34711597

<sup>\*</sup>No changes to content of the statistical analysis plan occurred between submission of the Protocol and Statistical Analysis Plan and its publication.